# An Open-Label, Randomized, Crossover Study to Assess Nicotine Uptake, Tobacco-Related Biomarkers of Exposure, Biomarkers of Potential Harm, and Puff Topography with Use of mybluTM Electronic Cigarettes in Adult Smokers

NCT# NCT04429932

Study SAP – 26 February 2020

#### Statistical Analysis Plan

An Open-Label, Randomized, Crossover Study to Assess Nicotine Uptake, Tobacco-Related Biomarkers of Exposure, Biomarkers of Potential Harm, and Puff Topography with Use of *my*blu<sup>TM</sup> Electronic Cigarettes in Adult Smokers

Protocol No: NER 01/003 Final Protocol Date: 4 November 2019 Amendment 1 Date: 4 December 2019

Product Names: *my*blu<sup>TM</sup> (freebase), Gold Leaf flavor, 2.4%; *my*blu<sup>TM</sup> (freebase), Polar Mint flavor, 2.4%; *my*blu<sup>TM</sup> (freebase), Cherry flavor, 2.4%; *my*blu<sup>TM</sup> (freebase), Vanilla flavor, 2.4%; *my*blu<sup>TM</sup> (freebase), Gold Leaf flavor, 1.2%; *my*blu<sup>TM</sup> (freebase), Polar Mint flavor, 1.2%; *my*blu<sup>TM</sup> (freebase), Menthol flavor, 2.4%; *my*blu<sup>TM</sup> Intense (nicotine salts), Fresh Mint flavor, 2.4%

Project CA22736 Final Version 1.0 Date: 26 February 2020

Nerudia Ltd Wellington House, Physics Rd, Speke Liverpool L24 9HP, United Kingdom

621 Rose Street Lincoln, Nebraska 68502, USA

# Statistical Analysis Plan Signature Page

Product Names: myblu<sup>™</sup> (freebase), Gold Leaf flavor, 2.4%; myblu<sup>™</sup> (freebase), Polar Mint flavor, 2.4%; myblu<sup>™</sup> (freebase), Cherry flavor, 2.4%; myblu<sup>™</sup> (freebase), Vanilla flavor, 2.4%; myblu<sup>™</sup> (freebase), Gold Leaf flavor, 1.2%; myblu<sup>™</sup> (freebase), Polar Mint flavor, 1.2%; myblu<sup>™</sup> (freebase), Menthol flavor, 2.4%; myblu<sup>™</sup> Intense (nicotine salts), Fresh Mint flavor, 2.4%

Protocol: NER 01/003

Study Title: An Open-Label, Randomized, Crossover Study to Assess Nicotine Uptake, Tobacco-Related Biomarkers of Exposure, Biomarkers of Potential Harm, and Puff Topography with Use of myblu<sup>TM</sup> Electronic Cigarettes in Adult Smokers

Issue Date: 26 February 2020



# **Table of Contents**

| 1. | INTRODUCTION | | | |
|---|---|---|---|---|
| 2. | OBJ | ECTIV | ES AND ENDPOINTS | 5 |
| | 2.1 | | tives | |
| | 2.2 Endpoints | | | |
| 3. | STU | TUDY DESIGN | | |
| 4. | ANA | ANALYSIS POPULATIONS | | |
| | 4.1 | Analy | vsis Populations | 12 |
| | | 4.1.1 | Safety Population | 12 |
| | | 4.1.2 | Outcomes Population | 12 |
| | 4.2 | Prelin | ninary Data and Interim Analysis | |
| 5. | PRO | DUCT | AND STUDY ARM DESCRIPTIONS | 12 |
| 6. | ANA | LYSIS | S OF STUDY ENDPOINTS | 14 |
| | 6.1 | Produ | ct Use Behavior | 14 |
| | | 6.1.1 | Product Use and Data Collection | 14 |
| | | 6.1.2 | Product Use Data Summarization | 14 |
| 6.2 Plasma Nicotine Pharmacokinetics (Part | | | na Nicotine Pharmacokinetics (Part 1 only) | 15 |
| | | 6.2.1 | Measurements and Collection Schedule | 15 |
| | | 6.2.2 | Pharmacokinetic Concentrations | 15 |
| | | 6.2.3 | Plasma Nicotine Pharmacokinetic Parameters | 16 |
| | | 6.2.4 | PK Data Summarization and Presentation | 17 |
| | 6.3 | Biomarkers of Exposure and Potential Harm. | | |
| | | 6.3.1 | Biomarker Sample Collection | 18 |
| | | 6.3.2 | Biomarker Calculations | 19 |
| | | Calcu | lation of Urine Nicotine Equivalents | 19 |
| | | Calcu | lation of Total Mass Excreted | 19 |
| | | Creati | inine Adjustments | 19 |
| | | | Biomarker Data Summarization | |
| | 6.4 | Topog | graphy (Part 1 only) | 20 |
| | | 6.4.1 | Data Collection | 20 |
| | | 6.4.2 | Data Summarization | 20 |
| | 6.5 | Physic | ologic Assessments | 21 |
| | | 6.5.1 | Data Collection | 21 |
| | | 6.5.2 | Data Summarization | 21 |
| | 6.6 | Subje | ctive Measures | 22 |
| | | 6.6.1 | Data Collection | 22 |

# Nerudia Ltd.

# NER 01/003 *my*blu™ E-cigarettes Clinical Study Report No. CA22736

| | _ | 6.6.2 Data Summarization | 23 |
|---|---|---|---|
| | 6.7 | Statistical Analyses | 24 |
| 7. | SAFI | ETY | 27 |
| | 7.1 | Subject Discontinuation | |
| | 7.2 | Demographics | |
| | 7.3 | Smoking History | |
| | 7.4 | Adverse Events | 28 |
| | 7.5 | Clinical Laboratory Tests (Serum Chemistry, Hematology, and Urinalysis) | 28 |
| | 7.6 | Vital Signs | 29 |
| | 7.7 | Electrocardiogram | 29 |
| | 7.8 | Concomitant Medications | 29 |
| | 7.9 | Physical Examination | 30 |
| | 7.10 | Exhaled CO | 30 |
| | 7.11 | Lung Function (Spirometry) | 30 |
| 8. | SUM | MARY OF CHANGES FROM PROTOCOL-PLANNED ANALYSIS | 30 |
| 9. | SUMMARY TABLES AND FIGURES | | |
| | Section 14 Summary Tables and Figures | | 30 |
| | Section 16 Data Listings | | |
| 10. | TAB | LE AND FIGURE SHELLS | 52 |
| | 10.1 | Figures Shells | 53 |
| | 10.2 | Post-Text Summary Tables Shells | 60 |
| 11. | LIST | ING SHELLS | 113 |

#### 1. INTRODUCTION

The following statistical analysis plan (SAP) provides the framework for the summarization of the data from this study. The SAP may change due to unforeseen circumstances. Any changes made from the planned analysis within protocol, after the locking of the database will be documented in the clinical study report (CSR). The section referred to as Table Shells within this SAP describes the traceability of the tables, figures, and listings (TFLs) back to the data.

Any additional exploratory analyses not addressed within this SAP and/or driven by the data, or requested by Nerudia Ltd., will be considered out of scope and must be described in the CSR.

#### 2. OBJECTIVES AND ENDPOINTS

# 2.1 Objectives

#### Primary:

- 1. To characterize nicotine uptake following controlled use of *my*blu<sup>TM</sup> electronic cigarettes (e-cigarettes)
- 2. To assess the change-from-baseline differences in the primary tobacco-related biomarkers of exposure (BoE) following a 9-day use period of *my*blu<sup>TM</sup> e-cigarettes.

#### Secondary:

- 1. To assess the change-from-baseline differences in the primary tobacco-related BoE following a 14-day use period of *my*blu<sup>TM</sup> e-cigarettes.
- 2. To assess the change-from-baseline differences in the secondary tobacco-related BoE following 9-day and 14-day use periods of *my*blu<sup>TM</sup> e-cigarettes.
- 3. To characterize the change in the primary and secondary tobacco-related BoE and biomarkers of potential harm (BoPH) during a 14-day period of use of *my*blu<sup>TM</sup> ecigarettes and compare between exclusive e-cigarette use, exclusive combustible cigarette use and dual (combustible cigarette and e-cigarette) use.
- 4. To assess the change-from-baseline differences in the primary and secondary tobaccorelated BoE between Day 9 and Day 14 in subjects using *my*blu<sup>TM</sup> e-cigarettes, both exclusively and alongside use of combustible cigarettes.
- 5. To assess change-from-baseline differences in BoPH following 9-day and 14-day use periods of *my*blu<sup>TM</sup> e-cigarettes.
- 6. To assess measures of subjective effects associated with use of *my*blu<sup>TM</sup> e-cigarettes.
- 7. To determine puffing topography parameters (puff count, puff duration, puff volume, peak puff flow rate, average puff flow rate, inter puff interval) following an 8-day use period of *my*blu<sup>TM</sup> e-cigarettes and assess change-from-baseline differences (if applicable).

# Clinical Study Report No. CA22736

- 8. To assess change-from-baseline differences in physiologic endpoints (i.e., blood pressure [BP], heart rate [HR], and spirometry) following 9-day and 14-day use periods of *my*blu<sup>TM</sup> e-cigarettes.
- 9. To characterize product use of *my*blu<sup>TM</sup> e-cigarettes under short-term controlled and *ad libitum* use conditions.
- 10. To assess the safety and tolerability of myblu<sup>TM</sup> e-cigarettes following short-term use.

# 2.2 Endpoints

#### **Primary Study Endpoints:**

#### 1. Pharmacokinetics

 $AUC_{0-180}$ ,  $C_{max}$ , and  $T_{max}$  from each controlled product use session on Days 2, 4, 6, and 8.

# 2. Biomarkers of Exposure

Concentration (blood BoE) or 24-hour mass excreted (Urine BoE) for the primary biomarkers of exposure listed below:

| Biomarker | Matrix | <b>Chemical Constituent</b> |
|-----------------------------|--------|-----------------------------|
| Carboxyhemoglobin | Blood | Carbon monoxide (CO) |
| (COHb) | | |
| 4-(methylnitrosamino)-1-(3- | Urine | 4-(methylnitrosamino)-1-(3- |
| pyridyl)-1-butanol (NNAL) | | pyridyl)-1-butanone (NNK) |
| 3-hydroxypropylmercapturic | Urine | Acrolein |
| acid (3-HPMA) | | |
| S-phenyl mercapturic acid | Urine | Benzene |
| (S-PMA) | | |

# **Secondary Study Endpoints:**

#### 1. Biomarkers of Exposure

24-hour mass excreted for the secondary biomarkers of exposure listed below:

| Biomarker | Matrix | <b>Chemical Constituent</b> |
|-------------------------------|--------|-----------------------------|
| N-nitrosonornicotine (NNN) | Urine | NNN |
| 2-cyanoethyl-mercapturic acid | Urine | Acrylonitrile |
| (CEMA) | | |
| Hydroxyethyl mercapturic acid | Urine | Ethylene oxide |
| (HEMA) | | |
| 3-hydroxy-1- | Urine | Crotonaldehyde |
| methylpropylmercapturic acid | | , |
| (HMPMA) | | |

#### Clinical Study Report No. CA22736

| Monohydroxybutenylmercapturic acid (MHBMA) | Urine | 1,3-butadiene |
|--------------------------------------------|-------|---------------|
| Hydroxypyrene (1-OHP) | Urine | Pyrene |
| o-toluidine (o-tol) | Urine | Toluidine |
| 3-hydroxybenzo[a]pyrene (3-OH | Urine | B[a]P |
| B[a]P) | | |
| 1-aminonaphthalene (1-AN) | Urine | Naphthalene |
| 2-aminonaphthalene (2-AN) | Urine | Naphthalene |
| Nicotine equivalents | Urine | Nicotine |

#### 2. Biomarkers of Potential Harm

Concentration (blood BoPH) or 24-hour mass excreted (urine BoPH) for the secondary biomarkers of exposure listed below:

| Biomarker | Matrix | <b>Biological Effect</b> |
|--------------------------------------|--------|--------------------------|
| Soluble intracellular adhesion | Blood | Inflammation |
| molecule (sICAM) | | |
| White blood cells (WBCs) | Blood | Inflammation |
| High density lipoprotein cholesterol | Blood | Inflammation |
| (HDL-C) | | |
| Monocyte chemoattractant protein 1 | Blood | Inflammation |
| (MCP-1) | | |
| Type III isoprostane (8-epi- | Urine | Oxidative stress |
| prostaglandin $F_{2\alpha}$ ) | | |
| 11-dehydrothromboxane B <sub>2</sub> | Urine | Platelet activation |

#### 3. Subjective measures

- Urge to Smoke (Part 1)
  - o Maximum reduction from baseline score (E<sub>max R</sub>)
  - $\circ$  Time of the  $E_{max R}$  ( $TE_{max}$ )
  - Area under the reduction from baseline "Urge to Smoke" visual analog scale (VAS) score versus time curve (AUEC\_R)
- Product Liking Questionnaire VAS responses
- Product Evaluation Scale (PES) factor scores
- Future Intent to Use Questionnaire bipolar VAS scores
- Questionnaire of Smoking Urges-Brief (QSU-Brief) factor scores
- Minnesota Tobacco Withdrawal Scale-Revised (MTWS-R) total score
- Penn State [Electronic] Cigarette Dependence Index (PSCDI, PSECDI) total score
- 4. <u>Puff Topography parameters:</u> puff count, puff duration, puff volume, peak puff flow rate, average flow rate, inter-puff interval
- 5. Physiological Endpoints
- Blood Pressure and Heart Rate: Change from Baseline AUEC0-t, Emax, TEMax

• Pre-bronchodilator and change from pre to post-bronchodilator lung function variables: FEV1, FVC, FEV1:FVC ratio, FEF25-75%

#### 6. Product Use Behavior

# Days 1, 3, 5, 7, and 9

• Pod weight differences

# Days 2, 4, 6, and 8

- Number of inhalations (first (controlled) product use session)
- Duration of each inhalation (first (controlled) product use session)
- Pod weight differences (first (controlled) and second (*ad libitum*) product use sessions)

#### Days 10-14

- Pod weight differences (Arm I and Arm K)
- Number of cigarettes smoked (Arm J and Arm K)

#### 7. <u>Safety Assessments</u>

Safety endpoints will include physical examinations, vital signs, electrocardiograms (ECGs), clinical laboratory tests, AEs, and use of concomitant medications.

#### 3. STUDY DESIGN

This will be an open-label, randomized, 2-part study in adult smokers. All subjects will participate in both study parts. Part 2 will begin immediately after Part 1.

Screening procedures will be performed within 28 days prior to study procedures on Day -2.

Subjects who successfully complete the screening procedures and meet the eligibility criteria will be eligible to check in to the clinical research unit (CRU) on Day -2 and will complete all subjective effects questionnaires for the purpose of familiarization with the questions, scales, and computerized tablet. Subjects will also participate in a brief trial on Day -2 (approximately 30 minutes) using the *my*blu<sup>TM</sup> device with a 0% nicotine e-liquid, to familiarize with the use of the device. Baseline study assessments, including BoE, BoPH, spirometry (Day -1 only), BP, HR, and puff topography (in a subset of 16 subjects [2 subjects from each sequence in Part 1] on Day -1 only) will be performed on Days -2 through -1, as appropriate. Subjects will continue to smoke their usual brand combustible cigarette from check-in through Day -1, but will abstain from use of any tobacco- or nicotine-containing products for at least 12 hours prior to the start of product use on Day 1. Subjects will be randomized to 1 of 8 sequences (Part 1) on Day -1. Sequences are shown in Figure 3.1

Part 1 (Days 1 to 9)

On Days 1, 3, 5, and 7, subjects will use the study product they are assigned to use the following day according to the randomization scheme. Subjects will use the assigned study product *ad libitum* until the start of the abstinence period (i.e., at least 12 hours prior to the start of the first product use session on the next day). A fully charged battery and a fresh pod will be provided on each day. Additional pods will be provided as needed. Pods will be weighed within 24 hours before the start and after completion of product use on each day. On Day 1, puff topography measurements will be performed in the same subset of 16 subjects (2 subjects from each sequence in Part 1) for 1 hour during *ab libitum* product use. Puff topography should be performed within  $\pm$  2 hours of the time of the baseline assessment on Day -1.

On Days 2, 4, 6, and 8, subjects will participate in two product use sessions on each day, using the assigned study product according to the randomization scheme. In the first (controlled) product use session, subjects will use the assigned study product under controlled conditions (i.e., 10 puffs taken at 30-second intervals, with puffs 3 seconds in duration). Blood samples for nicotine pharmacokinetic (PK) assessment will be collected prior to and for 3 hours following the start of the first product use session. Subjects will complete the Urge to Smoke questionnaire during and following the first product use session and the Product Liking, Product Evaluation Scale (PES), and Future Intent to Use questionnaires following the first product use session. Following collection of the last PK blood sample (180-minute time point) and completion of the subjective effects questionnaires, subjects will start the second (ad libitum) product use session, during which they will use the same assigned study product ad libitum (with no limits on puff duration or inter-puff interval) until approximately 23:00. Subjects will complete the Urge to Smoke, Product Liking, PES, and Future Intent to Use questionnaires at least 6 hours after the start of the second product use session. A fresh pod and fully charged device will be provided for each product use session. Pod weights will be measured before and after each product use session. On Day 8, puff topography measurements will be performed in the same subset of 16 subjects (2 subjects from each sequence in Part 1) for 1 hour during the second (ab libitum) product use session. Puff topography will be performed at least 4 hours after the start of the second (ab libitum) product use session and should be within  $\pm 2$  hours of the time of the baseline assessment on Day -1.

On Day 9, subjects may use all or any of the 4 study products (used previously on Days 1 to 8) *ad libitum* until approximately 23:00. For BoE and BoPH assessments, blood samples will be collected on Day 9 and urine samples will be collected over 24 hours (starting on Day 8 after completion of the second [*ab libitum*] product use session). BP and HR measurements will be taken throughout the period of *ad libitum* product use. Subjects will complete the Questionnaire on Smoking Urges-Brief (QSU-Brief), the Minnesota Tobacco Withdrawal Scale-Revised (MTWS-R), and the Penn State [Electronic] Cigarette Dependence Index (PSCDI/PSECDI) questionnaires at least 6 hours after the start of the *ad libitum* product use session on Day 9. Spirometry measurements will be conducted following completion of all subjective effects questionnaires on Day 9. Fresh pods and a fully charged device will be provided on Day 9 and pod weights will be measured.

Depending on the availability of topography equipment, puff topography may not be performed at all scheduled time points and may not be performed for some or all assigned subjects.

Part 2 (Days 10 to 14)

Subjects will be randomized to 1 of 3 study arms (Part 2) on Day 10. Subjects will use any or all of the 8 study products and/or smoke their usual brand combustible cigarettes *ad libitum* for 5 days (until approximately 23:00 on each day) according to the randomization scheme. For BoE and BoPH assessments, blood samples will be collected on Day 14 and urine samples will be collected over 24 hours (starting on Day 13 after the end of product use for that day). On Day 14, BP and HR measurements will be taken throughout the period of *ad libitum* product use/smoking. The QSU-Brief, MTWS-R, and PSCDI/PSECDI questionnaires will be completed at least 6 hours after the start of the *ad libitum* product use session on Day 14. Spirometry measurements will be conducted following completion of all subjective effects questionnaires on Day 14. Product use behavior will be assessed by documenting the number of cigarettes smoked, the flavor and strength of the *my*blu<sup>TM</sup> products, and pod weights, per day, as appropriate. On each study day, fresh pods and a fully charged device will be provided, as appropriate.

The CRU will attempt to contact all subjects who used at least one study product (including subjects who terminate the study early) using their standard procedures approximately 14 days after the last study product use to determine if any adverse event (AE) has occurred since the last study visit.

An overview of the study design is shown in the Figure 3.1.

# Figure 3.1. Study Design Overview



- a: To be performed within 28 days prior to study procedures on Day -2.
- b: Baseline study assessments will be performed on Days -2 and -1 while subjects continue to smoke their usual brand combustible cigarette.
- c: Subjects may use all or any of the 4 study products (i.e., A, B, C, and/or D) *ad libitum* (Ad lib) until approximately 23:00.
- d: Subjects may use all or any of the 4 study products (i.e., E, F, G, and/or H) *ad libitum* (Ad lib) until approximately 23:00.
- e: Subjects will be randomized to 1 of 3 study arms (Part 2) on Day 10 and will use any or all of the 8 study products (Products A to H) and/or smoke their usual brand combustible cigarettes *ad libitum* for 5 days according to the randomization scheme.
- f: The CRU will attempt to contact all subjects who used at least one study product (including subjects who terminate the study early) using their standard procedures approximately 14 days after the last study product used.
- g: Subjects will use *ad libitum* the study product they are assigned to use the following day according to the randomization scheme. Subjects will use the assigned study product *ad libitum* until the start of the abstinence period (i.e., at least 12 hours prior to the start of the first product use session on the next day).
- h: Subjects will complete one set of questionnaires for the purpose of familiarization with subjective effects questions, appropriate use of the VAS, and use of the computerized tablet system.

i: A total of 16 subjects (2 subjects from each sequence in Part 1) will have puff topography evaluated for 1 hour during *ad libitum* product use.

#### 4. ANALYSIS POPULATIONS

# 4.1 Analysis Populations

#### 4.1.1 Safety Population

For Part 1, the Safety Population will include all subjects who used at least one study product from Day -2.

For Part 2, the Safety Population will include all subjects who completed Part 1 and were randomized in Part 2 on Day 10.

# **4.1.2** Outcomes Population

The Outcomes Population (Part 1) is a subset of the Part 1 safety population and will consist of subjects who used a study product and have evaluable Part 1 PK, biomarkers, subjective effects, or topography data. This population will be used in the summary and analysis of Part 1 PK, subjective effects, topography, biomarkers, and product use, and all available data will be included in the summary tables to the extent possible.

The Outcomes Population (Part 2) is a subset of the Part 2 safety population and will consist of subjects who completed Part 1 and have evaluable Part 2 biomarkers, subjective effects, BP, HR, or spirometry data. This population will be used in the summary and analysis of Part 2 biomarkers, subjective effects, BP, HR, spirometry, and product use, and all available data will be included in the summary tables to the extent possible.

#### 4.2 Preliminary Data and Interim Analysis

Biometrics will not perform interim analyses.

#### 5. PRODUCT AND STUDY ARM DESCRIPTIONS

Subjects will be required to bring with them to the CRU a sufficient supply (i.e., 2-week supply [unopened packs]) of their usual brand combustible cigarettes for personal use throughout confinement (if applicable).

The e-cigarette products in Table 5.1 will be used in Part 1 of this study. In the CSR text and table headings, products will be referred to by the short descriptions. In the table footers, the 8 products will be referred to as Products A through H referenced to the long descriptions as shown in the following table:

**Table 5.1. Product Description** 

| Products | Short Description | Long Description |
|---|---|---|
| A | <i>my</i> blu™ Gold Leaf 2.4% | myblu <sup>TM</sup> (freebase), Gold Leaf flavor, 2.4% |
| В | <i>my</i> blu™ Polar Mint 2.4% | <i>my</i> blu <sup>TM</sup> (freebase), Polar Mint flavor, 2.4% |
| С | <i>my</i> blu™ Cherry 2.4% | <i>my</i> blu <sup>™</sup> (freebase), Cherry flavor, 2.4% |
| D | myblu™ Vanilla 2.4% | <i>my</i> blu <sup>™</sup> (freebase), Vanilla flavor, 2.4% |
| Е | <i>my</i> blu™ Gold Leaf 1.2% | <i>my</i> blu <sup>TM</sup> (freebase), Gold Leaf flavor, 1.2% |
| F | <i>my</i> blu™ Polar Mint 1.2% | <i>my</i> blu <sup>™</sup> (freebase), Polar Mint flavor, 1.2% |
| G | <i>my</i> blu™ Menthol 2.4% | <i>my</i> blu <sup>™</sup> (freebase), Menthol flavor, 2.4% |
| Н | <i>my</i> blu <sup>TM</sup> Intense Fresh Mint 2.4% | <i>my</i> blu <sup>TM</sup> Intense (nicotine salts), Fresh Mint flavor, 2.4% |

Similarly, in Part 2, the following descriptions of study arms will be used:

| Arm | Short Description | Long Description |
|---|---|---|
| I | <i>my</i> blu™ | Exclusive use of $my$ blu <sup>TM</sup> products ad libitum |
| J | Combustible Cigarette | Exclusive smoking of usual brand combustible cigarettes <i>ad libitum</i> |
| K | Dual Use | Smoking of usual brand combustible cigarettes (up to 50% of the subject's self-reported CPD) and use of <i>my</i> blu <sup>TM</sup> products <i>ad libitum</i> |

#### 6. ANALYSIS OF STUDY ENDPOINTS

#### 6.1 Product Use Behavior

#### 6.1.1 Product Use and Data Collection

#### Part 1

On Days -2 and -1, subjects will smoke their usual brand combustible cigarette *ad libitum*.

On Days 1, 3, 5, and 7, Subjects will use the assigned study product *ad libitum* until the start of the abstinence period.

On Days 2, 4, 6, and 8, subjects will participate in two product use sessions on each day, using the assigned study product according to the randomization scheme. In the first (controlled) product use session, subjects will use the assigned study product under controlled conditions (i.e., 10 puffs taken at 30-second intervals, with puffs 3 seconds in duration). In the second (*ad libitum*) product use session, they will use the same assigned study product *ad libitum* (with no limits on puff duration or interpuff interval)

On Day 9, subjects may use all or any of the 4 study products (used previously on Days 1 to 8) *ad libitum*.

Pods will be weighed before the start and after completion of product use on each day for Days 1 through 9.

#### Part 2

On Days 10 to 14, subjects will use any or all of the 8 study products and/or smoke their usual brand combustible cigarettes *ad libitum*. The number of cigarettes smoked, the flavor and strength of the *my*blu<sup>TM</sup> products, and pod weights will be documented each day, as appropriate.

#### 6.1.2 Product Use Data Summarization

The following product use variables will be determined:

#### Part 1

Days 1, 3, 5, 7, and 9

• Pod weight differences

#### Days 2, 4, 6, and 8

- Number of inhalations (first (controlled) product use session)
- Duration of each inhalation (first (controlled) product use session)

#### Clinical Study Report No. CA22736

• Pod weight differences (first (controlled) and second (ad libitum) product use sessions)

### Part 2

#### Days 10-14

- Pod weight differences (Arm I and Arm K)
- Number of cigarettes smoked (Arm J and Arm K)

Product use variables will be summarized by study product, product use session, and study day as applicable (Part 1) and by study arm and study day (Part 2) using descriptive statistics presented overall and by sex. When multiple pods are used, the pod weight differences will be calculated using the sums of the weights before and after product use.

The level of precision for each statistic will be presented as follows:

- minimum/maximum in same precision as the data,
- arithmetic mean/median in one more level of precision than minimum/maximum.
- SD in one more level of precision than mean/median,
- n will be presented as an integer,
- arithmetic CV% will be presented to 1 decimal point

#### 6.2 Plasma Nicotine Pharmacokinetics (Part 1 only)

#### **6.2.1** Measurements and Collection Schedule

On each of Days 2, 4, 6, and 8, a 4 mL blood sample for plasma nicotine analysis will be drawn into a plastic K2-EDTA (lavender top) vacutainer tube approximately 5 minutes prior to and at 3, 5, 7, 10, 12, 15, 20, 30, 60, 120 and 180 minutes following the start of the controlled product use episode.

#### **6.2.2** Pharmacokinetic Concentrations

Plasma concentrations of nicotine as determined at the collection times described in Section 6.2.1 will be used for the calculation of the plasma nicotine PK parameters.

All concentration data will be included in the calculation of the individual PK parameters, the individual concentration-time plots (based on actual sample times), and in the mean concentration-time plots (based on nominal sample times). However, if there are any significant deviations from nominal sample times, some concentration data may be excluded from mean concentration-time plots and/or additional concentration-time plots of the mean data may be provided. All deviations and excluded data will be provided and discussed in the CSR.

#### **6.2.3** Plasma Nicotine Pharmacokinetic Parameters

The appropriate noncompartmental PK parameters will be calculated for each controlled product use episode from the baseline adjusted plasma nicotine concentration-time data using Phoenix® WinNonlin® Version 7.0 or higher. Actual sample times will be used in the calculations of the PK parameters. The calculation of the actual time for nicotine will be in respect to the start of product use episodes. All PK parameters included in the protocol are listed in Table 6.1 below, and are defined as appropriate for study design.

Table 6.1. Noncompartmental Pharmacokinetic Parameters to be Calculated (Baseline Adjusted)

| Label to be<br>Used in the<br>Text, Tables<br>and Figures | Definition | Method of<br>Determination |
|---|---|---|
| AUC0-t | Area under the nicotine concentration-time curve from time 0 (defined as the start of product use) to 180 minutes (or the last quantifiable concentration during the interval) | Calculated using the<br>Linear Trapezoidal with<br>Linear Interpolation<br>Method |
| Cmax | Maximum measured plasma concentration over the duration of the measurement interval | Taken directly from bioanalytical data |
| Tmax | Time to reach the maximum measured plasma concentration over the duration of the measurement interval. If the maximum value occurs at more than one time point, Tmax is defined as the first time point with this value. | Taken from clinical database as the difference in the time of administration and the time of the blood draw which is associated with the Cmax. |

Pharmacokinetic parameters will not be calculated for subjects with less than 3 consecutive post-product use time points with quantifiable concentrations. Subjects for whom there are insufficient data to calculate the PK parameters will be included in the concentration tables only and excluded from the descriptive statistics.

Plasma concentrations below the limit of quantitation will be set to one-half of the lower limit of quantitation for the calculation of descriptive statistics of unadjusted plasma nicotine concentrations and for the calculation of baseline-adjusted nicotine concentrations.

Baseline (pre-product use) adjustments will be performed for calculation of PK parameters. The values used for all pre-product use adjustments is the plasma nicotine concentration value obtained before the first product use on each study day.

Baseline-adjustment method: For each PK profile, the pre-product administration nicotine concentration value for each subject will be subtracted from each nicotine

concentration obtained after test product administration on that day using the following equation:

$$C_t = C_{t \; uncorrected} - [C_0 \cdot e^{\text{-Kel} \cdot \; t1}]$$

Where:

 $C_t$  = Corrected concentration.

 $C_{t \text{ uncorrected}}$  = the uncorrected concentration.

 $C_0$  = the pre-product administration concentration.

$$Kel = \frac{\ln(2)}{t\frac{1}{2}}$$

Where t½ is 120 minutes for all subjects (estimated nicotine half-life)

t = actual sampling time since product administration.

t1 = actual sampling time since pre-product administration sampling.

After correction for pre-product administration values, some concentrations may be below the lower limit of quantitation and some may be negative values. Negative values will be assigned a value of zero in the analyses and all other values obtained will be reported as is even if these values are BLQ.

#### 6.2.4 PK Data Summarization and Presentation

All nicotine PK concentrations and/or PK parameters descriptive statistics will be generated using SAS® version 9.4.

The plasma concentrations of nicotine will be listed and summarized by product and time point for all subjects in the Outcomes Population. Unadjusted and baseline adjusted plasma concentrations of nicotine will be presented with the same level of precision as received from the bioanalytical laboratory. Summary statistics, including number of observations (n), arithmetic mean (Mean), standard deviation (SD), coefficient of variation (CV%), minimum, median, maximum will be calculated for all nominal concentration time points. Excluded subjects will be included in the concentration listings, but will be excluded from the summary statistics and noted as such in the tables. All BLQ values will be presented as "BLQ" in the concentration listings and footnoted accordingly.

Mean and individual concentration-time profiles will be presented on linear and semilog scales. Linear mean plots will be presented with and without SD.

Plasma nicotine PK parameters will be listed and summarized by product (overall and by sex) for all subjects in the Outcomes Population. Pharmacokinetic parameters will be reported to 3 significant figures for individual parameters, with the exception of Tmax, which will be presented with 2 decimal places. Summary statistics (n, arithmetic mean, geometric mean, SD, CV%, geometric CV% (Geom CV%), minimum, median, maximum), will be calculated for plasma nicotine PK parameters AUC0-t, Cmax, and Tmax. Excluded subjects will be listed in the PK parameter

tables, but will be excluded from the summary statistics and noted as such in the tables.

The level of precision for each concentration and PK parameter statistic will be presented as follows:

- minimum/maximum in same precision as in bioanalytical data and/or parameter output,
- mean/geometric mean/median in one more level of precision than minimum/maximum,
- SD in one more level of precision than mean/median,
- n will be presented as an integer, and
- CV% and Geom CV% will be presented to the nearest tenth.

Statistical analyses will be performed using SAS and are described in <u>Section 6.7</u>.

#### 6.3 Biomarkers of Exposure and Potential Harm

# **6.3.1** Biomarker Sample Collection

### **Blood Biomarker Sample Collection**

Blood samples for COHb (2 x 4 mL) in whole blood, sICAM in plasma (1 x 4 mL), WBCs (1 x 4 mL) in whole blood, and HDL-C in serum (1 x 3.5 mL), and MCP-1 in serum (1 x 3.5 mL) will be collected on Days -1, 9, and 14. Samples for COHb will be collected in the afternoon and samples for the other biomarkers will be collected following a fast of at least 8 hours.

#### **Urine Biomarker Sample Collection**

24-hour urine collections for biomarker measurements (NNAL, 3-HPMA, S-PMA, NNN, CEMA, HEMA, HMPMA, MHBMA, 1-OHP, (o-tol, 3-OH B[a]P, 1-AN, 2-AN, nicotine equivalents, 8-epi-prostaglandin  $F_{2\alpha}$ , and 11-dehydrothromboxane  $B_2$ ) will take place on Day -2 to -1, Day 8 to 9, and Day 13-14. Each 24-hour urine collection will begin at the start of overnight abstinence.

Subjects will be instructed to attempt to void prior to the beginning and at the end of each interval. All urine must be collected during the entire 24-hour interval. The start and stop time of each 24-hour interval and the total weight of the collection will be documented. The weight of the 24-hour urine collection containers will be documented prior to the collection (tare weight) and following completion of the collection.

Collections for each subject will be pooled into one labeled container throughout the interval and the total weight (g) will be recorded at the end of the 24-hour interval. Any missed voids will be documented, including the reason for missing.

#### 6.3.2 Biomarker Calculations

#### **Calculation of Urine Nicotine Equivalents**

Nicotine equivalents will be calculated as the molar sum of nicotine and 5 major nicotine metabolites. Values of individual components reported as below the limit of quantitation (BLQ) will be set to one-half of the limit of quantitation in the calculation below. Missing urine data will not be imputed.

```
Nicotine equivalents (\mu g/mL) = (nicotine [ng/mL]/162.23 [mg/mmol] + nicotine-gluc (ng/mL)/338.36 [mg/mmol] + cotinine [ng/mL]/176.22 [mg/mmol] + cotinine-gluc [ng/mL]/352.34 [mg/mmol] + trans-3'-hydroxycotinine [ng/mL]/192.22 [mg/mmol] + trans-3'-hydroxycotinine-gluc [ng/mL]/368.34 [mg/mmol]) x 162.23 (mg/mmol) x 1 \mu g/1000 ng
```

#### **Calculation of Total Mass Excreted**

Urine biomarker concentrations will be converted into biomarker quantities excreted in 24 hours by multiplying the measured concentration by the total weight (i.e., 1 kilogram = 1 liter) of urine produced by the subject during the 24-hour period.

#### **Creatinine Adjustments**

Urine creatinine will be measured and used to adjust the values of the primary and secondary urine BoPH and BoE as follows.

```
Biomarker = \underline{\text{Biomarker (units) x 100}}
(unit/g creatinine) = \underline{\text{creatinine (mg/dL)}}
```

#### 6.3.3 Biomarker Data Summarization

Biomarker concentrations reported as below the limit of quantitation will be reported as "BLQ" in the listings and set to one-half of the limit of quantitation for summarization and statistical analysis.

The following variables will be determined and summarized for each urine biomarker.

- Measured concentration
- Total biomarker mass excreted per 24 hours
- Creatinine-adjusted excretion level

Absolute and percent change-from-baseline will be determined for the mass excreted and creatinine-adjusted values. The total urine biomarker mass excreted per 24 hours change-from-baseline value will be used in the statistical analysis.

Data will be listed by subject, sequence, and study day and summarized by study day (Day -1 and Day 9) in Part 1, by study day (Day -1 and Day 14) in Part 2 for Arm I only, and by study arm and study day (Day 9 and Day 14) in Part 2. All summaries will be presented overall and by sex. Absolute and percent change-from-baseline values will also be listed and summarized.

Descriptive statistics (number of observations, mean, median, standard deviation, standard error of the mean, CV%, minimum, and maximum) will be presented using the level of precision details in section 6.1.2. Figures will be used to display the data graphically as applicable. All data summarizations and figures will be generated using the Outcomes Population. Data summarizations and statistical analyses will be performed using SAS procedures. Statistical analyses are described in <u>Section 6.7</u>.

# 6.4 Topography (Part 1 only)

#### 6.4.1 Data Collection

Puff topography will be performed in a subset of 16 subjects (2 subjects from each sequence in Part 1). Subjects will engage in a 1-hour *ad libitum* product use with their usual brand combustible cigarette (Day -1) or the assigned study product (Days 1 and 8), using the topography device (SPA-M). The topography session should start at least 4 hours after the start of the *ad libitum* product use of that day.

#### 6.4.2 Data Summarization

The following topography parameters will be assessed:

- Total Puff count
- Average Puff Duration
- Total Puff Duration
- Average Puff volume
- Total Puff Volume
- Average Peak flow rate
- Average flow rate
- Average Inter-puff interval

Topography parameters will be listed by subject and summarized by study day, overall and by sex. Other summaries by usual brand cigarette flavor (non-menthol or menthol), age, number of years smoking, or CPD may be done if the data permit.

Correlation analyses may be performed to determine the potential relationship between puff topography parameters and pod weight change.

#### 6.5 Physiologic Assessments

#### 6.5.1 Data Collection

On Days -1, 9, and 14, BP and HR will be measured within 2 hours prior to and at every hour after the start of *ad libitum* product use, and at 0, 3, and at least 30 minutes prior to the start of product use on the next day, to generate 24-hour profiles.

Spirometry assessments will be done on Days -1, 9, and 14.

#### 6.5.2 Data Summarization

#### BP and HR

The following parameters will be calculated from the change-from-baseline BP and HR profiles for myblu<sup>TM</sup> exclusive use Arm I:

AUEC0-24 The area under the change from baseline versus time curve from

time 0 to 24 hours, calculated using the linear trapezoidal method with

linear interpolation using nominal sample times.

Emax The maximum change from baseline.

TEmax Time of the Emax. If the maximum value occurs at more than one time

point, TEmax will be defined as the first time point with this value.

Change from baseline will be calculated by subtracting the time-matched post-baseline values from Day 9 and Day 14 from the baseline (Day -1) using nominal sample times. Original data, change from baseline data, and change from baseline parameters will be listed by subject and study day and summarized by study day. Parameters will be summarized by sex and overall.

#### Spirometry

The following pre- and post-bronchodilator lung function variables will be listed by subject and study arm (as applicable):

- Measured and percent of predicted FEV1
- Measured and percent of predicted FVC
- Measured and percent of predicted FEV1:FVC ratio
- Measured and percent of predicted FEF25-75%

The following pre- and post-bronchodilator lung function variables as well as change from baseline (Day -1) pre values and post-pre for each variable will be listed by subject and summarized by study day, for subjects in *my*blu<sup>TM</sup> exclusive use arm (Arm I) using descriptive statistics:

- percent of predicted FEV1
- percent of predicted FVC
- Percent of predicted FEV1:FVC ratio
- Percent of predicted FEF25-75%

Descriptive statistics (number of observations, mean, median, standard deviation, standard error of the mean, CV%, minimum, and maximum) will be used for summarizations. Summaries for the change variables will be by sex and overall.

Figures may be used to display the data graphically, as applicable. All data summarizations including figures will be generated using the Outcomes population. Data summarizations and statistical analyses will be performed using SAS procedures. Statistical analyses are described in <u>Section 6.7</u>.

# 6.6 Subjective Measures

The Urge to Smoke (VAS), Product Liking (VAS), PES (7-point scale), Future Intent to Use (VAS), QSU-Brief, MTWS-R, and PSCDI/PSECDI questionnaires will be completed using a computerized tablet device.

#### 6.6.1 Data Collection

#### Days 2, 4, 6, and 8

Urge to smoke (UTS) will be assessed using a 100 mm VAS approximately 10 minutes prior to the start of the controlled product use session and within approximately 30 seconds prior to the scheduled blood draws at 5, 10, 15, 30, 60, and 120 minutes following the start of the controlled product use session.

PES, Product Liking, and Future Intent to Use questionnaires will be administered following the completion of the controlled product use session.

UTS, PES, Product Liking, and Future Intent to Use questionnaires will be administered at least 6 hours following the start of the *ad libitum* product use session.

#### Days 9 and 14

The Penn State [Electronic] Cigarette Dependence Index (PSCDI/PSECDI) questionnaires, the Minnesota Tobacco Withdrawal Scale-Revised (MTWS-R), and the Questionnaire on Smoking Urges-Brief (QSU-Brief) will be administered at least 6 hours after the start of the *ad libitum* product use session.

#### 6.6.2 Data Summarization

# Days 2, 4, 6, and 8 of Part 1

The following parameters and subscales will be calculated and summarized. UTS parameters will be calculated from urge to smoke assessments taken during the controlled product use sessions using Phoenix WinNonlin Version 7.0 or higher (model 202). For questionnaires without summary parameters (Product Liking Questionnaire, Future Intent to Use Questionnaire, and UTS after *ad libitum* session), each item on the subjective measures questionnaires will be summarized.

- UTS parameters calculated from the reduction from baseline (VASpreuse VAS postuse) vs time profiles:
  - Emax\_R The maximum reduction from baseline VAS score.
  - o TEmax Time of the Emax\_R. If the maximum value occurred at more than one time point, TEmax will be defined as the first time point with this value.
  - AUEC0-120\_R The area under the reduction from baseline "Urge to Smoke" VAS score versus time curve from 0 to 120 minutes, calculated using the linear trapezoidal method with linear interpolation using actual sample times.
- PES subscales (controlled and ad libitum product use sessions):
  - o Satisfaction average of items 1, 2, 3, and 12
  - o Psychological reward average of items 4 through 8
  - o Aversion average of items 9, 10, 16, and 18
  - o Relief average of items 11, 13, 14, 15, and reversed for item 20
  - o Items 17, 19, 21 will be summarized as individual item scores.

UTS, Product Liking, PES, and Future Intent to Use responses will be listed by subject, product, day, and product use session (and time point as applicable). UTS parameters, PES subscales, and Product Liking and Future Intent to Use responses will be summarized by product (and product use session as applicable). For Future Intent to Use, responses recorded as VAS scores will also be treated as bipolar categorical variables (-50 to <0, 0, >0 to 50) and summarized by study product using frequency count tables. The bipolar score for the Future Intent to Use questionnaire is calculated by subtracting 50 from the original VAS score. The bipolar scores will also be treated as continuous variables and summarized using descriptive statistics.

#### Days 9 and 14

The following total scores and factor scores will be calculated and summarized. Total scores, factor scores, and responses to individual questionnaire items will be listed.

PSCDI/PSECDI total score

- MTWS-R total score
- QSU-brief factor scores:
  - Factor 1 (anticipation of pleasure from smoking) average of items 1, 3, 6, 7, and 10
  - o Factor 2 (anticipation of relief of nicotine withdrawal) average of items 2, 4, 5, 8, and 9

(QSU-Brief), the Minnesota Tobacco Withdrawal Scale-Revised (MTWS-R), and the Penn State [Electronic] Cigarette Dependence Index (PSCDI/PSECDI)

QSU-Brief, MTWS-R, PSCDI/PSECDI responses and factor/total scores will be listed by subject and day and study arm. Factor and total scores will be summarized by study day and study arm.

Descriptive statistics (number of observations, mean, median, standard deviation, standard error of the mean, CV%, minimum, and maximum) will be used for all questionnaire summarizations, and summaries will be presented overall and by sex.

Figures may be used to display the data graphically, as applicable. All data summarizations and figures will be generated using the Outcomes Population. Data summarizations and statistical analyses will be performed using SAS procedures. Statistical analyses are described in Section 6.7.

#### 6.7 Statistical Analyses

#### a. Pharmacokinetics (primary objective 1)

A linear mixed model for analysis of variance will be performed on the log-transformed PK parameters Cmax and AUC following the first product use session on each of Days 2, 4, 6, and 8. The two blocks of subjects (ABCD, EFGH) will be modeled separately. Each model will include sequence, study product, and day as fixed effects and subject-nested-within-sequence as a random effect. Sequence will be tested using subject-nested-within-sequence as the error term. Geometric least-squares means (LSM) and 95% confidence intervals (CIs) will be provided for the PK parameters of Cmax and AUC by study product. Geometric LSM ratio, 95% CIs of geometric LSM ratio, and p-values will be provided for the study product comparisons in Cmax and AUC. The comparisons of interest will include each of the study products compared to each other.

#### ABCD Block:

Product A versus Product B

Product A versus Product C

Product A versus Product D

Product B versus Product C

Product B versus Product D

Product C versus Product D

EFGH Block:

Product E versus Product F

Product E versus Product G

Product E versus Product H

Product F versus Product G

Product F versus Product H

Product G versus Product H

The above statistical analyses will be performed using the following SAS codes.

Proc MIXED data=<>;

Class subject sequence product day;

Model LN dependent variable = sequence product day /DDFM=KR;

Random Subject(sequence);

LSMeans product/pdiff CL alpha=0.05;

Run;

Non-parametric analysis (Wilcoxon signed rank test) will be performed for the comparisons of  $T_{max}$  between each product.

# b. Primary and Secondary Biomarkers Day 9 for myblu<sup>TM</sup> (primary objective 2 and secondary objectives 2 and 5)

Comparisons of the Day 9 and Day -1 primary and secondary BoE and BoPH values will be made using a linear mixed model analysis of variance (ANOVA).

The ANOVA model will include day as a fixed effect and subject as a random effect. Least square means (LSMs) will be provided for each day. LSM differences, 95% confidence intervals of LSM differences, and p-values will be provided for the day comparisons. The above statistical analyses will be performed using the following SAS codes.

Proc MIXED data=<>;

Class subject day;

Model dependent variable = day/DDFM=KR;

Random subject;

LSMeans day/pdiff CL alpha=0.05;

Run;

LSM differences, 95% confidence intervals of LSM differences, and p-values will be provided for the day comparisons.

# c. <u>Primary and Secondary Biomarkers Day 14 for myblu<sup>TM</sup> (secondary objectives 1, 2, and 5)</u>

Comparisons of the Day 14 and Day -1 primary and secondary BoE and BoPH values in exclusive *my*blu<sup>TM</sup> arm will be made using the same linear mixed model ANOVA as for Day 9 above.

# d. <u>Change-from-baseline differences (Day 14 – Day 9) in the primary and secondary tobacco-related BoE and BoPH between study arms (secondary objective 4)</u>

Comparisons of the change-from-baseline differences in the primary and secondary BoE and BoPH values among the study arms will be made using a linear mixed model analysis of variance (ANOVA).

The ANOVA model will include arm as fixed effects and subject as a random effect. Least square means (LSMs) will be provided for each arm. LSM differences, 95% confidence intervals of LSM differences, and p-values will be provided for the day comparisons. The above statistical analyses will be performed using the following SAS codes.

```
Proc MIXED data=<>;
Class arm;
Model dependent variable = arm/DDFM=KR;
LSMeans arm/pdiff CL alpha=0.05;
Run;
```

The comparisons of interest are:

*my*blu<sup>TM</sup> vs Combustible Cigarette *my*blu<sup>TM</sup> vs Dual Use
Dual Use vs Combustible Cigarette

#### e. Other Secondary Objectives:

Changes in the primary and secondary tobacco-related BoE in the exclusive e-cigarette use, exclusive combustible cigarette use and dual use groups at Day 14 (Secondary objective 3) will be summarized descriptively.

Urge to smoke parameters from the controlled product use session will be analyzed using analysis a. Other questionnaire information will be summarized descriptively (Secondary objective 6).

Puff topography and product use (secondary objectives 7 and 9) will be summarized descriptively.

Analyses b and c will be used to assess in physiologic endpoints following 9-day and 14-day use periods of myblu<sup>TM</sup> e-cigarettes (secondary objective 8):

• change from baseline blood pressure [BP] and heart rate [HR] parameters

- change from baseline pre-bronchodilator values for percent of predicted parameters
- change from baseline in post-pre bronchodilator values for percent of predicted parameters

#### 7. SAFETY

All case report form (CRF) data will be listed by subject and chronologically by assessment time points. This will include rechecks, unscheduled assessments, and early termination.

Applicable continuous variables will be summarized using n, arithmetic mean, SD, minimum, median, and maximum.

The level of precision will be presented as follows: minimum/maximum in the same precision as in the database, mean/median in one more precision level than minimum/maximum, SD in one more precision level than mean/median, and n will be presented as an integer.

Where individual data points are missing because of dropouts or other reasons, the data will be summarized based on reduced denominators.

# 7.1 Subject Discontinuation

Subjects will be summarized by number of subjects enrolled, randomized, completed, and discontinued the study with discontinuation reasons by randomized product sequence (Part 1) or study arm (Part 2) and overall for each study part.

#### 7.2 Demographics

Descriptive statistics will be calculated for continuous variables (age, weight, height, and body mass index) by randomized product sequence (Part 1) or study arm (Part 2) and overall for each study part.

Frequency counts will be provided for categorical variables (race, ethnicity, and sex, and other characteristics) for each randomized product sequence (Part 1) or study arm (Part 2) and overall for each study part.

# 7.3 Smoking History

Descriptive statistics will be calculated for continuous variables (cigarettes smoked per day [CPD] and number of years smoked) by randomized randomized product sequence (Part 1) or study arm (Part 2) and overall for each study part.

Frequency counts will be provided for subject's usual brand for each randomized product sequence (Part 1) or study arm (Part 2) and overall for each study part.

#### 7.4 Adverse Events

All adverse events (AEs) occurring during this clinical trial will be coded using the Medical Dictionary for Regulatory Activities (MedDRA®), Version 22.1.

All AEs captured in the database will be listed in by-subject data listings including verbatim term, coded term, product, severity, relationship to study product (Part 1) or study arm (Part 2), and action; however, only product use-emergent AEs (PUEAEs) will be summarized

A PUEAE is defined as an AE that is starting or worsening at the time of or after the first randomized study product use. Each PUEAE will be attributed to a study product (Part 1) or study arm (Part 2) based on the onset date and time of the AE.

If the onset time of an AE is missing and the onset date is the same as the first study product use date, then the AE will be considered product use emergent in the study product. If onset time of an AE is missing and the onset date does not fall on a study product use date, then the AE will be considered product use emergent for the last study product administered. If the onset date of an AE is missing, then the AE will be considered product use emergent, unless the onset date is known to have occurred within or between specific product use days.

PUEAEs will be tabulated by System Organ Class (SOC) and Preferred Term. Summary tables will include number of subjects reporting the AE and as percent of number of subjects who used study product by product. The number of AEs will be tabulated in a similar manner. Tables which tabulate the number of PUEAEs by severity and relationship to study product will also be included.

In addition, adverse events occurred during baseline period on Day -2 and day -1 will be summarized separately.

Serious adverse events (SAEs), if present, will also be listed. Applicable narratives will be included in the CSR.

# 7.5 Clinical Laboratory Tests (Serum Chemistry, Hematology, and Urinalysis)

Serum Chemistry, hematology, and urinalysis samples will be collected at screening, check-in (Day -2), and prior to discharge or prior to early termination from the study.

Descriptive statistics will be reported for numeric clinical data and change from baseline for each assessment timepoint. Rechecked values prior to randomization will be used in calculating summary statistics. Baseline is the last non-missing value including recheck and unscheduled event before randomization (usually on Day -2 Check-in). Normal ranges will be listed.

Out of normal range and clinically significant laboratory values will be listed by subject. Results that are indicated as CS by the PI will be listed in the table.

A urine cotinine test will be completed at Screening.

Urine drug tests and alcohol breath tests will be completed at Screening and Check-in (Day -2).

For females, serum pregnancy tests will be completed at Screening and urine pregnancy tests will be completed at Check-in (Day -2).

Results for these tests will be listed as "Negative" or "Positive."

# 7.6 Vital Signs

Vital signs (pulse, blood pressure, respiration rate, and body temperature) will be measured at Screening and Check-in (Day -2). BP and HR will also be measured within 2 hours prior to and at every hour after the start of *ad libitum* product use and throughout the period of *ad libitum* product use. Following completion of *ad libitum* product use on that day, BP and HR will be measured at 00:00, 03:00, and at least 30 minutes prior to the start of product use on the next day on Days -1, Day 9, and Day 14 (for Day 14, the last measurement will be collected at approximately 06:00 on Day 15). Respiration rate and body temperature will also be measured prior to the start of the first product use session.

Descriptive statistics will be reported for vital sign measurements by product (Part 1) or study arm (Part 2) and time point. Unscheduled events or rechecks post randomization will not be included in summaries. Similarly early termination results will not be included in summaries.

#### 7.7 Electrocardiogram

A single 12-lead electrocardiogram (ECG) will be recorded at collected at screening, check-in (Day -2), and prior to discharge or prior to early termination from the study.

Descriptive statistics will be reported for ECG parameters by time point. Unscheduled events or rechecks post randomization will not be included in summaries. Similarly early termination results will not be included in summaries.

ECG results will be listed by subject.

#### 7.8 Concomitant Medications

All concomitant medications recorded during the study will be coded with the WHO Drug Dictionary Version 01SEP2019 b3 and listed by subject.

#### 7.9 Physical Examination

Full physical examinations will be performed at Screening and prior to discharge or prior to early termination from the study.

Physical examinations will be listed by subject. Changes in physical examinations (if any) will be described in the text of the final report.

#### 7.10 Exhaled CO

Exhaled CO will be collected at Screening.

Exhaled CO will be listed by subject.

# 7.11 Lung Function (Spirometry)

Subjects will undergo lung function testing at Screening to affirm eligibility (FEV<sub>1</sub>, FEV<sub>1</sub>:FVC ratio) and as a safety endpoint (FEV<sub>1</sub>, FVC, FEV<sub>1</sub>:FVC ratio, and forced expiratory flow (FEF)<sub>25-75%</sub>) at Day -1, Day 9, and Day 14.

Descriptive statistics will be reported for measured and percent of predicted spirometry parameters. Unscheduled events or rechecks post randomization will not be included in summaries. Similarly early termination results will not be included in summaries.

Spirometry results will be listed by subject.

#### 8. SUMMARY OF CHANGES FROM PROTOCOL-PLANNED ANALYSIS

The analyses described in this SAP are aligned with those analyses described in the protocol.

#### 9. SUMMARY TABLES AND FIGURES

Summary tables and figures are numbered following the International Conference on Harmonization (ICH) structure but may be renumbered as appropriate during the compilation of the tables and figures for the CSR. Note that all summary tables and figures will be generated using  $SAS^{@}$  Version 9.4.

# **Section 14 Summary Tables and Figures**

The following is a list of table and figure titles that will be included in Section 14 of the report. Tables and figures may be renumbered as appropriate during the compilation of the report.

#### 14.1 Demographic Data Summary Tables

Table 14.1.1.1 Summary of Disposition - Part 1 (Safety Population)

- Table 14.1.2 Disposition of Subjects Part 1 (Safety Population)
- Table 14.1.3.1 Demographic Summary Part 1 (Safety Population)
- Table 14.1.3.2 Demographic Summary Part 2 (Safety Population)
- Table 14.1.4.1 Smoking History Summary Part 1 (Safety Population)
- Table 14.1.4.2 Smoking History Summary Part 2 (Safety Population)
- Table 14.1.5.1 Summary of Disposition –Part 1 (Outcome Population)
- Table 14.1.5.2 Summary of Disposition –Part 2 (Outcome Population)
- Table 14.1.6.1 Demographic Summary Part 1 (Outcome Population)
- Table 14.1.6.2 Demographic Summary Part 2 (Outcome Population)
- Table 14.1.7.1 Smoking History Summary Part 1 (Outcome Population)
- Table 14.1.7.2 Smoking History Summary Part 2 (Outcome Population)

# 14.2 Study Product Use, Pharmacokinetics, Biomarkers, Physiologic Assessments, Questionnaires, and Topography Data Summary Tables and Figures

#### **14.2.1 Product Use Tables**

| Table 14.2.1.1 | Summary of Pod Weight Changes by Study Product<br>and Study Day Following Controlled Use (Outcomes<br>Population) |
|---|---|
| Table 14.2.1.2 | Summary of Number of Inhalations by Study Product<br>and Study Day Following Controlled Use (Outcomes<br>Population) |
| Table 14.2.1.3 | Summary of Duration of Inhalations by Study Product<br>and Study Day Following Controlled Use (Outcomes<br>Population) |
| Table 14.2.1.4 | Summary of Pod Weight Changes by Study Product<br>Study Day Following Ad Libitum Use (Outcomes<br>Population) |
| Table 14.2.1.5 | Summary of Pod Weight Changes by Study Product<br>and Study Day Following Ad libitum Use on Day 9<br>(Outcomes Population) |
| Table 14.2.1.6 | Summary of Pod Weight Changes and Number of Cigarettes Smoked by Study Arm and Study Day (Outcomes Population) |

#### 14.2.2 Pharmacokinetics Tables

Table 14.2.2.1.1 Unadjusted Plasma Nicotine Concentrations (ng/mL) Following Controlled Use of *my*blu<sup>TM</sup> (freebase), Gold Leaf flavor, 2.4% (Product A) (Outcomes Population)

| 003 myblu ··· E-cigalettes | |
|-----------------------------------|---|
| Clinical Study Report No. CA22736 | |
| = | Ξ |

| Table 14.2.2.1.2 | Unadjusted Plasma Nicotine Concentrations (ng/mL) Following Controlled Use of <i>my</i> blu <sup>TM</sup> (freebase), Polar Mint flavor, 2.4% (Product B) (Outcomes Population) |
|---|---|
| Table 14.2.2.1.3 | Unadjusted Plasma Nicotine Concentrations (ng/mL) Following Controlled Use of <i>my</i> blu <sup>TM</sup> (freebase), Cherry flavor, 2.4% (Product C) (Outcomes Population) |
| Table 14.2.2.1.4 | Unadjusted Plasma Nicotine Concentrations (ng/mL) Following Controlled Use of <i>my</i> blu <sup>TM</sup> (freebase), Vanilla flavor, 2.4% (Product D) (Outcomes Population) |
| Table 14.2.2.1.5 | Unadjusted Plasma Nicotine Concentrations (ng/mL) Following Controlled Use of <i>my</i> blu <sup>TM</sup> (freebase), Gold Leaf flavor, 1.2% (Product E) (Outcomes Population) |
| Table 14.2.2.1.6 | Unadjusted Plasma Nicotine Concentrations (ng/mL) Following Controlled Use of <i>my</i> blu <sup>TM</sup> (freebase), Polar Mint flavor, 1.2% (Product F) (Outcomes Population) |
| Table 14.2.2.1.7 | Unadjusted Plasma Nicotine Concentrations (ng/mL) Following Controlled Use of <i>my</i> blu <sup>TM</sup> (freebase), Menthol flavor, 2.4% (Product G) (Outcomes Population) |
| Table 14.2.2.1.8 | Unadjusted Plasma Nicotine Concentrations (ng/mL) Following Controlled Use of <i>my</i> blu <sup>TM</sup> Intense (nicotine salts), Fresh Mint flavor, 2.4% (Product H) (Outcomes Population) |
| Table 14.2.2.2.1 | Baseline-Adjusted Plasma Nicotine Concentrations (ng/mL) Following Controlled Use of <i>my</i> blu <sup>TM</sup> (freebase), Gold Leaf flavor, 2.4% (Product A) (Outcomes Population) |
| Table 14.2.2.2.2 | Baseline-Adjusted Plasma Nicotine Concentrations (ng/mL) Following Controlled Use of <i>my</i> blu <sup>TM</sup> (freebase), Polar Mint flavor, 2.4% (Product B) (Outcomes Population) |
| Table 14.2.2.2.3 | Baseline-Adjusted Plasma Nicotine Concentrations (ng/mL) Following Controlled Use of <i>my</i> blu <sup>TM</sup> (freebase), Cherry flavor, 2.4% (Product C) (Outcomes Population) |
| Table 14.2.2.2.4 | Baseline-Adjusted Plasma Nicotine Concentrations (ng/mL) Following Controlled Use of <i>my</i> blu <sup>TM</sup> (freebase), Vanilla flavor, 2.4% (Product D) (Outcomes Population) |
| Table 14.2.2.2.5 | Baseline-Adjusted Plasma Nicotine Concentrations (ng/mL) Following Controlled Use of <i>my</i> blu <sup>TM</sup> |

| | (freebase), Gold Leaf flavor, 1.2% (Product E) (Outcomes Population) |
|---|---|
| Table 14.2.2.2.6 | Baseline-Adjusted Plasma Nicotine Concentrations (ng/mL) Following Controlled Use of <i>my</i> blu <sup>TM</sup> (freebase), Polar Mint flavor, 1.2% (Product F) (Outcomes Population) |
| Table 14.2.2.2.7 | Baseline-Adjusted Plasma Nicotine Concentrations (ng/mL) Following Controlled Use of <i>my</i> blu <sup>TM</sup> (freebase), Menthol flavor, 2.4% (Product G) (Outcomes Population) |
| Table 14.2.2.2.8 | Baseline-Adjusted Plasma Nicotine Concentrations (ng/mL) Following Controlled Use of <i>my</i> blu <sup>TM</sup> Intense (nicotine salts), Fresh Mint flavor, 2.4% (Product H) (Outcomes Population) |
| Table 14.2.2.3.1 | Baseline-Adjusted Plasma Nicotine PK Parameters Following Controlled Use of <i>my</i> blu <sup>TM</sup> (freebase), Gold Leaf flavor, 2.4% (Product A) (Outcomes Population) |
| Table 14.2.2.3.2 | Baseline-Adjusted Plasma Nicotine PK Parameters Following Controlled Use of <i>my</i> blu <sup>TM</sup> (freebase), Polar Mint flavor, 2.4% (Product B) (Outcomes Population) |
| Table 14.2.2.3.3 | Baseline-Adjusted Plasma Nicotine PK Parameters Following Controlled Use of <i>my</i> blu <sup>TM</sup> (freebase), Cherry flavor, 2.4% (Product C) (Outcomes Population) |
| Table 14.2.2.3.4 | Baseline-Adjusted Plasma Nicotine PK Parameters Following Controlled Use of <i>my</i> blu <sup>TM</sup> (freebase), Vanilla flavor, 2.4% (Product D) (Outcomes Population) |
| Table 14.2.2.3.5 | Baseline-Adjusted Plasma Nicotine PK Parameters Following Controlled Use of <i>my</i> blu <sup>TM</sup> (freebase), Gold Leaf flavor, 1.2% (Product E) (Outcomes Population) |
| Table 14.2.2.3.6 | Baseline-Adjusted Plasma Nicotine PK Parameters Following Controlled Use of <i>my</i> blu <sup>TM</sup> (freebase), Polar Mint flavor, 1.2% (Product F) (Outcomes Population) |
| Table 14.2.2.3.7 | Baseline-Adjusted Plasma Nicotine PK Parameters Following Controlled Use of <i>my</i> blu <sup>TM</sup> (freebase), Menthol flavor, 2.4% (Product G) (Outcomes Population) |
| Table 14.2.2.3.8 | Baseline-Adjusted Plasma Nicotine PK Parameters Following Controlled Use of <i>my</i> blu <sup>TM</sup> Intense (nicotine salts), Fresh Mint flavor, 2.4% (Product H) (Outcomes Population) |

# Clinical Study Report No. CA22736

| Table 14.2.2.4.1 | Statistical Comparisons of Baseline-Adjusted Plasma Nicotine PK Parameters Among <i>my</i> blu <sup>TM</sup> Products A, B, C, and D Following Controlled Use (Outcomes Population) |
|---|---|
| Table 14.2.2.4.2 | Statistical Comparisons of Baseline-Adjusted Plasma Nicotine PK Parameters Among <i>my</i> blu <sup>TM</sup> Products E, F, G, and H Following Controlled Use (Outcomes Population) |
| Table 14.2.2.4.3 | Nonparametric Statistical Comparisons of Plasma<br>Nicotine PK Parameter Tmax Among <i>my</i> blu <sup>TM</sup><br>Products A, B, C, and D following Controlled Use<br>(Outcomes Population) |
| Table 14.2.2.4.4 | Nonparametric Statistical Comparisons of Plasma<br>Nicotine PK Parameter Tmax Among <i>my</i> blu <sup>TM</sup><br>Products A, B, C, and D following Controlled Use<br>(Outcomes Population) |

# 14.2.3 Biomarker Tables

# 14.2.3.1 Part 1

| Table 14.2.3.1.1 | Summary of Blood COHb (% saturation) by Study Day |
|---|---|
| | in Part 1: 9-Day Switch to Exclusive <i>my</i> blu <sup>™</sup> Use |
| | (Outcomes Population) |

Table 14.2.3.1.2 through 14.2.3.1.21 (one per biomarker) will be generated similarly:

| Sillillally. | |
|-------------------|----------------------------|
| Table 14.2.3.1.2 | Urine NNAL |
| Table 14.2.3.1.3 | Urine 3-HPMA |
| Table 14.2.3.1.4 | Urine S-PMA |
| Table 14.2.3.1.5 | Urine NNN |
| Table 14.2.3.1.6 | Urine CEMA |
| Table 14.2.3.1.7 | Urine HEMA |
| Table 14.2.3.1.8 | Urine 3-HMPMA |
| Table 14.2.3.1.9 | Urine MHBMA |
| Table 14.2.3.1.10 | Urine 1-OHP |
| Table 14.2.3.1.11 | Urine o-tol |
| Table 14.2.3.1.12 | Urine 3-OH B[a]P |
| Table 14.2.3.1.13 | Urine 1-AN |
| Table 14.2.3.1.14 | Urine 2-AN |
| Table 14.2.3.1.15 | Urine Nicotine Equivalents |
| Table 14.2.3.1.16 | Plasma sICAM (ng/mL) |
| Table 14.2.3.1.17 | WBCs $(x10^3/\mu L)$ |

# Clinical Study Report No. CA22736

| Serum HDL-C (mg/dL) |
|--------------------------------|
| Serum MCP-1 (units) |
| Urine 8-epi-prostaglandin F2α |
| Urine 11-dehydrothromboxane B2 |

Note: units are in the table header for urine biomarkers

Table 14.2.3.1.22 Statistical Comparisons of BoE and BoPH Between Study Days in Part 1: 9-Day Switch to Exclusive *my*blu<sup>TM</sup> Use (Outcomes Population)

# **14.2.3.2** Part **2** by Study Day

Table 14.2.3.2.1 Summary of Blood COHb (% Saturation) by Study Day in Part 2: Continue Exclusive *my*blu<sup>TM</sup> Use (Outcomes Population)

Table 14.2.3.2.2 through 14.2.3.2.21 (one per biomarker) will be generated similarly:

| Table 14.2.3.2.2 | Urine NNAL |
|-------------------|---------------------------------------|
| Table 14.2.3.2.3 | Urine 3-HPMA |
| Table 14.2.3.2.4 | Urine S-PMA |
| Table 14.2.3.2.5 | Urine NNN |
| Table 14.2.3.2.6 | Urine CEMA |
| Table 14.2.3.2.7 | Urine HEMA |
| Table 14.2.3.2.8 | Urine 3-HMPMA |
| Table 14.2.3.2.9 | Urine MHBMA |
| Table 14.2.3.2.10 | Urine 1-OHP |
| Table 14.2.3.2.11 | Urine o-tol |
| Table 14.2.3.2.12 | Urine 3-OH B[a]P |
| Table 14.2.3.2.13 | Urine 1-AN |
| Table 14.2.3.2.14 | Urine 2-AN |
| Table 14.2.3.2.15 | Urine Nicotine Equivalents |
| Table 14.2.3.2.16 | Plasma sICAM (ng/mL) |
| Table 14.2.3.2.17 | WBCs $(x10^3/\mu L)$ |
| Table 14.2.3.2.18 | Serum HDL-C (mg/dL) |
| Table 14.2.3.2.19 | Serum MCP-1 (units) |
| Table 14.2.3.2.20 | Urine 8-epi-prostaglandin F2 $\alpha$ |
| Table 14.2.3.2.21 | Urine 11-dehydrothromboxane B2 |

Note: units are in the table header for urine biomarkers
Table 14.2.3.2.22 Statistical Comparisons of BoE and BoPH Between

Study Days in Part 2: Continue Exclusive myblu<sup>TM</sup> Use

(Outcomes Population)

#### 14.2.3.3 Part 2 by Study Arm

Table 14.2.3.3.1 Summary of Blood COHb (% Saturation) by Study Arm in Part 2 (Outcomes Population)

Tables 14.2.3.3.2 through 14.2.3.3.21 will be generated for each biomarker similarly:

| Table 14.2.3.3.2 | Urine NNAL |
|-------------------|--------------------------------|
| Table 14.2.3.3.3 | Urine 3-HPMA |
| Table 14.2.3.3.4 | Urine S-PMA |
| Table 14.2.3.3.5 | Urine NNN |
| Table 14.2.3.3.6 | Urine CEMA |
| Table 14.2.3.3.7 | Urine HEMA |
| Table 14.2.3.3.8 | Urine 3-HMPMA |
| Table 14.2.3.3.9 | Urine MHBMA |
| Table 14.2.3.3.10 | Urine 1-OHP |
| Table 14.2.3.3.11 | Urine o-tol |
| Table 14.2.3.3.12 | Urine 3-OH B[a]P |
| Table 14.2.3.3.13 | Urine 1-AN |
| Table 14.2.3.3.14 | Urine 2-AN |
| Table 14.2.3.3.15 | Urine Nicotine Equivalents |
| Table 14.2.3.3.16 | Plasma sICAM (ng/mL) |
| Table 14.2.3.3.17 | WBCs $(x103/\mu L)$ |
| Table 14.2.3.3.18 | Serum HDL-C (mg/dL) |
| Table 14.2.3.3.19 | Serum MCP-1 (units) |
| Table 14.2.3.3.20 | Urine 8-epi-prostaglandin F2α |
| Table 14.2.3.3.21 | Urine 11-dehydrothromboxane B2 |

Note: units are in the table header for urine biomarkers

Table 14.2.3.3.22 Statistical Comparisons of BoE and BoPH Differences From Baseline Among *my*blu<sup>TM</sup>, Combustible Cigarette, and Dual Use Arms in Part 2 (Outcomes Population)

Clinical Study Report No. CA22736

### 14.2.4 Physiologic Assessments Tables

| 14.2.4 I hysiologic Assessments Tables | |
|---|---|
| 14.2.4.1 SPB, DPB, and HR | |
| Table 14.2.4.1.1 | Summary of Systolic Blood Pressure (mm Hg) by Time Point in Exclusive <i>my</i> blu <sup>TM</sup> Use (Arm I) (Outcomes Population) |
| Table 14.2.4.1.2 | Summary of Systolic Blood Pressure Change from Baseline (mm Hg) by Time Point in Exclusive <i>my</i> blu <sup>TM</sup> Use (Arm I) (Outcomes Population) |
| Table 14.2.4.1.3 | Summary of Systolic Blood Pressure Change from Baseline Parameters in Exclusive <i>my</i> blu <sup>TM</sup> Use (Arm I) (Outcomes Population) |
| Table 14.2.4.1.4 | Summary of Diastolic Blood Pressure (mm Hg) by Time Point in Exclusive <i>my</i> blu <sup>TM</sup> Use (Arm I) (Outcomes Population) |
| Table 14.2.4.1.5 | Summary of Diastolic Blood Pressure Change from Baseline (mm Hg) by Time Point in Exclusive myblu <sup>TM</sup> Use (Arm I) (Outcomes Population) |
| Table 14.2.4.1.6 | Summary of Systolic Blood Pressure Change from Baseline Parameters in Exclusive <i>my</i> blu <sup>TM</sup> Use (Arm I) (Outcomes Population) |
| Table 14.2.4.1.7 | Summary of Heart Rate (bpm) by Time Point in Exclusive <i>my</i> blu <sup>TM</sup> Use (Arm I) (Outcomes Population) |
| Table 14.2.4.1.8 | Summary of Heart Rate (bpm) Change from Baseline by Time Point in Exclusive <i>my</i> blu <sup>TM</sup> Use (Arm I) (Outcomes Population) |
| Table 14.2.4.1.9 | Summary of Heart Rate Change from Baseline Parameters in Exclusive <i>my</i> blu <sup>TM</sup> Use (Arm I) (Outcomes Population) |
| Table 14.2.4.1.10 | Statistical Comparisons of Change From Baseline<br>Systolic Blood Pressure, Diastolic Blood Pressure, and<br>Heart Rate Heart Rate Parameters in Exclusive <i>my</i> blu <sup>TM</sup><br>Use (Arm I) |
| <b>14.2.4.2 Spirometry</b> | |
| Table 14.2.4.2.1 | Summary of Lung Function Variables by Time Point in Exclusive <i>my</i> blu <sup>TM</sup> Use (Arm I) (Outcomes Population) |
| Table 14.2.4.2.2 | Summary of Lung Function Variables Changes by Time Point in Exclusive <i>my</i> blu <sup>TM</sup> Use (Arm I) (Outcomes Population) |
| Table 14.2.4.2.3 | Statistical Comparisons of Change From Baseline<br>Systolic Blood Pressure, Diastolic Blood Pressure, and<br>Heart Rate Heart Rate Parameters in Exclusive <i>my</i> blu <sup>TM</sup><br>Use (Arm I) |

| 14.2.5 | Urge to Smoke Tables |
|---|---|
| Table 14.2.5.1.1 | Urge to Smoke VAS Score Following Controlled and Ad libitum use of <i>my</i> blu <sup>™</sup> (freebase), Gold Leaf flavor, 2.4% (Product A) (Outcomes Population) |
| Table 14.2.5.1.2 | Urge to Smoke VAS Score Following Controlled and Ad Libitum use of <i>my</i> blu <sup>TM</sup> (freebase), Polar Mint flavor, 2.4% (Product B) (Outcomes Population) |
| Table 14.2.5.1.3 | Urge to Smoke VAS Score Following Controlled and Ad Libitum use of <i>my</i> blu <sup>TM</sup> (freebace), Charry flavor, 2.4% (Product C) (Outcomes Population) |
| Table 14.2.5.1.4 | Urge to Smoke VAS Score Following Controlled and Ad Libitum use of <i>my</i> blu <sup>TM</sup> (freebase), Vanilla flavor, 2.4% (Product D) (Outcomes Population) |
| Table 14.2.5.1.5 | Urge to Smoke VAS Score Following Controlled and Ad Libitum use of <i>my</i> blu <sup>TM</sup> (freebase), Gold Leaf flavor, 1.2% (Product E) (Outcomes Population) |
| Table 14.2.5.1.6 | Urge to Smoke VAS Score Following Controlled and Ad Libitum use of <i>my</i> blu <sup>TM</sup> (freebase), Polar Mint flavor, 1.2% (Product F) (Outcomes Population) |
| Table 14.2.5.1.7 | Urge to Smoke VAS Score Following Controlled and Ad Libitum use of <i>my</i> blu <sup>TM</sup> (freebase), Menthol flavor, 2.4% (Product G) (Outcomes Population) |
| Table 14.2.5.1.8 | Urge to Smoke VAS Score Following Controlled and Ad Libitum use of <i>my</i> blu <sup>TM</sup> Intense (nicotine salts), Fresh Mint flavor, 2.4% (Product H) (Outcomes Population) |
| Table 14.2.5.2.1 | Urge to Smoke VAS Parameters Following Controlled and Ad libitum use of $my$ blu <sup>TM</sup> (freebase), Gold Leaf flavor, 2.4% (Product A) (Outcomes Population) |
| Table 14.2.5.2.2 | Urge to Smoke VAS Parameters Following Controlled and Ad Libitum use of <i>my</i> blu <sup>TM</sup> (freebase), Polar Mint flavor, 2.4% (Product B) (Outcomes Population) |
| Table 14.2.5.2.3 | Urge to Smoke VAS Parameters Following Controlled and Ad Libitum use of <i>my</i> blu <sup>TM</sup> (freebase), Cherry flavor, 2.4% (Product C) (Outcomes Population) |
| Table 14.2.5.2.4 | Urge to Smoke VAS Parameters Following Controlled and Ad Libitum use of <i>my</i> blu <sup>TM</sup> (freebase), Vanilla flavor, 2.4% (Product D) (Outcomes Population) |
| Table 14.2.5.2.5 | Urge to Smoke VAS Parameters Following Controlled and Ad Libitum use of <i>my</i> blu <sup>TM</sup> (freebase), Gold Leaf flavor, 1.2% (Product E) (Outcomes Population) |

| O1:: - 1 | 04-1 | D 4 M - | C 4 22726 |
|----------|-------|-----------|-----------|
| Ciinicai | Stuav | Keport No | . CA22736 |

| Table 14.2.5.2.6 | Urge to Smoke VAS Parameters Following Controlled and Ad Libitum use of <i>my</i> blu <sup>TM</sup> (freebase), Polar Mint flavor, 1.2% (Product F) (Outcomes Population) |
|---|---|
| Table 14.2.5.2.7 | Urge to Smoke VAS Parameters Following Controlled and Ad Libitum use of <i>my</i> blu <sup>TM</sup> (freebase), Menthol flavor, 2.4% (Product G) (Outcomes Population) |
| Table 14.2.5.2.8 | Urge to Smoke VAS Parameters Following Controlled and Ad Libitum use of <i>my</i> blu <sup>™</sup> Intense (nicotine salts), Fresh Mint flavor, 2.4% (Product H) (Outcomes Population) |
| Table 14.2.5.3.1 | Statistical Comparisons of Urge to Smoke Parameters Among <i>my</i> blu <sup>™</sup> Products A, B, C, and D Following Controlled Use (Outcomes Population) |
| Table 14.2.5.3.2 | Statistical Comparisons of Urge to Smoke Parameters Among <i>my</i> blu <sup>TM</sup> Products E, F, G, and H Following Controlled Use (Outcomes Population) |

#### 14.2.6 Questionnaire Tables

#### **14.2.6.1 PES Subscales**

Table 14.2.6.1

| | Controlled Product Use Session (Outcomes Population) |
|---|---|
| Table 14.2.6.2 | Summary of PES Subscales by Study Product for Ad<br>Libitum Product Use Session (Outcomes Population) |
| 14.2.6.2 Product Liking VAS Score | |
| Table 14.2.6.2.1 | Summary of Product Liking VAS Score by Study<br>Product for Controlled Product Use Session (Outcomes<br>Population) |
| Table 14.2.6.2.2 | Summary of Product Liking VAS Score by Study<br>Product for Ad Libitum Product Use Session<br>(Outcomes Population) |
| 14.2.6.3 Future Intent to Use VAS Score | |

Summary of PES Subscales by Study Product for

| Table 14.2.6.3.1 | Frequency of Responses to Future Intent to Use in Each<br>Category by Study Product for Controlled Product Use<br>Session (Outcomes Population) |
|---|---|
| Table 14.2.6.3.2 | Frequency of Responses to Future Intent to Use in Each<br>Category by Study Product for Ad Libitum Product Use<br>Session (Outcomes Population) |
| Table 14.2.6.3.3 | Summary of Future Intent to Use VAS Score in Each<br>Category by Study Product for Controlled Product Use<br>Session (Outcomes Population) |

| inical Study Report No. CA22736 | |
|---|---|
| Table 14.2.6.3.4 | Summary of Future Intent to Use VAS Score in Each<br>Category by Study Product for Ad Libitum Product Use<br>Session (Outcomes Population) |
| Table 14.2.6.3.5 | Summary of Future Intent to Use VAS Raw Scores by<br>Study Product for Contolled Product Use Session<br>(Outcomes Population) |
| Table 14.2.6.3.6 | Summary of Future Intent to Use VAS Raw Scores by Study Product for Ad Libitum Product Use Session (Outcomes Population) |
| 14.2.6.4 PSCDI or | PSECDI Total Score |
| Table 14.2.6.4 | Summary of PSCDI or PSECDI Total Score by Study<br>Arm and Study Day (Outcomes Population) |
| 14.2.6.5 MTWS-R | Total Score |
| Table 14.2.6.5 | Summary of MTWS-R Total Score by Study Arm and Study Day (Outcomes Population) |
| 14.2.6.6 QSU-brie | f Factor Scores |
| Table 14.2.6.6 | Summary of QSU-brief Factor Scores by Study Arm and Study Day (Outcomes Population) |
| 14.2.7 Topograph | y |
| Table 14.2.7 | Summary of Puff Topography Parameters by Study Day (Outcomes Population) |
| 14.2.8 Ph | narmacokinetics Figures |
| Figure 14.2.8.1 | Arithmetic Mean (SD) Baseline-adjusted Plasma<br>Nicotine Concentration Versus Time Profiles Following<br>Controlled Use (Linear Scale) (Outcomes Population) |
| Figure 14.2.8.2 | Arithmetic Mean Plasma Baseline-adjusted Nicotine<br>Concentration Versus Time Profiles Following<br>Controlled Use (Linear Scale) (Outcomes Population) |
| Figure 14.2.8.3 | Arithmetic Mean Plasma Baseline-adjusted Nicotine<br>Concentration Versus Time Profiles Following<br>Controlled Use (Semi-log Scale) (Outcomes<br>Population) |
| Note: Individual ba | seline-adjusted profiles will be presented in Appendix 16.2.6.1 of the report. |
| 14.2.9 Biomarker | Figures |

#### 14.2.9.1 Part 1

Figure 14.2.9.1.1 Arithmetic Mean (SD) Blood COHb by Study Day in Part 1: 9-Day Switch to Exclusive myblu<sup>TM</sup> Use (Outcomes Population)

#### Clinical Study Report No. CA22736

Figures 14.2.9.1.2 through 14.2.9.1.19 (one per biomarker) will be generated similarly:

Figure 14.2.9.1.2 Urine NNAL Figure 14.2.9.1.3 Urine 3-HPMA Figure 14.2.9.1.4 Urine S-PMA Figure 14.2.9.1.5 Urine NNN Figure 14.2.9.1.6 Urine CEMA Figure 14.2.9.1.7 Urine HEMA Figure 14.2.9.1.8 Urine 3-HMPMA Figure 14.2.9.1.9 Urine 1-OHP Figure 14.2.9.1.10 Urine o-tol Figure 14.2.9.1.11 Urine 3-OH B[a]P Figure 14.2.9.1.12 Urine 1-AN Figure 14.2.9.1.13 Urine 2-AN Figure 14.2.9.1.14 Plasma sICAM Figure 14.2.9.1.15 **WBCs** Figure 14.2.9.1.16 Serum HDL-C Figure 14.2.9.1.17 Serum MCP-1 Figure 14.2.9.1.18 Urine 8-epi-prostaglandin F2α Figure 14.2.9.1.19 Urine 11-dehydrothromboxane B2

#### **14.2.9.2** Part 2 by Study Day

Figure 14.2.9.2.1 Arithmetic Mean (SD) Blood COHb (% Saturation) by Study Day in Part 2: Continue Exclusive myblu<sup>TM</sup> Use (Outcomes Population)

Figures 14.2.9.2.2 through 14.2.9.2.19 (one per biomarker) will be generated similarly:

| Figure 14.2.9.2.2 | Urine NNAL |
|--------------------|---------------------|
| Figure 14.2.9.2.3 | Urine 3-HPMA |
| Figure 14.2.9.2.4 | Urine S-PMA |
| Figure 14.2.9.2.5 | Urine NNN |
| Figure 14.2.9.2.6 | Urine CEMA |
| Figure 14.2.9.2.7 | Urine HEMA |
| Figure 14.2.9.2.8 | Urine 3-HMPMA |
| Figure 14.2.9.2.9 | Urine 1-OHP |
| Figure 14.2.9.2.10 | Urine o-tol |
| Figure 14.2.9.2.11 | Urine 3- 3-OH B[a]P |
| Figure 14.2.9.2.12 | Urine 1-AN |

#### Clinical Study Report No. CA22736

| Figure 14.2.9.2.13 | Urine 2-AN |
|---|---|
| Figure 14.2.9.2.14 | Plasma sICAM |
| Figure 14.2.9.2.15 | WBCs |
| Figure 14.2.9.2.16 | Serum HDL-C |
| Figure 14.2.9.2.17 | Serum MCP-1 |
| Figure 14.2.9.2.18 | Urine 8-epi-prostaglandin F2α |
| Figure 14.2.9.2.19 | Urine 11-dehydrothromboxane B2 |
| 14.2.9.3 Part 2 by Study Arm | |
| Figure 14.2.9.3.1 | Arithmetic Mean (SD) Blood COHb (% Saturation) by |
| | $C_{i}$ 1 D : D $i$ 2 $i$ 0 $i$ D $i$ 1 $i$ 1 |

Study Day in Part 2 (Outcomes Population)

Figures 14.2.9.3.2 through 14.2.9.3.19 (one per biomarker) will be generated

similarly: Figure 14.2.9.3.2 Urine NNAL

Figure 14.2.9.3.3 Urine 3-HPMA

Figure 14.2.9.3.4 Urine S-PMA

Figure 14.2.9.3.5 Urine NNN

Figure 14.2.9.3.6 Urine CEMA

Figure 14.2.9.3.7 Urine HEMA

Figure 14.2.9.3.8 Urine 3-HMPMA

Figure 14.2.9.3.9 Urine 1-OHP

Figure 14.2.9.3.10 Urine o-tol

Figure 14.2.9.3.11 Urine 3- 3-OH B[a]P

Figure 14.2.9.3.12 Urine 1-AN

Figure 14.2.9.3.13 Urine 2-AN

Figure 14.2.9.3.14 Plasma sICAM

Figure 14.2.9.3.15 WBCs

Figure 14.2.9.3.16 Serum HDL-C

Figure 14.2.9.3.17 Serum MCP-1

Figure 14.2.9.3.18 Urine 8-epi-prostaglandin F2α

Figure 14.2.9.3.19 Urine 11-dehydrothromboxane B2

#### 14.2.10 Physiologic Assessments Figures

#### 14.2.10.1 SBP, DBP, HR

Figure 14.2.10.1.1 Change from Baseline Systolic Blood Pressure Versus Time (Arm I) (Outcomes Population)

| Figure 14.2.10.1.2 | Change From Baseline Diastolic Blood Pressure Versus |
|--------------------|------------------------------------------------------|
| | Time (Arm I) (Outcomes Population) |
| Figure 14.2.10.1.3 | Change From Baseline Heart Rate Versus Time (Arm I) |
| | (Outcomes Population) |

The 24-hour change-from-baseline profiles for each endpoint, for Day 9 and Day 14, will be plotted, with y axis = Change from Baseline (unit) and x axis = time (hr)

#### **14.2.10.2 Lung Function**

| Figure 14.2.10.2.1 | Box Plot of Change From Baseline Pre-Bronchodilator<br>Percent of Predicted FEV1 by Study Day (Outcomes<br>Population) |
|---|---|
| Figure 14.2.10.2.2 | Box Plot of Change From Baseline Pre-Bronchodilator<br>Percent of Predicted FVC by Study Day (Outcomes<br>Population) |
| Figure 14.2.10.2.3 | Box Plot of Change From Baseline Pre-Bronchodilator<br>Percent of Predicted FEV1:FVC by Study Day<br>(Outcomes Population) |
| Figure 14.2.10.2.4 | Box Plot of Change From Baseline Pre-Bronchodilator<br>Percent of Predicted FEF25-75% by Study Day<br>(Outcomes Population) |
| Figure 14.2.10.2.5 | Box Plot of Change From Baseline Post-Pre-<br>Bronchodilator Percent of Predicted FEV1 by Study<br>Day (Outcomes Population) |
| Figure 14.2.10.2.6 | Box Plot of Change From Baseline Post-Pre-<br>Bronchodilator Percent of Predicted FVC by Study Day<br>(Outcomes Population) |
| Figure 14.2.10.2.7 | Box Plot of Change From Baseline Post-Pre-<br>Bronchodilator Percent of Predicted FEV1:FVC by<br>Study Day (Outcomes Population) |
| Figure 14.2.10.2.8 | Box Plot of Change From Baseline Post-Pre-<br>Bronchodilator Percent of Predicted FEF25-75% by<br>Study Day (Outcomes Population) |

#### 14.2.11 Urge to Smoke Figures

Figure 14.2.11.1 Arithmetic Mean (SD) of Urge to Smoke Versus Time by Study Product Following Controlled Use (Outcomes Population)

Figure 14.2.11.2 Arithmetic Mean of Urge to Smoke Versus Time by Study Product Following Controlled Use (Outcomes Population)

### 14.2.12 Questionnaire Figures

#### 14.2.12.1 PES Subscales

| 14.2.12.1 PES Subs | scales |
|---|---|
| Figure 14.2.12.1.1 | Box Plot of PES Subscales (Satisfaction) by Study<br>Product Following Controlled Product Use (Outcomes<br>Population) |
| Figure 14.2.12.1.2 | Box Plot of PES Subscales (Satisfaction) by Study<br>Product Following Ad Libitum Product Use (Outcomes<br>Population) |
| Figure 14.2.12.2.1 | Box Plot of PES Subscales (Psychological Reward)<br>Following Controlled Product Use Episode (Outcomes<br>Population) |
| Figure 14.2.12.2.2 | Box Plot of PES Subscales (Psychological Reward) by<br>Study Product Following Ad Libitum Product Use<br>(Outcomes Population) |
| Figure 14.2.12.3.1 | Box Plot of PES Subscales (Aversion) by Study Product<br>Following Controlled Product Use (Outcomes<br>Population) |
| Figure 14.2.12.3.2 | Box Plot of PES Subscales (Aversion) by Study Product<br>Following Ad Libitum Product Use (Outcomes<br>Population) |
| Figure 14.2.12.4.1 | Box Plot of PES Subscales (Relief) by Study Product<br>Following Controlled Product Use |
| Figure 14.2.12.4.2 | Box Plot of PES Subscales (Relief) by Study Product<br>Following Ad Libitum Product Use (Outcomes<br>Population) |
| Figure 14.2.12.5.1 | Box Plot of PES Subscales (Item 17) by Study Product Following Controlled Product Use (Outcomes Population) |
| Figure 14.2.12.5.2 | Box Plot of PES Subscales (Item 17) by Study Product<br>Following Ad Libitum Product Use (Outcomes<br>Population) |
| Figure 14.2.12.6.1 | Box Plot of PES Subscales (Item 19) by Study Product Following Controlled Product Use (Outcomes Population) |
| Figure 14.2.12.6.2 | Box Plot of PES Subscales (Item 19) by Study Product<br>Following Ad Libitum Product Use (Outcomes<br>Population) |

| Figure 14.2.12.7.1 | Box Plot of PES Subscales (Item 21) by Study Product Following Controlled Product Use (Outcomes Population) |
|---|---|
| Figure 14.2.12.7.2 | Box Plot of PES Subscales (Item 21) by Study Product Following Ad Libitum Product Use (Outcomes Population) |
| 14.2.13 Product Li | king VAS Score |
| Figure 14.2.13.1 | Box Plot of Product Liking VAS Score by Study Product Following Controlled Product Use |
| Figure 14.2.13.2 | Box Plot of Product Liking VAS Score by Study Product Following Ad Libitum Product Use (Outcomes Population) |
| 14.2.14 Future Inte | ent to Use VAS Score |
| Figure 14.2.14.1.1 | Frequency of Future Intent to Use (Likely to Smoke) by Study Product Following Controlled Product Use |
| Figure 14.2.14.1.2 | Frequency of Future Intent to Use (Likely to Smoke) by<br>Study Product Following Ad Libitum Product Use<br>(Outcomes Population) |
| Figure 14.2.14.2.1 | Frequency of Future Intent to Use (Not Likely to Smoke) by Study Product Following Controlled Product Use |
| Figure 14.2.14.2.2 | Frequency of Future Intent to Use (Not Likely to Smoke) by Study Product Following Ad Libitum Product Use (Outcomes Population) |
| Figure 14.2.14.3.1 | Frequency of Future Intent to Use (Likely to Buy<br>Assigned Product) by Study Product Following<br>Controlled Product Use |
| Figure 14.2.14.3.2 | Frequency of Future Intent to Use (Likely to Buy<br>Assigned Product) by Study Product Following Ad<br>Libitum Product Use (Outcomes Population) |
| Figure 14.2.14.4.1 | Frequency of Future Intent to Use (Not Likely to Buy<br>Assigned Product by Study Product Following<br>Controlled Product Use |
| Figure 14.2.14.4.2 | Frequency of Future Intent to Use (Not Likely to Buy<br>Assigned Product) by Study Product Following Ad<br>Libitum Product Use (Outcomes Population) |
| Figure 14.2.14.5.1 | Frequency of Future Intent to Use (Likely to Buy<br>Another E-Cigarette) by Study Product Following<br>Controlled Product Use |
| Figure 14.2.14.5.2 | Frequency of Future Intent to Use (Likely to Buy<br>Another E-Cigarette) by Study Product Following Ad<br>Libitum Product Use (Outcomes Population) |

Figure 14.2.14.6.1 Frequency of Future Intent to Use (Not Likely to Buy Another E-Cigarette) by Study Product Following Controlled Product Use

Figure 14.2.14.7.2 Frequency of Future Intent to Use (Not Likely to Buy Another E-Cigarette) by Study Product Following Ad Libitum Product Use (Outcomes Population)

### Note: Above figures will be bar graphs

#### 14.2.15 PSCDI or PSECDI Total Score

Figure 14.2.15 Box plot of PSCDI or PSECDI Total Score by Study Arm and Study Day (Outcomes Population)

#### 14.2.16 MTWS-R Total Score

Figure 14.2.16 Box Plot of MTWS-R Total Score by Study Arm and Study Day (Outcomes Population)

#### 14.2.17 QSU-brief Factor Scores

Figure 14.2.17.1 Box Plot of QSU-brief Factor Scores (Factor 1) by Study Product and Study Day (Outcomes Population)

Figure 14.2.17.3 Box Plot of QSU-brief Factor Scores (Factor 2) by Study Product and Study Day (Outcomes Population)

#### 14.3 Safety Data Summary Tables

#### 14.3.1 Displays of Adverse Events

- Table 14.3.1.1.1 Product Use-emergent Adverse Event Frequency by Study Product – Number of Subjects Reporting the Event (% of Subjects Who Used Study Product) - Part 1 (Safety Population)
- Table 14.3.1.1.2 Product Use-emergent Adverse Event Frequency by Study Product – Number of Adverse Events (% of Total Adverse Events) – Part 1 (Safety Population)
- Table 14.3.1.1.3 Product Use-emergent Adverse Event Frequency by Study Product, Severity, and Relationship to Study Product – Number of Subjects Reporting Events - Part 1 (Safety Population)
- Table 14.3.1.2.1 Product Use-emergent Adverse Event Frequency by Study Arm – Number of Subjects Reporting the Event (% of Subjects Who Used Study Product) - Part 2 (Safety Population)

- Table 14.3.1.2.2 Product Use-emergent Adverse Event Frequency by Study Arm – Number of Adverse Events (% of Total Adverse Events) – Part 2 (Safety Population)
- Table 14.3.1.2.3 Product Use-emergent Adverse Event Frequency by Study Arm, Severity, and Relationship to Study Product – Number of Subjects Reporting Events - Part 2 (Safety Population)

#### 14.3.2 Listings of Deaths, other Serious and Significant Adverse Events

Table 14.3.2.1 Serious Adverse Events (Safety Population) <if no serious adverse event occurred, a statement 'No serious adverse event is reported'>

## 14.3.3 Narratives of Deaths, other Serious and Certain other Significant Adverse Events

#### 14.3.4 Abnormal Laboratory Value Listing (each subject)

- Table 14.3.4.1 Out-of-Range Values and Recheck Results Serum Chemistry (Safety Population)
- Table 14.3.4.2 Out-of-Range Values and Recheck Results Hematology (Safety Population)
- Table 14.3.4.3 Out-of-Range Values and Recheck Results Urinalysis (Safety Population)
- Table 14.3.4.4 Clinically Significant Values and Recheck Results (Safety Population)

## 14.3.5 Displays of Other Laboratory, Vital Signs, Electrocardiogram, Physical Examination, and Other Safety Data

- Table 14.3.5.1 Clinical Laboratory Summary Serum Chemistry (Safety Population)
- Table 14.3.5.2 Clinical Laboratory Summary Hematology (Safety Population)
- Table 14.3.5.3 Clinical Laboratory Summary Urinalysis (Safety Population)
- Table 14.3.5.4 Vital Sign Summary (Safety Population)
- Table 14.3.5.5 12-Lead Electrocardiogram Summary (Safety Population)
- Table 14.3.5.6 Spirometry Summary (Safety Population)

#### **Section 16 Data Listings**

Note: Hepatitis and HIV results that are provided by the clinical laboratory will not be presented in subject data listings and will not be included in any database transfer.

Data listings are numbered following the ICH structure but may be renumbered as appropriate during the compilation of the TFLs for the CSR. The following is a list of appendix numbers and titles that will be included as data listings:

#### **16.1** Study Information

Appendix 16.1.9 Statistical Methods

Appendix 16.1.10.1 Clinical Laboratory Reference Ranges

#### 16.2 Subject Data Listings

#### 16.2.1 Subject Discontinuation

Appendix 16.2.1.1 Subject Discontinuation (Safety Population)

#### **16.2.2 Protocol Deviations**

Appendix 16.2.2 Protocol Deviations

#### 16.2.3 Subjects Excluded from Analysis

Appendix 16.2.3 Subjects Excluded from Analysis

Note: Appendix 16.2.3 is generated in MS Word for inclusion in the study report.

#### 16.2.4 Demographic Data

| Appendix 16.2.4.1.1 | Demographics (Safety Population) |
|---|---|
| Appendix 16.2.4.1.2 | Reproductive Status (Safety Population) |
| Appendix 16.2.4.2 | Physical Examination (Safety Population) |
| Appendix 16.2.4.3.1 | Medical History (Safety Population) |
| Appendix 16.2.4.3.2 | Allergy History (Safety Population) |
| Appendix 16.2.4.3.3 | Surgical History (Safety Population) |
| Appendix 16.2.4.4 | Smoking History (Safety Population) |
| Appendix 16.2.4.5 | Caffeine, Alcohol, and Drug History (Safety Population) |

#### 16.2.5 Compliance and/or Concentration Data

| Appendix 16.2.5.1.1 | Inclusion Criteria |
|---------------------|-------------------------------------------|
| Appendix 16.2.5.1.2 | Exclusion Criteria |
| Appendix 16.2.5.2 | Subject Eligibility (Safety Population) |
| Appendix 16.2.5.3 | Randomization (Safety Population) |
| Appendix 16.2.5.4.1 | Usual Brand Cigarette (Safety Population) |

| Appendix 16.2.5.4.2 | Test Product Administration (Safety Population) |
|---|---|
| Appendix 16.2.5.4.3 | Ad Libitum Product Use (Safety Population) |
| Appendix 16.2.5.4.4 | Product Use Behavior – Pod Weight (Safety Population) |
| Appendix 16.2.5.5.1 | Blood Draw Times (Safety Population) |
| Appendix 16.2.5.5.2 | 24-Hour Urine Collection (Safety Population) |
| Appendix 16.2.5.6 | Meal Times (Safety Population) |
| Appendix 16.2.5.7 | Prior and Concomitant Medications (Safety Population) |
| 16.2.6 | Individual Pharmacokinetics, Biomarker, Subjective |
| 10.2.0 | Effects and Topography Data |
| Appendix 16.2.6.1 Inc | dividual Baseline-Adjusted Plasma Nicotine<br>Concentrations For Subject # |
| Appendix 16.2.6.2.1 | Blood COHb (Outcomes Population) |
| Appendix 16.2.6.2.2 | Urine NNAL (Outcomes Population) |
| Appendix 16.2.6.2.3 | Urine 3-HPMA (Outcomes Population) |
| Appendix 16.2.6.2.4 | Urine S-PMA (Outcomes Population) |
| Appendix 16.2.6.2.5 U | Urine NNN (Outcomes Population) |
| Appendix 16.2.6.2.6 | Urine CEMA (Outcomes Population) |
| Appendix 16.2.6.2.7 | Urine HEMA (Outcomes Population) |
| Appendix 16.2.6.2.8 | Urine HMPMA (Outcomes Population) |
| Appendix 16.2.6.2.9 | Urine MHBMA (Outcomes Population) |
| Appendix 16.2.6.2.10 | Urine 1-OHP (Outcomes Population) |
| Appendix 16.2.6.2.11 | Urine o-tol (Outcomes Population) |
| Appendix 16.2.6.2.12 | Urine 3-OH B[a]P (Outcomes Population) |
| Appendix 16.2.6.2.13 | Urine 1-AN (Outcomes Population) |
| Appendix 16.2.6.2.14 | Urine 2-AN (Outcomes Population) |
| Appendix 16.2.6.2.15 | .1 Urine Nicotine and Metabolites (Outcomes |
| | Population) |
| = = | .2 Urine Nicotine Equivalents (Outcomes Population) |
| | Plasma sICAM (Outcomes Population) |
| | WBCs (Outcomes Population) |
| | Serum HDL-C (Outcomes Population) |
| | Serum MCP-1 (Outcomes Population) |
| Appendix 16.2.6.2.20 | Urine Type III isoprostane (8-epi-prostaglandin F2α) (Outcomes Population) |
| Appendix 16.2.6.2.21 | Urine 11-dehydrothromboxane B2 (Outcomes Population) |

| | <b>7</b> 1 | |
|---|---|---|
| | Appendix 16.2.6.3.1 | PES Questionnaire (Outcomes Population) |
| | Appendix 16.2.6.3.2 | PES Questionnaire Responses (Outcomes Population) |
| | Appendix 16.2.6.3.3 | PES Questionnaire Subscales (Outcomes Population) |
| Appendix 16.2.6.4 | | Product Liking Questionnaire Responses (Outcomes Population) |
| | Appendix 16.2.6.5 | Future Intent to Use Questionnaire Responses (Outcomes Population) |
| | Appendix 16.2.6.6.1 | PSCDI, PSECDI Questionnaire (Outcomes Population) |
| | Appendix 16.2.6.6.2 | PSCDI, PSECDI Questionnaire Responses (Outcomes Population |
| | Appendix 16.2.6.7.1 | MTWS-R Questionnaire (Outcomes Population) |
| | Appendix 16.2.6.7.2 | MTWS-R Questionnaire Responses (Outcomes Population) |
| | Appendix 16.2.6.8.1 | QSU-brief Questionnaire (Outcomes Population) |
| | Appendix 16.2.6.8.2 | QSU-brief Questionnaire Responses (Outcomes Population |
| | Appendix 16.2.6.9 | Individual Puff Topography Parameters (Outcomes Population) |
| | 16.2.7 Adverse Ev | rents Listings |
| | Appendix 16.2.7.1.1 | Adverse Events (I of II) (Safety Population) |
| | Appendix 16.2.7.1.2 | Adverse Events (II of II) (Safety Population) |
| | Appendix 16.2.7.2 | Adverse Event Non- Medication Therapy (Safety Population) |
| | Appendix 16.2.7.3 | Adverse Event Preferred Term Classification (Safety Population) |
| | 16.2.8 Listings of Safety Obse | Individual Laboratory Measurements and Other ervations |
| | Appendix 16.2.8.1.1 | Clinical Laboratory Report - Serum Chemistry (Safety Population) |
| | Appendix 16.2.8.1.2 | Clinical Laboratory Report - Hematology (Safety Population) |
| | Appendix 16.2.8.1.3 | Clinical Laboratory Report - Urinalysis (Safety Population) |
| | Appendix 16.2.8.1.4 | Clinical Laboratory Report - Urine Drug Screen (Safety Population) |
| | Appendix 16.2.8.1.5 | Clinical Laboratory Report - Comments (Safety |

Population)

| Appendix 16.2.8.1.6 | Alcohol Breath Testing (Safety Population) |
|---------------------|---------------------------------------------------|
| Appendix 16.2.8.2 | Vital Signs (Safety Population) |
| Appendix 16.2.8.3 | 12-Lead Electrocardiogram (Safety Population) |
| Appendix 16.2.8.4 | Carbon Monoxide Breath Test (Safety Population) |
| Appendix 16.2.8.5 | Administration of Albuterol (Safety Population) |
| Appendix 16.2.8.6 | Spirometry (Safety Population) |
| Appendix 16.2.8.7 | Tobacco Cessation Information (Safety Population) |

#### 10. TABLE AND FIGURE SHELLS

The following table and figure shells provide a framework for the display of data from this study. The shells may change due to unforeseen circumstances. These shells may not be reflective of every aspect of this study, but are intended to show the general layout of the tables that will be presented and included in the final report. Unless otherwise noted, all tables will be presented in Times New Roman font size 8. These tables will be generated off of the ADaM Version 1.0.

#### 10.1 Figures Shells

In-text and post-text PK Figures of mean plasma concentrations and UTS on linear scale will be in the following format: Figure 11-X, 14.X, and appendix 16.2.6.1:

Figure X.X Arithmetic Mean Baseline-Adjusted Plasma Nicotine Concentration-Time Profiles Following Controlled Product Use by Product (Linear Scale) (Outcomes Population)



Program: /CAXXXXX/sas\_prg/pksas/adam\_meangraph.sas DDMMMYYY HH:MM Program: /CAXXXXX/sas\_prg/pksas/meangraph.sas DDMMMYYY HH:MM

#### Notes for Generating the Actual Mean Figure:

- I. Legend will use the short descriptions
- II. Y axis label will be "Plasma Nicotine Concentration (ng/mL)" for PK figures and "Urge to Smoke" for UTS figure
- III. X axis label will be "Minutes from Product Use" for all figures

Program: /CAXXXXX/sas\_prg/pksas/meangraph.sas DDMMYYYY HH:MM
Program: /CAXXXXX/sas\_prg/pksas/adam\_meangraph.sas DDMMYYYY HH:MM

Post-text PK Figures of mean (SD) plasma concentrations and UTS on linear scale will be in the following format:

Figure 14.X: Arithmetic Mean (SD) Baseline-Adjusted Plasma Nicotine Concentration-Time Profiles Following Controlled Product Use by Product (Linear Scale) (Outcomes Population)



Treatments B and C are shifted to the right for ease of reading

Program: /CAXXXXX/sas\_prg/pksas/adam\_meangraph.sas DDMMMYYY HH:MM Program: /CAXXXXX/sas\_prg/pksas/meangraph.sas DDMMMYYY HH:MM

#### Notes for Generating the Actual Mean Figure:

- IV. Legend will use the short descriptions
- V. Y axis label will be "Plasma Nicotine Concentration (ng/mL)" for PK figures and "Urge to Smoke" for UTS figure
- VI. X axis label will be "Minutes from Product Use" for all figures
- VII. Please add the footnote for products that are shifted to the right for ease of reading

Program: /CAXXXX/sas\_prg/pksas/meangraph.sas DDMMYYYY HH:MM
Program: /CAXXXXX/sas\_prg/pksas/adam\_meangraph.sas DDMMYYYY HH:MM

Post-text PK Figures of mean plasma concentrations on semi-log scale (Figure 14.X, Appendix 16.2.6.1) will be in the following format:

Figure 14.X: Arithmetic Mean Baseline-Adjusted Plasma Nicotine Concentration-Time Profiles Following Controlled Product Use by Product (Semi-Log Scale) (Outcomes Population)



Program: /CAXXXX/sas\_prg/pksas/adam\_meangraph.sas DDMMMYYY HH:MM Program: /CAXXXXX/sas\_prg/pksas/meangraph.sas DDMMMYYY HH:MM

#### Notes for Generating the Actual Mean Figure:

- I. Legend will use the short descriptions
- II. Y axis label will be "Plasma Nicotine Concentration (ng/mL)" for all figures
- III. X axis label will be "Minutes from Product Use" for all figures

Program: /CAXXXX/sas\_prg/pksas/meangraph.sas DDMMYYYY HH:MM
Program: /CAXXXXX/sas\_prg/pksas/adam\_meangraph.sas DDMMYYYY HH:MM

Post-text Figure(s) for Total Scores will be in the following format:

Figure 14.X: Box Plot of PSCDI or PSECDI Total Score by Study Arm and Study Day (Outcomes Population)

#### Notes for Generating the Actual Mean Figure:

- I. Note: this figure will be a boxplot figure
- II. Please present each subjective measurement on different graphs but associated with Figure 14.2.9.1 or similar graphs. Present each question (or factor scale, subscale, or total score) in the title of each graph.
- III. Y axis label will be "Subjective Measurement Score"
- IV. X axis label will be labelled with "A, B, C, D, E, F, G, H" for each figure representing each product or Arm I, J, K as appropriate

### **10.2** Post-Text Summary Tables Shells

#### **14.1 Demographic Tables**

Tables 14.1.1.1 and 14.1.5.1 will have the following format.

Table 14.1.1.1 Summary of Disposition - Part 1 (Safety Population)

Study Product Sequence

Page 1 of  ${\tt X}$ 

| Category | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX | -<br>Overall |
|---|---|---|---|---|---|---|---|---|---|
| Enrolled | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| Completed | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| Discontinued Early | X | X | X | X | X | X | X | X | X |
| <reason1></reason1> | X | X | X | X | X | X | X | X | X |
| <reason2></reason2> | X | X | X | X | X | X | X | X | X |
| <reason3></reason3> | X | X | X | X | X | X | X | X | X |

Note: Product X = < >

Program: /CAXXXXX/ sas\_prg/stsas/tab cdash\_tbldisp1.sas DDMMMYYYY HH:MM

#### Nerudia Ltd.

#### NER 01/003 *my*blu™ E-cigarettes

### Clinical Study Report No. CA22736

#### Tables 14.1.1.2 and 14.1.5.2 will have the following format.

Table 14.1.1.2 Summary of Disposition - Part 2 (Safety Population)

Study Product Arm

| Category | X | X | X | Overall |
|---------------------|----|----|----|---------|
| Enrolled | XX | XX | XX | XX |
| Completed | XX | XX | XX | XX |
| Discontinued Early | X | X | X | X |
| <reason1></reason1> | X | X | X | X |
| <reason2></reason2> | X | X | X | X |
| <reason3></reason3> | X | X | X | X |

Note: Study Arm X = < >

Program: /CAXXXXX/ sas\_prg/stsas/tab cdash\_tbldisp1.sas DDMMMYYYY HH:MM

Statistical Analysis Plan, 26 February 2020


#### Table 14.1.2 will have the following format.


Table 14.1.2 Disposition of Subjects (Safety Population)

| Cubicat | | Study Product Administration/ Completed | | | | | Study Completion | |
|---|---|---|---|---|---|---|---|---|
| Subject Product Number Sequence/Arm | | Period 1 | Period 2 | Period 3 | Period 4 | Part 2 | Status | Date |
| X | XXXX/X | Yes/Yes | Yes/Yes | Yes/Yes | Yes/ No | Yes/ No | Terminated Study Prematurely | DDMMMYYYY |
| X | XXXX/X | Yes/Yes | Yes/Yes | Yes/Yes | Yes/Yes | Yes/Yes | Completed Study | DDMMMYYYY |
| X | XXXX/X | Yes/Yes | Yes/Yes | Yes/Yes | Yes/Yes | Yes/Yes | Completed Study | DDMMMYYYY |
| X | XXXX/X | Yes/Yes | Yes/Yes | Yes/Yes | Yes/Yes | Yes/Yes | Completed Study | DDMMMYYYY |
| | | XX/XX | XX/XX | XX/XX | XX/XX | xx/xx | | |

Note: Product X = < >

Program: /CAXXXXX/sas\_prg/stsas/tab cdash\_tbldisp2.sas DDMMMYYYY HH:MM

Tables 14.1.3.1 and 14.1.6.1 will have the following format.

Table 14.1.3.1 Demographic Summary - Part 1 (Safety Population)


| | | | | Study | Product Se | equence | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Trait | | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX | Overall |
| Sex | Male<br>Female | X (XX.X%)<br>X (XX.X%) | X (XX.X%)<br>X (XX.X%) | X (XX.X%)<br>X (XX.X%) | X (XX.X%)<br>X (XX.X%) | X (XX.X%)<br>X (XX.X%) | X (XX.X%)<br>X (XX.X%) | X (XX.X%)<br>X (XX.X% | | X (XX.X%)<br>X (XX.X%) |
| Race | XXXXXXXXX<br>XXXXX | X (XX.X%)<br>X (XX.X%)<br>X (XX.X%) | X (XX.X%)<br>X (XX.X%)<br>X (XX.X%) | X (XX.X%)<br>X (XX.X%)<br>X (XX.X%) | X (XX.X%)<br>X (XX.X%)<br>X (XX.X%) | X (XX.X%)<br>X (XX.X%)<br>X (XX.X%) | X (XX.X%)<br>X (XX.X%)<br>X (XX.X%) | X (XX.X%<br>X (XX.X%<br>X (XX.X% | X (XX.X%) | X (XX.X%)<br>X (XX.X%)<br>X (XX.X%) |
| Ethnicity | Hispanic or Latino<br>Not Hispanic or<br>Latino | X(XX.X%)<br>X(XX.X%) | X (XX.X%)<br>X (XX.X%) | X (XX.X%)<br>X (XX.X%) | X (XX.X%)<br>X (XX.X%) | X (XX.X%)<br>X (XX.X%) | X (XX.X%)<br>X (XX.X%) | X (XX.X%<br>X (XX.X% | | X(XX.X%)<br>X(XX.X%) |
| Age (yrs) | n<br>Mean<br>SD<br>Minimum<br>Median<br>Maximum | x<br>x.x<br>x.xx<br>xx<br>xx<br>xx<br>xx | x<br>x.x<br>x.xx<br>xx<br>xx<br>xx<br>xx | X<br>X.X<br>X.XX<br>XX<br>XX<br>XX | X<br>X.X<br>X.XX<br>XX<br>XX<br>XX | X<br>X.X<br>X.XX<br>XX<br>XX<br>XX | X<br>X.X<br>X.XX<br>XX<br>XX<br>XX | x<br>x.x<br>x.xx<br>x.xx<br>xx | X<br>X<br>X.X<br>X.XX<br>XX<br>XX | X<br>X.X<br>X.XX<br>XX<br>XX<br>XX |

Note: Product X = < >

Program: /CAXXXXX/sas\_prg/stsas/tab cdash\_demsum.sas DDMMMYYYY HH:MM

Programmer Note: Weight (kg), Height (cm), and BMI (kg/m^2) will also be included in the demographic summary table.

#### Nerudia Ltd.

#### NER 01/003 *my*blu™ E-cigarettes

Clinical Study Report No. CA22736

Tables 14.1.3.2 and 14.1.6.2 will have the following format.

Table 14.1.3.2 Demographic Summary - Part 2 (Safety Population)

Study Product Arm


| | | | _ | | |
|---|---|---|---|---|---|
| Trait | | Х | Х | Х | Overall |
| Sex | Male | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| | Female | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| Race | XXXXXXXXX | X(XX.X%) | X (XX.X%) | X(XX.X%) | X (XX.X%) |
| | XXXXX | X(XX.X%) | X(XX.X%) | X(XX.X%) | X(XX.X%) |
| | XXXXX | X(XX.X%) | X(XX.X%) | X(XX.X%) | X (XX.X%) |
| Ethnicity | Hispanic or Latino | X(XX.X%) | X (XX.X%) | X(XX.X%) | X (XX.X%) |
| | Not Hispanic or<br>Latino | X(XX.X%) | X(XX.X%) | X(XX.X%) | X (XX.X%) |
| Age (yrs) | n | X | X | X | X |
| | Mean | X.X | X.X | X.X | X.X |
| | SD | X.XX | X.XX | X.XX | X.XX |
| | Minimum | XX | XX | XX | XX |
| | Median | X.X | X.X | X.X | X.X |
| | Maximum | XX | XX | XX | XX |

Note: Study Product Arm X = < >

Program: /CAXXXXX/sas\_prg/stsas/tab cdash\_demsum.sas DDMMMYYYY HH:MM

Programmer Note: Weight (kg), Height (cm), and BMI (kg/m^2) will also be included in the demographic summary table.

Tables 14.1.4.1 and 14.1.7.1 will have the following format.


Table 14.1.4.1 Smoking History Summary - Part 1 (Safety Population)

| | | Study Product Sequence | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Trait | | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX | Overall |
| Brand | XXXX | X (XX.X%)<br>X (XX.X%) | X (XX.X%)<br>X (XX.X%) | X (XX.X%)<br>X (XX.X%) | X (XX.X%)<br>X (XX.X%) | X (XX.X%)<br>X (XX.X%) | X (XX.X%)<br>X (XX.X%) | X (XX.X%)<br>X (XX.X%) | , | X (XX.X%)<br>X (XX.X%) |
| Flavor | XXXXXX<br>XXXXX | X(XX.X%)<br>X(XX.X%) | X (XX.X%)<br>X (XX.X%) | X (XX.X%)<br>X (XX.X%) | X(XX.X%)<br>X(XX.X%) | X(XX.X%)<br>X(XX.X%) | X (XX.X%)<br>X (XX.X%) | X (XX.X%)<br>X (XX.X%) | . , | X (XX.X%)<br>X (XX.X%) |
| Number of Cigarettes<br>Smoked per Day | n<br>Mean<br>SD<br>Minimum<br>Median<br>Maximum | X<br>X.X<br>X.XX<br>XX<br>XX<br>X.X | X<br>X.X<br>X.XX<br>XX<br>XX<br>XX | X<br>X.X<br>X.XX<br>XX<br>XX<br>X.X | X<br>X.X<br>X.XX<br>XX<br>XX<br>XX | X<br>X.X<br>X.XX<br>XX<br>XX<br>XX | X<br>X.X<br>X.XX<br>XX<br>XX<br>X.X | X<br>X.X<br>X.XX<br>XX<br>XX<br>XX | X<br>X.X<br>X.XX<br>XX<br>XX<br>XX | X<br>X.X<br>X.XX<br>XX<br>XX<br>XX |

Note: Product X = < >

Program: /CAXXXXX/sas prg/stsas/tab cdash demsum.sas DDMMMYYYY HH:MM

Programmer Note: Flavor and cigarette length will also be included in the smoking history summary table.

Clinical Study Report No. CA22736

Tables 14.1.4.2 and 14.1.7.2 will have the following format.

Table 14.1.4.2 Smoking History Summary - Part 2 (Safety Population)

Page 1 of  ${\tt X}$ 

| Trait | | X | X | Х | Overall |
|---|---|---|---|---|---|
| Brand | XXXX | X (XX.X%) | X (XX.X%) | X (XX.X%) | X (XX.X%) |
| | XXXXXX | X(XX.X%) | X(XX.X%) | X(XX.X%) | X(XX.X%) |
| Flavor | XXXXXX | X(XX.X%) | X (XX.X%) | X(XX.X%) | X(XX.X%) |
| | XXXXX | X(XX.X%) | X(XX.X%) | X(XX.X%) | X(XX.X%) |
| Number of Cigarettes | n | X | X | Х | Х |
| Smoked per Day | Mean | X.X | X.X | X.X | X.X |
| | SD | X.XX | X.XX | X.XX | X.XX |
| | Minimum | XX | XX | XX | XX |
| | Median | X.X | X.X | X.X | X.X |
| | Maximum | XX | XX | XX | XX |

Study Product Arm

Note: Study Product Arm X = < >

Program: /CAXXXXX/sas\_prg/stsas/tab cdash\_demsum.sas DDMMMYYYY HH:MM

Programmer Note: Flavor and cigarette length will also be included in the smoking history summary table.

Clinical Study Report No. CA22736

#### **14.2.1 Product Use Tables**

Note: Summary Tables 14.2.1.1 through 14.2.1.4 will have the following format:

Page 1 of X Table 14.2.1.1 Summary of Pod Weight Changes by Study Product and Study Day Following Controlled Use (Outcomes Population)

| | | | Study Day | | | |
|---|---|---|---|---|---|---|
| Pro | oduct | Statistic | 2 | 4 | 6 | 8 |
| Overall | <br>А | n | X | X | X | X |
| | | Mean | X.X | X.X | X.X | X.X |
| | | SD | X.XX | X.XX | X.XX | X.XX |
| | | CV (%) | XX.X | XX.X | XX.X | XX.X |
| | | SEM | X.XX | X.XX | X.XX | X.XX |
| | | Minimum | XX | XX | XX | XX |
| | | Median | X.X | X.X | X.X | X.X |
| | | Maximum | XX | XX | XX | XX |
| | В | n | X | X | X | X |
| | | Mean | X.X | X.X | X.X | X.X |
| | | SD | X.XX | X.XX | X.XX | X.XX |
| | | CV (%) | XX.X | XX.X | XX.X | XX.X |
| | | SEM | X.XX | X.XX | X.XX | X.XX |
| | | Minimum | XX | XX | XX | XX |
| | | Median | X.X | X.X | X.X | X.X |
| | | Maximum | XX | XX | XX | XX |
| | С | n | X | X | X | X |
| | | Mean | X.X | X.X | X.X | X.X |
| | | SD | X.XX | X.XX | X.XX | X.XX |
| | | CV (%) | XX.X | XX.X | XX.X | XX.X |
| | | SEM | X.XX | X.XX | X.XX | X.XX |
| | | Minimum | XX | XX | XX | XX |
| | | Median | X.X | X.X | X.X | X.X |
| | | Maximum | XX | XX | XX | XX |
| D, E, F, 0 | G <b>,</b> H | <same abo<="" as="" td=""><td>ve&gt;</td><td></td><td></td><td></td></same> | ve> | | | |

Female <Same as above>

Male <Same as above>

Note: Product < X >

Programming Note: Table 14.2.1.4 will present Days 1 through 8


Table 14.2.1.5 Summary of Pod Weight Changes by Study Product and Study Day Following Ad libitum Use on Day 9 (Outcomes Population)

| | | Product | |
|----------|-----------|--------------|--------------|
| Category | Statistic | A, B, C,or D | E, F, G,or H |
| Overall | n | X | X |
| | Mean | X.X | X.X |
| | SD | X.XX | X.XX |
| | CV (%) | XX.X | XX.X |
| | SEM | X.XX | X.XX |
| | Minimum | XX | XX |
| | Median | X.X | X.X |
| | Maximum | XX | XX |

Female <Same as above>

Male <Same as above>

Note: Product: <X>


Table 14.2.1.6 Summary of Pod Weight Changes and Number of Cigarettes Smoked by Study Arm and Study Day (Outcomes Population)

| | | | Weight | Changes | Number of Cigarettes | |
|---|---|---|---|---|---|---|
| Category | Arm | Statistic | Day 9 | Day 14 | Day 9 | Day 14 |
| Overall | I | n | X | X | X | X |
| | | Mean | X.X | X.X | X.X | X.X |
| | | SD | X.XX | X.XX | X.XX | X.XX |
| | | CV (%) | XX.X | XX.X | XX.X | XX.X |
| | | SEM | X.XX | X.XX | X.XX | X.XX |
| | | Minimum | XX | XX | XX | XX |
| | | Median | X.X | X.X | X.X | X.X |
| | | Maximum | XX | XX | XX | XX |
| | J | n | X | X | X | X |
| | | Mean | X.X | X.X | X.X | X.X |
| | | SD | X.XX | X.XX | X.XX | X.XX |
| | | CV (%) | XX.X | XX.X | XX.X | XX.X |
| | | SEM | X.XX | X.XX | X.XX | X.XX |
| | | Minimum | XX | XX | XX | XX |
| | | Median | X.X | X.X | X.X | X.X |
| | | Maximum | XX | XX | XX | XX |
| | K | n | X | X | X | X |
| | | Mean | X.X | X.X | X.X | X.X |
| | | SD | X.XX | X.XX | X.XX | X.XX |
| | | CV (%) | XX.X | XX.X | XX.X | XX.X |
| | | SEM | X.XX | X.XX | X.XX | X.XX |
| | | Minimum | XX | XX | XX | XX |
| | | Median | X.X | X.X | X.X | X.X |
| | | Maximum | XX | XX | XX | XX |

Female <Same as above>

Male <Same as above>

Note: Arm I: Exclusive use of  $\mathsf{myblu^{\mathtt{TM}}}$  products ad libitum

Arm J: Exclusive smoking of usual brand combustible cigarettes ad libitum

Arm K: Smoking of usual brand combustible cigarettes (up to 50% of the subject's self-reported CPD) and use of myblu™ products ad libitum

Programming note: Arm I will have no data under number of cigarettes and Arm J will have no data under weight changes

#### 14.2.2 Pharmacokinetic Tables and 14.2.5 Urge to Smoke Tables

Tables 14.2.2.1.1 through 14.2.2.1.8 for unadjusted and Tables 14.2.2.2.1 through 14.2.2.2.8 for baseline-adjusted concentration data and Tables 14.2.5.1.1 through 14.2.5.1.8 for UTS data will be in the following format:

Table 14.2.2.1.1 Unadjusted Plasma Nicotine Concentrations (ng/mL) Following Controlled Use of myblu™ (freebase), Gold Leaf flavor, 2.4% (Product A) (Outcomes Population)

| Subject | Product Use | | | | | | S | ample Time | es (min) - | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Number | Sequence | Product | Pre-use | XX | XX | XX | XX | XX | XX | XX | XX |
| X | XXX | X | BLQ | XX | XX | XX | XX | XX | XX | XX | XX |
| X | XXX | X | BLQ | XX | XX | XX | XX | XX | XX | XX | XX |
| X | XXX | X | BLQ | XX | XX | XX | XX | XX | XX | XX | XX |
| n | | | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| Mean | | | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| CV% | | | | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SEM | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Minimum | | | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| Median | | | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Maximum | | | XX | XX | XX | XX | XX | XX | XX | XX | XX |

For the calculation of summary statistics, values that are below the limit of quantitation (BLQ) of <XX> are treated as 1/2 LLOQ.

<sup>. =</sup> Value missing or not reportable.

#### Notes for Generating the Actual Table:

#### Presentation of Data:

For baseline-adjusted table, Pre-use will be replaced with 0.

Concentrations will be presented to same precision as in bio data.

Summary statistics presentation with respect to the precision of the bio data: n = integer; Mean and Median +1; SD and SEM +2, Min and Max +0, CV% to 1 decimal

#### Programmer Note:

PK Time points are: pre-use and 3, 5, 7, 10, 12, 15, 20, 30, 60, 120 and 180 minutes following the start of product use Please also present the geometric mean and geometric CV around the geometric mean for all concentration tables UTS Time points are: pre-use and 5, 10, 15, 30, 60, and 120 minutes following the start of the fixed product use session and one value for 6 hours after ad libitum session (can be labelled "ad libitum\*" with footnote \*6 hours following the start of ad libitum product use session). Please add column for Day

Program: /CAXXXX/sas\_prg/pksas/pk-conc-tables.sas DDMMYYYY HH:MM
Program: /CAXXXX/sas\_prg/pksas/pk-conc-tables-sig.sas DDMMYYYY HH:MM
Program: /CAXXXX/sas\_prg/pksas/adam conc.sas DDMMYYYY HH:MM
Tables 14.2.2.3.1 through 14.2.2.3.8 (PK) and Tables 14.2.5.2.1 through 14.2.5.2.8 (UTS) will be in the following format:

Table 14.2.2.3.1 Baseline-Adjusted Plasma Nicotine PK Parameters Following Controlled Use of myblu™ (freebase), Gold Leaf flavor, 2.4% (Product A) (Outcomes Population)

| Subject<br>Number | Product Use<br>Sequence | Product | paraml<br>(units) | param2<br>(units) | param3<br>(units) | param4<br>(units) | param5<br>(units) | param6<br>(units) |
|---|---|---|---|---|---|---|---|---|
| X | XXX | X | XXX | X.XX | XXX | XXX | XX.X | X <b>.</b> XXX |
| X | XXX | X | XX.X | X.XX | XXX | XXX | XX.X | X.XXX |
| X | XXX | X | XXX | X.XX | XXX | XXX | XX.X | X.XXX |
| X | XXX | X | XX.X | X.XX | XXX | XXX | XX.X | X.XXX |
| X | XXX | X | XX.X | X.XX | XXX | XXX | XX.X | X.XXX |
| X | XXX | X | X.XX | X.XX | XXX | XXX | XX.X | X.XXX |
| X | XXX | X | XXX | X.XX | XXX | XXX | XX.X | X.XXX |
| n | | | XX | XX | XX | XX | XX | XX |
| Mean | | | XXX.X | X.XXX | XXX.X | XXX.X | XX.XX | X.XXXX |
| SD | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| CV% | | | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SEM | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Minimum | | | XX.X | X.XX | XXX | XXX | XX.X | X.XXX |
| Median | | | XX.XX | X.XXX | XXX.X | XXX.X | XX.XX | X.XXXX |
| Maximum | | | XXX | X.XX | XXX | XXX | XX.X | X.XXX |
| Geom Mean | | | XXX.X | X.XXX | XXX.X | XXX.X | XX.XX | X.XXXX |
| Geom CV% | | | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |

. = Value missing or not reportable.

#### Notes for Generating the Actual Table:

#### Presentation of Data:

- PK Parameters will be presented in the following order and with following units: AUCO-t (ng\*min/mL), Cmax (ng/mL), Tmax (min)
- UTS Parameters will be presented in the following order and with the following units: Emax R, TEmax (min), AUECO-120 R
- n will be presented as an integer (with no decimal);
- Parameter values for exposure based parameters (i.e. AUCO-t and Cmax) will be presented with, at maximum, the precision of the bio data, and, at minimum, 3 significant figures (to be determined by the PKist once bio data are received). Summary statistics for exposure parameters will be presented as: Mean, Median, and Geom Mean+1; SD and SEM +2, Min and Max +0.
- Values for time-based parameters (i.e. Tmax) will be presented with 2 decimals. Summary statistics for time-based parameters will be presented as: Mean, Median, and Geom Mean +1; SD +2, Min and Max +0 (omit Geom mean for UTS tables).
- CV% and Geom CV% for all parameters will be presented with 1 decimal (please omit Geom CV% for UTS tables)
- Summarize by overall, female, male
- Add column for Day

Program: /CAXXXX/sas\_prg/pksas/pk-tables.sas DDMMYYYYY HH:MM
Program: /CAXXXXX/sas\_prg/pksas/adam\_pkparam.sas DDMMMYYYY HH:MM

### Clinical Study Report No. CA22736

### Tables 14.2.2.4.1 and 14.2.2.4.2 (PK) and Tables 14.2.5.3.1 and 14.2.5.3.2 (UTS) will be in the following format:

Table 14.2.2.4.1 Statistical Comparisons of Baseline-Adjusted Plasma Nicotine PK Parameters Among myblu™ Products A, B, C, and D Following Controlled Use (Outcomes Population)

| Comparison | Parameter | | metric<br>Means<br>Reference (n) | % Geometric<br>LS Mean Ratio<br>(Test/Reference) | Confidence Intervals<br>(95% Confidence) | p-value |
|---|---|---|---|---|---|---|
| Product A vs Product B | AUCO-t | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXX |
| | Cmax | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXX |
| Product A vs Product C | AUCO-t | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXX |
| | Cmax | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXX |
| Product A vs Product D | AUCO-t | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXX |
| | Cmax | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXX |
| Product B vs Product C | AUCO-t | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXX |
| | Cmax | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXX |
| Product B vs Product D | AUCO-t | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXX |
| | Cmax | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXX |
| Product C vs Product D | AUCO-t | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXX |
| | Cmax | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXX |

Test = The first product in the comparison; Reference = The second product in the comparison n = Number of observations used in the analysis

Product A = < > Product B = < >

Product C = < > Product D = < >

Parameters are log-transformed prior to analysis. Geometric least-squares means (LS Means) are calculated by exponentiating the LS Means from the ANOVA. % Geometric LS Mean Ratio = 100\* (Test Product/Reference Product)

Program: /CAXXXXX/sas prg/pksas PROGRAMNAME.SAS DDMMMYYYY HH:MM

Analyst note: UTS table will based on untransformed data (ie LS means, differences, CIs and p-value)

### Tables 14.2.2.4.3 and 14.2.2.4.4 will be in the following format:

Table 14.2.2.4.3 Nonparametric Statistical Comparisons of Plasma Nicotine PK Parameter Tmax Among myblu $^{\text{TM}}$  Products A, B, C, and D following Controlled Use (Outcomes Population)

| Comparison | Test (n) | Reference (n) | Differen<br>95% CI | ce Test-Refe<br>Median | erence<br>p-Value |
|---|---|---|---|---|---|
| Product A vs Product B | X.XX (X) | X.XX (X) | x.xx - x.xx | X.XX | X.XXX |
| Product A vs Product C | X.XX (X) | X.XX (X) | X.XX - X.XX | X.XX | X.XXXX |
| Product A vs Product D | X.XX (X) | X.XX (X) | X.XX - X.XX | X.XX | X.XXXX |
| Product B vs Product C | $X_{\bullet}XX$ (X) | X.XX (X) | X.XX - X.XX | X.XX | X.XXXX |
| Product B vs Product D | X.XX (X) | X.XX (X) | X.XX - X.XX | X.XX | X.XXXX |
| Product C vs Product D | X.XX (X) | X.XX (X) | X.XX - X.XX | X.XX | X.XXXX |

\_\_\_\_\_\_

Test = The first product in the comparison; Reference = The second product in the comparison n = Number of observations used in the analysis

Product A = < >
Product B = < >
Product C = < >
Product D = < >

p-values are from Wilcoxon signed rank test.

Program: /CAXXXXV/ECR/sas\_prg/pksas/PROGRAMNAME.SAS DDMMMYYYY HH:MM

#### 14.3 Biomarker Tables

Summary tables for blood biomarkers (Part 1) will be in the following format:


Table 14.2.3.1.1 Summary of Blood COHb (% saturation) by Study Day in Part 1: 9-Day Switch to Exclusive myblu™ Use (Outcomes Population)

| Statistic | Day -1 | Day 9 | Change | Percent Change |
|-----------|--------|-------|--------|----------------|
| n | Х | X | X | X |
| Mean | X.X | X.X | X.X | X.X |
| SD | X.XX | X.XX | X.XX | X.XX |
| CV (%) | XX.X | XX.X | XX.X | XX.X |
| SEM | X.XX | X.XX | X.XX | X.XX |
| Minimum | XX | XX | XX | XX |
| Median | X.X | X.X | X.X | X.X |
| Maximum | XX | XX | XX | XX |

Note: Change = Day 9 - Day -1; percent change = (Day 9 - Day -1)/Day -1\*100

Program: /CAXXXXX/sas prg/pksas PROGRAMNAME.SAS DDMMMYYYY HH:MM

Programming Notes: Footnotes to include under the table, as appropriate: <. = Value missing or not reportable. > <For the calculation of summary statistics, values that are below the limit of quantitation (BLQ) of <XX> are treated as 1/2 LLOQ>. Summarize by Overall, female, male

Summary tables for urine biomarkers (Part 1) will be in the following format:


Table 14.2.3.1.2 Summary of Urine NNAL by Study Day in Part 1: 9-Day Switch to Exclusive myblu™ Use (Outcomes Population)

| Statistic | <br>Day -1 | Amount Excreted Day 9 | | hours) Percent Change |
|---|---|---|---|---|
| n | X | X | X | X |
| Mean | X.X | X.X | X.X | X.X |
| SD | X.XX | X.XX | X.XX | X.XX |
| CV (%) | XX.X | XX.X | XX.X | XX.X |
| SEM | X.XX | X.XX | X.XX | X.XX |
| Minimum | XX | XX | XX | XX |
| Median | X.X | X.X | X.X | X.X |
| Maximum | XX | XX | XX | XX |

Note: Change = Day 9 - Day -1; percent change = (Day 9 - Day -1)/Day -1\*100

Program: /CAXXXXX/sas prg/pksas PROGRAMNAME.SAS DDMMMYYYY HH:MM

Programming Notes: Add four columns with the header "Creatinine-Adjusted (unit/g creatinine)" Footnotes to include under the table, as appropriate: <. = Value missing or not reportable. > <For the calculation of summary statistics, values that are below the limit of quantitation (BLQ) of <XX> are treated as 1/2 LLOQ>. Summarize by Overall, female, male.

Statistical comparison table for Part 1 will be in the following format:


Table 14.2.3.1.22 Statistical Comparisons of BoE and BoPH Between Study Days in Part 1: 9-Day Switch to Exclusive myblu™ Use (Outcomes Population)

| Biomarker (unit) | LS M<br>Day 9(n) | Day -1 (n) | LS Mean Difference<br>(Day 9 - Day -1) | 95% Confidence Interval | p-value |
|---|---|---|---|---|---|
| Blood COHb (% Saturation)<br>Urine NNAL (xg/24 hours) | X.XX (X)<br>X.XX (X) | X.XX (X)<br>X.XX (X) | XXX.XX<br>XXX.XX | XX.XX - XXX.XX<br>XX.XX - XXX.XX | X.XXXX<br>X.XXXX |
| <pre><add biomarkers="" remaining=""></add></pre> | | | | | |

Note: n = Number of observation used in the analysis; Least-squares means (LS Means) are calculated from the ANOVA.

Program: /CAXXXX/sas prg/pksas PROGRAMNAME.SAS DDMMYYYYY HH:MM

Programming Notes: List biomarkers in the same order as section 2.2

Summary tables for blood biomarkers by Study Day (Part 2) will be in the following format:


Table 14.2.3.2.1 Summary of Blood COHb (% Saturation) by Study Day in Part 2: Continue Exclusive myblu™ Use (Outcomes Population)

| Statistic | Day -1 | Day 14 | Change | Percent Change |
|-----------|--------|--------|--------|----------------|
| n | X | X | X | X |
| Mean | X.X | X.X | X.X | X.X |
| SD | X.XX | X.XX | X.XX | X.XX |
| CV (%) | XX.X | XX.X | XX.X | XX.X |
| SEM | X.XX | X.XX | X.XX | X.XX |
| Minimum | XX | XX | XX | XX |
| Median | X.X | X.X | X.X | X.X |
| Maximum | XX | XX | XX | XX |

Note: Change = Day 14 - Day -1; percent change = (Day 14 - Day -1)/Day -1\*100

Program: /CAXXXXX/sas prg/pksas PROGRAMNAME.SAS DDMMMYYYY HH:MM

Programming Notes: Add four columns for with the header "Creatinine-Adjusted unit/g creatinine" Footnotes to include under the table, as appropriate: < . = Value missing or not reportable. > <For the calculation of summary statistics, values that are below the limit of quantitation (BLQ) of <XX> are treated as 1/2 LLOQ>. Summarize by Overall, female, male

Summary tables for urine biomarkers by Study Day (Part 2) will be in the following format:


Table 14.2.3.2.2 Summary of Urine NNAL by Study Day in Part 2: Continue Exclusive myblu™ Use (Outcomes Population)

| Statistic | <br>Day -1 | Amount Excre<br>Day 14 | ted (xg/24 hou: | rs)<br>cent Change |
|---|---|---|---|---|
| n | X | X | X | X |
| Mean | X.X | X.X | X.X | X.X |
| SD | X.XX | X.XX | X.XX | X.XX |
| CV (%) | XX.X | XX.X | XX.X | XX.X |
| SEM | X.XX | X.XX | X.XX | X.XX |
| Minimum | XX | XX | XX | XX |
| Median | X.X | X.X | X.X | X.X |
| Maximum | XX | XX | XX | XX |

Note: Change = Day 14 - Day -1; percent change = (Day 14 - Day -1)/Day -1\*100

Program: /CAXXXXX/sas prg/pksas PROGRAMNAME.SAS DDMMMYYYY HH:MM

Programming Notes: Add four columns for with the header "Creatinine-Adjusted unit/g creatinine" Footnotes to include under the table, as appropriate: <. = Value missing or not reportable. > <For the calculation of summary statistics, values that are below the limit of quantitation (BLQ) of <XX> are treated as 1/2 LLOQ>. Summarize by Overall, female, male

Statistical comparison table of biomarkers between study days for Part 2 will be in the following format:


Table 14.2.3.2.22 Statistical Comparison of BoE and BoPH Between Study Days in Part 2: Continue Exclusive myblu™ Use (Outcomes Population)

| Biomarker (unit) | LS Mea<br>Day 14(n) | - | LS Mean Difference<br>(Day 14 - Day -1) | 95% Confidence Interval | p-value |
|---|---|---|---|---|---|
| Blood COHb (% Saturation)<br>Urine NNAL (xg/24 hours) | X.XX (X)<br>X.XX (X) | X.XX (X)<br>X.XX (X) | XXX.XX<br>XXX.XX | XX.XX - XXX.XX<br>XX.XX - XXX.XX | X.XXXX<br>X.XXXX |
| <pre><add biomarkers="" remaining=""></add></pre> | | | | | |

Note: n = Number of observation used in the analysis; Least-squares means (LS Means) are calculated from the ANOVA.

Program: /CAXXXX/sas prg/pksas PROGRAMNAME.SAS DDMMMYYYY HH:MM

Programming Notes: List biomarkers in the same order as section 2.2

### Summary tables for blood biomarkers by Study Arm and Study Day (Part 2) will be in the following format:


Table 14.2.3.3.1 Summary of Blood COHb (% Saturation) by Study Arm in Part 2 (Outcomes Population)

| | Arm | Statistic | Day 9 | Day 14 | Change | Percent Change |
|---------|-----|-----------|-------|--------|--------|----------------|
| Overall | I | n | X | X | X | X |
| | | Mean | X.X | X.X | X.X | X.X |
| | | SD | X.XX | X.XX | X.XX | X.XX |
| | | CV (%) | XX.X | XX.X | XX.X | XX.X |
| | | SEM | X.XX | X.XX | X.XX | X.XX |
| | | Minimum | XX | XX | XX | XX |
| | | Median | X.X | X.X | X.X | X.X |
| | | Maximum | XX | XX | XX | XX |
| | J | n | X | X | X | X |
| | | Mean | X.X | X.X | X.X | X.X |
| | | SD | X.XX | X.XX | X.XX | X.XX |
| | | CV (%) | XX.X | XX.X | XX.X | XX.X |
| | | SEM | X.XX | X.XX | X.XX | X.XX |
| | | Minimum | XX | XX | XX | XX |
| | | Median | X.X | X.X | X.X | X.X |
| | | Maximum | XX | XX | XX | XX |
| | K | n | X | X | X | X |
| | | Mean | X.X | X.X | X.X | X.X |
| | | SD | X.XX | X.XX | X.XX | X.XX |
| | | CV (%) | XX.X | XX.X | XX.X | XX.X |
| | | SEM | X.XX | X.XX | X.XX | X.XX |
| | | Minimum | XX | XX | XX | XX |
| | | Median | X.X | X.X | X.X | X.X |
| | | Maximum | XX | XX | XX | XX |

Female <Same as above>

Male <Same as above>

\_\_\_\_\_\_

Note: Change = Day 14 - Day 9; percent change = (Day 14 - Day 9)/Day 9\*100

Arm I: Exclusive use of myblu™ products ad libitum

Arm J: Exclusive smoking of usual brand combustible cigarettes ad libitum

Arm K: Smoking of usual brand combustible cigarettes (up to 50% of the subject's self-reported CPD) and use of myblu™ products ad libitum

Programming Notes: Footnotes to include under the table, as appropriate: < . = Value missing or not reportable. > <For the calculation of summary statistics, values that are below the limit of quantitation (BLQ) of <XX> are treated as 1/2 LLOQ>.

### Summary tables for urine biomarkers by Study Arm and Study Day (Part 2) will be in the following format:


| Table 14.2.3.3.2 | Summary | of IIrine | MNAT. by | Study Arm | in | Part 2. | (Outcomes | Population) |
|---|---|---|---|---|---|---|---|---|

| | Arm | Statistic | Day 9 | Amount Excreted Day 14 | | )<br>Percent Change |
|---|---|---|---|---|---|---|
| Overall | I | n | X | | X | X |
| | | Mean | X.X | | X.X | X.X |
| | | SD | X.XX | | X.XX | X.XX |
| | | CV (%) | XX.X | | XX.X | XX.X |
| | | SEM | X.XX | | X.XX | X.XX |
| | | Minimum | XX | | XX | XX |
| | | Median | X.X | | X.X | X.X |
| | | Maximum | XX | XX | XX | XX |
| | J | n | X | X | X | X |
| | | Mean | X.X | X.X | X.X | X.X |
| | | SD | X.XX | X.XX | X.XX | X.XX |
| | | CV (%) | XX.X | XX.X | XX.X | XX.X |
| | | SEM | X.XX | X.XX | X.XX | X.XX |
| | | Minimum | XX | XX | XX | XX |
| | | Median | X.X | X.X | X.X | X.X |
| | | Maximum | XX | XX | XX | XX |
| | K | n | X | X | X | Х |
| | | Mean | X.X | X.X | X.X | X.X |
| | | SD | X.XX | | X.XX | X.XX |
| | | CV (%) | XX.X | | XX.X | XX.X |
| | | SEM | X.XX | | X.XX | X.XX |
| | | Minimum | XX | | XX | XX |
| | | Median | X.X | | X.X | X.X |
| | | Maximum | XX | | XX | XX |

Female <Same as above>

Male <Same as above>

Note: Change = Day 14 - Day 9; percent change = (Day 14 - Day 9)/Day 9\*100

Arm I: Exclusive use of myblu™ products ad libitum

Arm J: Exclusive smoking of usual brand combustible cigarettes ad libitum

Arm K: Smoking of usual brand combustible cigarettes (up to 50% of the subject's self-reported CPD) and use of myblu™ products ad libitum

Program: /CAXXXX/sas prg/pksas PROGRAMNAME.SAS DDMMMYYYY HH:MM

Programming Notes: Add four columns for with the header "Creatinine-Adjusted unit/g creatinine" Footnotes to include under the table, as appropriate: < . = Value missing or not reportable. > <For the calculation of summary statistics, values that are below the limit of quantitation (BLQ) of <XX> are treated as 1/2 LLOQ>.

### Statistical comparison tables of biomarkers among study arms for Part 2 will be in the following format:


Table 14.2.3.3.22 Statistical Comparisons of BoE and BoPH Differences From Baseline Among myblu™, Combustible Cigarette, and Dual Use Arms in Part 2 (Outcomes Population) (Outcomes Population)

| Biomarker (unit) | Comparison | _ | eans<br>Day 9(n) | LS Mean Difference<br>(Day 14 - Day 9) | 95% Confidence Interval | p-value |
|---|---|---|---|---|---|---|
| Blood COHb (% Saturation) | Arm I vs Arm J<br>Arm I vs Arm K<br>Arm K vs Arm J | X.XX (X)<br>X.XX (X)<br>X.XX (X) | X.XX (X)<br>X.XX (X)<br>X.XX (X) | XXX.XX<br>XXX.XX<br>XXX.XX | XX.XX - XXX.XX<br>XX.XX - XXX.XX<br>XX.XX - XXX.XX | X.XXXX<br>X.XXXX<br>X.XXXX |
| Urine NNAL (xg/24 hours) | <same above<="" as="" td=""><td>for the rema</td><td>ining biomark</td><td>ers</td><td></td><td></td></same> | for the rema | ining biomark | ers | | |

Note: n = Number of observation used in the analysis; Least-squares means (LS Means) are calculated from the ANOVA.

Program: /CAXXXX/sas prg/pksas PROGRAMNAME.SAS DDMMYYYYY HH:MM

#### Programming Notes: List biomarkers in the same order as section 2.2

Arm I: Exclusive use of  $myblu^{m}$  products ad libitum

Arm J: Exclusive smoking of usual brand combustible cigarettes ad libitum

Arm K: Smoking of usual brand combustible cigarettes (up to 50% of the subject's self-reported CPD) and use of myblu™ products ad libitum

### 4.2.4 <u>Physiologic Assessments Tables</u> Tables 14.2.4.1.1, 14.2.4.1.2, 14.2.4.1.4, 14.2.4.1.5, 14.2.4.1.7, 14.2.4.1.8 will be in the following format:

Table 14.2.4.1.1 Summary of Systolic Blood Pressure (mm Hg) by Time Point in Exclusive myblu™ Use (Arm I) (Outcomes Population)

| | Sample Times (hr) | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Day | Pre-use | XX | XX | XX | XX | XX | XX | XX | XX |
| -1 n | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| CV% | | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SEM | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Minimum | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Maximum | XX | XX | XX | XX | XX | XX | XX | XX | XX |

Repeat for Days 9 and 14

Programmer note: For change from baseline tables, present values for Day 9 – Day -1 and Day 14 – Day -1

<sup>. =</sup> Value missing or not reportable.

### Tables 14.2.4.1.3, 14.2.4.1.6, and 14.2.4.1.9 will be in the following format:

Table 14.2.4.1.3 Summary of Systolic Blood Pressure Change from Baseline Parameters in Exclusive myblu™ Use (Arm I) (Outcomes Population)

| Day | Statistic | paraml<br>(units) | param2<br>(units) | param3<br>(units) | param4<br>(units) | param5<br>(units) | param6<br>(units) |
|---|---|---|---|---|---|---|---|
| 9 | n | XX | XX | XX | XX | XX | XX |
| | Mean | XXX.X | X.XXX | XXX.X | XXX.X | XX.XX | X.XXXX |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | CV% | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SEM | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Minimum | XX.X | X.XX | XXX | XXX | XX.X | X.XXX |
| | Median | XX.XX | X.XXX | XXX.X | XXX.X | XX.XX | X.XXXX |
| | Maximum | XXX | X.XX | XXX | XXX | XX.X | X.XXX |

14 (same as above)

#### Notes for Generating the Actual Table:

Presentation of Data:

- Parameters will be presented in the following order and with following units: AUECO-24 (mm Hg \* hr), Emax (mm hg), TEmax (min)
- n will be presented as an integer (with no decimal);
- Parameter values for exposure-based parameters (i.e. AUCO-t and Cmax) will be presented with, at maximum, the precision of the bio data, and, at minimum, 3 significant figures (to be determined by the PKist once bio data are received). Summary statistics for exposure parameters will be presented as: Mean, Median, +1; SD and SEM +2, Min and Max +0.
- Values for time-based parameters (i.e. TEmax) will be presented with 2 decimals. Summary statistics for time-based parameters will be presented as: Mean, Median, SD +2, Min and Max +0.
- Summarize by overall, female, male

Program: /CAXXXXX/sas prg/pksas/pk-tables.sas DDMMMYYYY HH:MM

<sup>. =</sup> Value missing or not reportable.


Table 14.2.4.1.10 Statistical Comparisons of Change From Baseline Systolic Blood Pressure, Diastolic Blood Pressure, and Heart Rate Heart Rate Parameters in Exclusive myblu™ Use (Arm I)

| Vital Sign | Parameter (unit) | _ | eans<br>Day 9(n) | LS Mean Difference<br>(Day 14 - Day 9) | 95% Confidence Interval | p-value |
|---|---|---|---|---|---|---|
| Systolic BP | AUEC (mmHg * hr) | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| | Emax (mmHg) | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| | TEmax (min) | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |

<Repeat for other vital signs>

Note: n = Number of observation used in the analysis; Least-squares means (LS Means) are calculated from the ANOVA.

Program: /CAXXXXX/sas\_prg/pksas PROGRAMNAME.SAS DDMMMYYYY HH:MM

Program: /CAXXXX/sas\_prg/pksas/adam\_pkparam.sas DDMMMYYYY HH:MM


Table 14.2.4.2.1 Summary of Lung Function Parameters by Time Point in Exclusive myblu™ Use (Arm I) (Outcomes Population)

| Parameter: | Statistics | Day -1 | Day 9 | Day -1 | Day 14 |
|---|---|---|---|---|---|
| ====================================== | n | X | X | X | X |
| | Mean | X.X | X.X | X.X | X.X |
| | SD | X.XX | X.XX | X.XX | X.XX |
| | CV (%) | XX.X | XX.X | XX.X | XX.X |
| | Minimum | XX | XX | XX | XX |
| | Median | X.X | X.X | X.X | X.X |
| | Maximum | XX | XX | XX | XX |
| FEV1 (post) | n | X | X | X | X |
| | Mean | X.X | X.X | X.X | X.X |
| | SD | X.XX | X.XX | X.XX | X.XX |
| | CV (%) | XX.X | XX.X | XX.X | XX.X |
| | Minimum | XX | XX | XX | XX |
| | Median | X.X | X.X | X.X | X.X |
| | Maximum | XX | XX | XX | XX |

FEV1 (Post - Pre)

<Continue with remaining parameters>

Note: \*Parameters values are are the percent of predicted

. = Value missing or not reportable.

Program: /CAXXXXX/sas\_prg/pksas PROGRAMNAME.SAS DDMMYYYYY HH:MM

Programmer note: Parameters are pre-, post-, and pre-post bronchodilator values for percent of predicted FEV1, FVC, FEV1:FVC ratio, and FEF25-25%


Table 14.2.4.2.2 Summary of Lung Function Variables Changes by Time Point in Exclusive myblu™ Use (Arm I) (Outcomes Population)

| Parameter: | Statistics | Day 9 - Day -1 | codilator<br>Day 14 - Day -1 |
|------------|------------|----------------|------------------------------|
| EV1 (%) | n | X | X |
| | Mean | X.X | X.X |
| | SD | X.XX | X.XX |
| | CV (%) | XX.X | XX.X |
| | Minimum | XX | XX |
| | Median | X.X | X.X |
| | Maximum | XX | XX |
| | n | X | X |
| | Mean | X.X | X.X |
| | SD | X.XX | X.XX |
| | CV (%) | XX.X | XX.X |
| | Minimum | XX | XX |
| | Median | X.X | X.X |
| | Maximum | XX | XX |

\*Parameters values are are the percent of predicted Note:

. = Value missing or not reportable.

Program: /CAXXXX/sas prg/pksas PROGRAMNAME.SAS DDMMMYYYY HH:MM

Programmer note: Parameters percent of predicted FEV1, FVC, FEV1:FVC, and FEF25-25%. Add the same two columns for "Post Bronchodilator – Pre-Bronchodilator". Present results for Overall, Female, Male


Table 14.2.4.2.3 Statistical Comparisons of Change From Baseline Lung Function Parameters in Exclusive myblu™ Use (Arm I)

| Parameter* | (unit) | LS N<br>Day 14 (n) | Means<br>Day 9(n) | LS Mean Difference<br>(Day 14 - Day 9) | 95% Confidence Interval | p-value |
|---|---|---|---|---|---|---|
| Pre-Bronchodi | llator | | | | | |
| FEV1 (%) | | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| FVC (%) | | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| FEV1:FVC | | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| FEF25-75% | | | | | | |
| Post-Bronchoo | dilator - Pre-B | ronchodilato | r. | | | |
| FEV1 (%) | | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| FVC (%) | | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| FEV1:FVC | | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| FEF25-75% | | | | | | |

\_\_\_\_\_\_

Note: \*Parmeters are percent of predicted

Program: /CAXXXXX/sas\_prg/pksas PROGRAMNAME.SAS DDMMMYYYY HH:MM
Program: /CAXXXXX/sas\_prg/pksas/adam pkparam.sas DDMMMYYYY HH:MM

n = Number of observation used in the analysis; Least-squares means (LS Means) are calculated from the ANOVA.

### **14.2.6 Questionnaires Tables**

### Tables 14.2.6.1.X and 14.2.6.2.X will be in the following format:


Table 14.2.6.1 Summary of < PES Subscales> by Study Product for Controlled Product Use Session (Outcomes Population)

| | | | Product | | | | | |
|---|---|---|---|---|---|---|---|---|
| < Subscale of Question> | or | Statistic | А | В | С | D | E | F |
| Satisfaction | Overall | n | X | Х | X | X | X | X |
| | | Mean | X.X | X.X | X.X | X.X | X.X | X.X |
| | | SD | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| | | CV% | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | SEM | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| | | Minimum | XX | XX | XX | XX | XX | XX |
| | | Median | X.X | X.X | X.X | X.X | X.X | X.X |
| | | Maximum | XX | XX | XX | XX | XX | XX |
| | Female | n | X | X | X | X | X | Х |
| | | Mean | X.X | X.X | X.X | X.X | X.X | X.X |
| | | SD | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| | | CV% | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | SEM | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| | | Minimum | XX | XX | XX | XX | XX | XX |
| | | Median | X.X | X.X | X.X | X.X | X.X | X.X |
| | | Maximum | XX | XX | XX | XX | XX | XX |
| | Male | n | X | X | Х | Х | X | Х |
| | | Mean | X.X | X.X | X.X | X.X | X.X | Х.Х |
| | | SD | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| | | CV% | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | SEM | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| | | Minimum | XX | XX | XX | XX | XX | XX |
| | | Median | X.X | X.X | Х.Х | X.X | Х.Х | Х.Х |
| | | Maximum | XX | XX | XX | XX | XX | XX |

Programmer note: Add columns for Products G, and H.

### Tables 14.2.6.3.1 and 14.2.6.3.2 will be in the following format:

Page 1 of X Table 14.2.6.3.1 Frequency of Responses to Use the Product Again Questionnaire in Each Category After the Ad Libitum Product Use Episode by Product (Outcome Population)

| Question | Product | Category | Statistics | | oduct Again Respo<br>0 | nse Category<br>>0 to 50 |
|---|---|---|---|---|---|---|
| 1 | A | Female | n (%)<br>n (%)<br>n (%) | XX (XX%)<br>XX (XX%)<br>XX (XX%) | XX (XX%)<br>XX (XX%)<br>XX (XX%) | XX (XX%)<br>XX (XX%)<br>XX (XX%) |
| | В | Female | n (%)<br>n (%)<br>n (%) | | XX (XX%)<br>XX (XX%)<br>XX (XX%) | XX (XX%)<br>XX (XX%)<br>XX (XX%) |
| | С | | n (%) | XX (XX%) | XX (XX%)<br>XX (XX%)<br>XX (XX%) | |
| | D | | n (%) | XX (XX%) | XX (XX%)<br>XX (XX%)<br>XX (XX%) | |
| | E | | n (응)<br>n (응)<br>n (응) | XX (XX%) | XX (XX%)<br>XX (XX%)<br>XX (XX%) | |
| | F | Overall<br>Female<br>Male | | XX (XX%)<br>XX (XX%)<br>XX (XX%) | XX (XX%)<br>XX (XX%)<br>XX (XX%) | XX (XX%)<br>XX (XX%)<br>XX (XX%) |
| | G | Overall<br>Female<br>Male | n (%)<br>n (%)<br>n (%) | XX (XX%)<br>XX (XX%)<br>XX (XX%) | XX (XX%)<br>XX (XX%)<br>XX (XX%) | XX (XX%)<br>XX (XX%)<br>XX (XX%) |
| | Н | Overall<br>Female<br>Male | n (%)<br>n (%)<br>n (%) | XX (XX%)<br>XX (XX%)<br>XX (XX%) | XX (XX%)<br>XX (XX%)<br>XX (XX%) | XX (XX%)<br>XX (XX%)<br>XX (XX%) |
| 2 | <repe< td=""><td>at for quest</td><td>tions 2 and 3&gt;</td><td>&gt;</td><td></td><td></td></repe<> | at for quest | tions 2 and 3> | > | | |

Question 1: How likely are you to continue to smoke after you complete this study?
Question 2: If available, how likely are you to buy your assigned study product in the future?
Question 3: How likely are you to buy an e-cigarette other than your assigned product in the future?

### Nerudia Ltd.

### NER 01/003 *my*blu™ E-cigarettes

### Clinical Study Report No. CA22736

```
Product A = <>
Product B = <>
Product C = <>
Product D = <>
Product E = <>
Product F = <>
Product G = <>
Product H = <>
```

Program: /CAXXXXX/sas\_prg/pksas/PROGRAMNAME.SAS DDMMMYYYY HH:MM

Programming Note: The percentage (%) is the row percentage.

### Tables 14.2.6.3.3 and 14.2.6.3.4 will be in the following format:

Page 1 of X Table 14.2.6.3.3 Summary of Future Intent to Use VAS Score in Each Category by Study Product for Ad Libitum Product Use Session (Outcomes Population)

| Question | Product | Category | Use<br>Statistics | e the Product Again | n Response Category<br>>0 to 50 |
|---|---|---|---|---|---|
| 1 | A | Overall | n<br>Mean<br>SD<br>CV(%)<br>SEM<br>Minimum<br>Median<br>Maximum | X<br>X.X<br>X.XX<br>XX.X<br>X.XX<br>XX<br>XX<br>XX | X<br>X.X<br>X.XX<br>XX.X<br>X.XX<br>XX<br>XX<br>XX<br>XX |
| | | Female | n<br>Mean<br>SD<br>CV(%)<br>SEM<br>Minimum<br>Median<br>Maximum | X<br>X.X<br>X.XX<br>XX.X<br>X.XX<br>XX<br>XX<br>XX | X<br>X.X<br>X.XX<br>XX.X<br>X.XX<br>XX<br>XX<br>XX<br>XX |
| | | Male | n<br>Mean<br>SD<br>CV(%)<br>SEM<br>Minimum<br>Median<br>Maximum | X<br>X.X<br>X.XX<br>XX.X<br>X.XX<br>XX<br>XX<br>XX | X<br>X.X<br>X.XX<br>XX.X<br>X.XX<br>XX<br>XX<br>XX<br>XX |

Question 1: How likely are you to continue to smoke after you complete this study?

Question 2: If available, how likely are you to buy your assigned study product in the future?

Question 3: How likely are you to buy an e-cigarette other than your assigned product in the future?

Product A = <>

Product B = <>

Product C = <>

Product D = <>

Product E = <>

Product F = <>

Product G = <>

Product H = <>

Programming Note: Summary for Products B, C, D, E, F, G, and H will also be included in the table. Include category 0 in the table if there sufficient data.

### Tables 14.2.6.3.5 and 14.2.6.3.6 will be in the following format:

Page 1 of X Table 14.2.6.3.5 Summary of Future Intent to Use VAS Raw Scores by Study Product for Ad Libitum Product Use Session (Outcomes Population)

| | | Product | | | |
|----------|------------|---------|------|------|------|
| Category | Statistics | А | В | С | D |
| Overall | n | X | X | X | X |
| | Mean | X.X | X.X | X.X | X.X |
| | SD | X.XX | X.XX | X.XX | X.XX |
| | CV (%) | XX.X | XX.X | XX.X | XX.X |
| | SEM | XX.X | XX.X | XX.X | XX.X |
| | Minimum | XX | XX | XX | XX |
| | Median | X.X | X.X | X.X | Х. |
| | Maximum | XX | XX | XX | XX |
| Female | n | X | X | X | X |
| | Mean | X.X | X.X | X.X | X.X |
| | SD | X.XX | X.XX | X.XX | X.XX |
| | CV (%) | XX.X | XX.X | XX.X | XX.X |
| | SEM | XX.X | XX.X | XX.X | XX.X |
| | Minimum | XX | XX | XX | XX |
| | Median | X.X | X.X | X.X | Х. |
| | Maximum | XX | XX | XX | XX |

Question 1: How likely are you to continue to smoke after you complete this study?

Question 2: If available, how likely are you to buy your assigned study product in the future? Question 3: How likely are you to buy an e-cigarette other than your assigned product in the future?

Product A = <>

Product B = <>

Product C = <>

Product D = <>

Product E = <>

Product F = <> Product G = <>

Product H = <>

Program: /CAXXXXX/sas prg/pksas/PROGRAMNAME.SAS DDMMMYYYY HH:MM

Programmer Note: Summary for Male and Products E, F, G, H will be included in the table. Add a column to the left for "Question"


### Tables 14.2.6.4, 14.2.6.5, and 14.2.6.6 will be in the following format:

Table 14.2.6.6 Summary of QSU-brief Factor Scores by Study Arm and Study Day (Outcomes Population)

| | | | | Day 9 | |
|----------|---------|-----------|-------|-------|-------|
| Subscale | | Statistic | Arm I | Arm J | Arm K |
| Factor 1 | Overall | n | X | Х | Х |
| | | Mean | X.X | X.X | X.X |
| | | SD | X.XX | X.XX | X.XX |
| | | CV% | XX.X | XX.X | XX.X |
| | | SEM | X.XX | X.XX | X.XX |
| | | Minimum | XX | XX | XX |
| | | Median | X.X | X.X | X.X |
| | | Maximum | XX | XX | XX |
| | Female | n | X | X | X |
| | | Mean | X.X | X.X | X.X |
| | | SD | X.XX | X.XX | X.XX |
| | | CV% | XX.X | XX.X | XX.X |
| | | SEM | X.XX | X.XX | X.XX |
| | | Minimum | XX | XX | XX |
| | | Median | X.X | X.X | X.X |
| | | Maximum | XX | XX | XX |
| | Male | n | X | X | Х |
| | | Mean | X.X | X.X | X.X |
| | | SD | X.XX | X.XX | X.XX |
| | | CV% | XX.X | XX.X | XX.X |
| | | SEM | X.XX | X.XX | X.XX |
| | | Minimum | XX | XX | XX |
| | | Median | X.X | X.X | X.X |
| | | Maximum | XX | XX | XX |

< Repeat for Factor 2>

\_\_\_\_\_\_

### Nerudia Ltd. NER 01/003 *my*blu™ E-cigarettes

### Clinical Study Report No. CA22736

Arm I =

Factor 1 = Anticipation of pleasure from smoking

Factor 2 = Anticipation of Relief of nicotine withdrawal

Scale: 1 = Strongly disagree; 7 = Strongly agree

Program: /AAXXXXX/ECR/sas\_prg/stsas/tab programname.sas DDMMMYYYY HH:MM

### Programmer note: Add columns for Day 14. Tables 14.2.6.4 and 14.2.6.5 will have no subscale column.

Footnote for Table 14.2.6.4: Total scoring: 0 - 3 = not dependent, 4 - 8 = low dependence, 9 - 12 = medium dependence, 13+ = high dependence


Table 14.2.7 Summary of Puff Topography Parameters by Study Day (Outcomes Population)

| Parameter (Units) | Category | Statistics | Day -1 | Day 1 | Day 8 |
|---|---|---|---|---|---|
| Total Puff Count | Overall | n | X | X | Х |
| | | Mean | X.X | X.X | X.X |
| | | SD<br>CV(%)<br>SEM | X.XX<br>XX.X<br>XX.X | X.XX<br>XX.X<br>XX.X | X.XX<br>XX.X<br>XX.X |
| | | Minimum | XX | XX | XX |
| | | Median | X.X | X.X | X.X |
| | | Maximum | XX | XX | XX |
| | Female | n | X | X | X |
| | | Mean | X.X | X.X | X.X |
| | | SD | X.XX | X.XX | X.XX |
| | | CV (%) | XX.X | XX.X | XX.X |
| | | SEM | XX.X | XX.X | XX.X |
| | | Minimum | XX | XX | XX |
| | | Median | X.X | X.X | X.X |
| | | Maximum | XX | XX | XX |

### Programming note: Parameters are:

- Total Puff count
- Average Puff Duration (sec)
- Total Puff Duration sec)
- Average Puff volume (mL)
- Total Puff Volume (mL)
- Average Peak flow rate (mL/sec)
- Average flow rate (mL/sec)
- Average Inter-puff interval (sec)

Adverse event summary table (Tables 14.3.1.1.1 and 14.3.1.2.1) will be in the following format.

Table 14.3.1.1.1 Product Use-emergent Adverse Event Frequency by Study Product - Number of Subjects Reporting the Event
(% of Subjects Who Used Study Product) - Part 1 (Safety Population)

| Product | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Adverse Event* | A | Α | | В | | С | | D | | | F | | G | | Over | all |
| Number of Subjects Who Received Study Product<br>Number of Subjects With Adverse Events<br>Number of Subjects Without Adverse Events | Х ( | X%) | , | XX%) | Х ( | 100%)<br>X%)<br>XX%) | Х ( | X%) | Х ( | X%) | XX (1<br>X (<br>XX (X | X%) | Х ( | X%) | XX (1<br>X (<br>XX (X | X%) |
| Eye disorders Vision blurred | X (<br>X ( | X%)<br>X%) | X (<br>X ( | X%)<br>X%) | X ( | X%)<br>X%) | X (<br>X ( | X%)<br>X%) | X (<br>X ( | X%)<br>X%) | X (<br>X ( | X%)<br>X%) | X (<br>X ( | X%)<br>X%) | X (<br>X ( | X%)<br>X%) |
| Gastrointestinal disorders Dyspepsia Nausea | X (<br>X (<br>X ( | X%)<br>X%)<br>X%) | X (<br>X (<br>X ( | X%)<br>X%)<br>X%) | X (<br>X (<br>X ( | X%)<br>X%)<br>X%) | X (<br>X (<br>X ( | X%)<br>X%)<br>X%) | X (<br>X (<br>X ( | X%)<br>X%)<br>X%) | X (<br>X (<br>X ( | X%)<br>X%)<br>X%) | X (<br>X (<br>X ( | X%)<br>X%)<br>X%) | X (<br>X (<br>X ( | X%)<br>X%)<br>X%) |
| Musculoskeletal and connective tissue disorders | X ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) |
| Back pain<br>Muscle cramps<br>Musculoskeletal pain | X (<br>X (<br>X ( | X%)<br>X%)<br>X%) | X (<br>X (<br>X ( | X%)<br>X%)<br>X%) | X (<br>X (<br>X ( | X%)<br>X%)<br>X%) | X (<br>X (<br>X ( | X%)<br>X%)<br>X%) | X (<br>X (<br>X ( | X%)<br>X%)<br>X%) | X (<br>X (<br>X ( | X%)<br>X%)<br>X%) | X (<br>X (<br>X ( | X%)<br>X%)<br>X%) | X (<br>X (<br>X ( | X%)<br>X%)<br>X%) |
| Nervous system disorders<br>Headache NOS | X (<br>X ( | X응)<br>X응) | X (<br>X ( | X%)<br>X%) | X (<br>X ( | X%)<br>X%) | X (<br>X ( | X용)<br>X용) | X (<br>X ( | X%)<br>X%) | X (<br>X ( | X%)<br>X%) | X (<br>X ( | X%)<br>X%) | X (<br>X ( | X%)<br>X%) |

Note: \* Adverse events are classified according to MedDRA Version 22.0. Product X = < >

Program: /CAXXXXX/sas prg/stsas/tab cdash tblae1a auto.sas DDMMMYYYY HH:MM

Programmer Note: Product H will also be presented in the table. Table 14.3.1.2.1 will have three columns for the three study arms and an overall column.

### Adverse event summary table (Tables 14.3.1.1.2 and 14.3.1.2.2) will be in the following format.


Table 14.3.1.1.2 Product Use-emergent Adverse Event Frequency by Study Product - Number of Adverse Events (% of Total Adverse Events) - Part 1 (Safety Population)

| | Product | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Adverse Event* | | A<br>XX (100%) | | B<br>XX (100%) | | C<br><br>XX (100%) | | D | | | F<br>XX (100%) | | | | Overall<br> | |
| Number of Adverse Events | XX (1 | | | | | | | .00%) | XX (100%) | | | | | | | |
| Eye disorders | X ( | X%) | Х( | X%) | X ( | X%) | Х ( | X%) | X ( | X%) | Х ( | X%) | Х ( | X%) | Х( | X%) |
| Vision blurred | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) |
| Gastrointestinal disorders | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) |
| Dyspepsia | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) |
| Nausea | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) |
| Musculoskeletal and connective tissue | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) |
| disorders | | | | | | | | | | | | | | | | |
| Back pain | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) |
| Muscle cramps | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) |
| Musculoskeletal pain | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) |
| Nervous system disorders | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) |
| Headache NOS | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) |
| Reproductive system and breast disorders | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) |
| Vaginal discharge | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) |

Note: \* Adverse events are classified according to MedDRA Version 22.0. Product X = < >

Program: /CAXXXXX/sas\_prg/stsas/tab cdash\_tblaela\_auto.sas DDMMMYYYY HH:MM

Programmer Note: Product H will also be presented in the table. Table 14.3.1.2.2 will have three columns for the three study arms and an overall column.

### Adverse event summary table (Tables 14.3.1.1.3 and 14.3.1.2.3) will be in the following format.


Product Use-emergent Adverse Event Frequency by Study Product, Severity, and Relationship to Study Product

- Number of Subjects Reporting Events - Part 1 (Safety Population)

| | O.b | Number of | | Inten | sity | Relationship to Study Product | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Adverse Event* | Study<br>Product | Subjects with<br>Adverse Events | Mild | Moderate | Severe | Not Related | Unlikely | Probably | Likely | Related |
| Abdominal pain | Х | X | Х | Х | X | Х | Х | Х | Х | Х |
| Constipation | X | X | X | X | X | X | X | X | X | X |
| Dry throat | X | X | X | X | X | X | X | X | X | X |
| Headache | X | X | X | X | X | X | X | X | X | X |
| | X | X | X | X | X | X | X | X | X | X |
| Study Product A | | X | Х | X | X | X | Х | Х | Х | Х |
| Study Product B | | X | X | X | X | X | X | X | X | X |
| Study Product C | | X | X | X | X | X | X | X | X | X |
| Study Product D | | X | X | X | X | X | X | X | X | X |
| Study Product E | | X | X | X | X | X | X | X | X | X |
| Study Product F | | X | X | X | X | X | X | X | X | X |
| Study Product G | | X | X | X | X | X | X | X | X | X |
| Study Product H | | X | X | X | X | X | X | X | X | X |
| Overall | | X | Χ | X | X | X | X | X | X | X |

Note: \* Adverse events are classified according to MedDRA Version 22.0.

When a subject experienced the same AE at more than one level of intensity during a product use period, only the most severe one was counted.

When a subject experienced the same AE at more than one level of product relationship during a product use period, only the one most closely related to study product was counted.

Product  $X = \langle \rangle$ 

Program: /CAXXXXX/sas prg/stsas/tab cdash tblae3a auto.sas DDMMMYYYY HH:MM

Programmer Note: Table 14.3.1.2.3 will have three rows for the three study arms and an overall row. The column header will be study product arm.

| Nerudia Ltd. |
|----------------------------------------|
| NER 01/003 <i>my</i> blu™ E-cigarettes |
| Clinical Study Report No. CA22736 |

Serious adverse event table (Table 14.3.2.1) will be in the following format.


Table 14.3.2.1 Serious Adverse Events

There were no serious adverse events recorded during the study

Program: /CAXXXXX/sas\_prg/stsas/tab cdash\_tblae\_ser.sas DDMMMYYYY HH:MM

### Post-text Tables 14.3.4.1, 14.3.4.2, and 14.3.4.3 will be in the following format:


Table 14.3.4.1 Out-of-Range Values and Recheck Results - Serum Chemistry (Safety Population)

| Subject<br>Number | Age#/<br>Sex | Study<br>Period | Day | Hour | Date | Time | Parameter1<br><range><br/>(Unit)</range> | Parameter2<br><range><br/>(Unit)</range> | Parameter3<br><range><br/>(Unit)</range> | Parameter4<br><range><br/>(Unit)</range> | Parameter5<br><range><br/>(Unit)</range> |
|---|---|---|---|---|---|---|---|---|---|---|---|
| X | XX/X | Screen | | | DDMMYYYY | | | | | XX LY | XX HY |
| | | X<br>X | -X | -X.XX<br>-X.XX | DDMMYYYY<br>DDMMYYYYY | | XX HY | XX LY | XX LY | | XX HY |
| | | | X | X.XX | DDMMYYYY | HH:MM:SS | | | XX HY | | |

Programmer Note: Table 14.3.4.2 (Hematology) and Table 14.3.4.3 (Urinalysis) will resemble Table 14.3.4.1. Replace Parameter1, 2 etc. with actual lab tests in the study. Sort unscheduled assessment and early termination chronologically with other scheduled assessments and rechecks. Recheck should be sorted with the scheduled time point the recheck is for.

Note: # Age is calculated from the date of informed consent. F = Female, M = Male H = Above Reference Range, L = Below Reference Range PI Interpretation: N = Not Clinically Significant, Y = Clinically Significant

Study Part 1 is up to Day 9 and Study Part 2 is from Day 10 onward.

Program: /CAXXXXX/sas prg/stsas/tab/programname.sas DDMMYYYY HH:MM
### Post-text Table 14.3.4.4 will be in the following format:


Table 14.3.4.4 Clinically Significant Values and Recheck Results (Safety Population)

| Subject<br>Number | | | Day | Hour | Date | Time | Department | Test | Result | = | Reference Range | Unit |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| X | XX/X | X | X | | | | Serum Chemistry<br>Serum Chemistry | | | | X - X<br>X - X | mg/dL<br>mg/dL |
| | | | | X.XX | DDMMYYYYY | HH:MM:SS | Serum Chemistry | XXXXXXXX | XXX | HY+ | X - X | ma/dL |

Programmer note: All time points for a subject/test with at least one value deemed as CS by the PI will be presented in this table. If no event meets this criteria then include a statement as follows: 'There were no clinical laboratory results documented as clinically significant by the Principal Investigator.'

Note: # Age is calculated from the date of informed consent. F = Female, M = Male

H = Above Reference Range

Computer: Y = Clinically Significant

PI Interpretation: R = Recheck Requested, + = Clinically Significant

Study Part 1 is up to Day 9 and Study Part 2 is from Day 10 and afterwards.

### Nerudia Ltd.

### NER 01/003 *my*blu™ E-cigarettes

### Clinical Study Report No. CA22736

Serum chemistry, hematology, and urinalysis summary tables (Table 14.3.5.1. Table 14.3.5.2, and 14.3.5.3) will be in the following format.

Table 14.3.5.1 Clinical Laboratory Summary - Serum Chemistry (Safety Population)

Time Point

| | Reference | | | | |
|---|---|---|---|---|---|
| Laboratory Test (units) | Range | Statistic | Screening | Check-in | End-of-Study |
| Testname (unit) | XX - XX # | n<br>Mean<br>SD<br>Minimum<br>Median<br>Maximum | X<br>X.X*<br>X.XX<br>XX<br>XX<br>X.X<br>XX | X<br>X.X<br>X.XX<br>XX<br>XX<br>XX<br>XX | X<br>X.X<br>X.XX<br>XX<br>XX<br>XX<br>XX |
| Testname (unit) | XX - XX | n<br>Mean<br>SD<br>Minimum<br>Median<br>Maximum | X<br>X.X<br>X.XX<br>XX<br>XX<br>X.X<br>XX | X<br>X.X<br>X.XX<br>XX<br>X.X<br>XX | X<br>X.X<br>X.XX<br>XX<br>X.X<br>XX |

Note: # = Lowest of the lower ranges and highest of the higher ranges are used. Refer to Appendix 16.1.10.1 for the breakdown.

Program: /CAXXXXX/sas prg/stsas/tab/programname.sas DDMMYYYY HH:MM


<sup>\*</sup> Above Reference Range, ^ Below Reference Range

## Nerudia Ltd. NER 01/003 *my*blu™ E-cigarettes

## Clinical Study Report No. CA22736

Vital sign summary table (Table 14.3.5.4) will be in the following format.

Table 14.3.5.4 Vital Sign Summary (Safety Population)

| Vital Sign (units) | Time Point | Statistic | |
|---|---|---|---|
| Testname (unit) | Screening | n<br>Mean<br>SD<br>Minimum<br>Median<br>Maximum | X<br>X.X<br>X.XX<br>XX<br>XX<br>XX |
| | Check-in | n<br>Mean<br>SD<br>Minimum<br>Median<br>Maximum | X<br>X.X<br>X.XX<br>XX<br>XX<br>X.X |

Note: Study Part 1 is up to Day 9 and Study Part 2 is from Day 10 and afterwards.

Program: /CAXXXXX/sas\_prg/stsas/tab cdash\_vitsummary.sas DDMMMYYYY HH:MM


## Nerudia Ltd.

## NER 01/003 *my*blu™ E-cigarettes

Clinical Study Report No. CA22736

### ECG summary tables (Table 14.3.5.5) will be in the following format.

Table 14.3.5.5 12-Lead Electrocardiogram Summary (Safety Population) (Safety Population)


| | | | Time Point | |
|---|---|---|---|---|
| Parameter (units) | Statistic | Screening | Check-in | End-of-Study |
| Testname (unit) | n<br>Mean<br>SD<br>Minimum<br>Median | X<br>X.X<br>X.XX<br>XX<br>XX<br>XX | X<br>X.X<br>X.XX<br>XX<br>XX<br>XX | X X X X X X X X X X X X X X X X X X X |
| | Maximum | XX | XX | XX |
| Testname (unit) | n<br>Mean<br>SD<br>Minimum<br>Median<br>Maximum | X<br>X.X<br>X.XX<br>XX<br>XX<br>XX<br>XX | X<br>X.X<br>X.XX<br>XX<br>XX<br>X.X | X<br>X.X<br>X.XX<br>XX<br>X.X<br>XX |

Spirometry summary tables (Table 14.3.5.6) will be in the following format.


Table 14.3.5.6 Spirometry Summary (Safety Population) (Safety Population)

| | | | Pre Broncho | dilator | Post Bronchodilator | | |
|---|---|---|---|---|---|---|---|
| Parameter (units) | Statistic | Screening | Day 9 | Day 14 | Screening | Day 9 | Day 14 |
| Testname (unit) | n | X | X | X | X | X | X |
| | Mean | X.X | X.X | X.X | X.X | X.X | X.X |
| | SD | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| | Minimum | XX | XX | XX | XX | XX | XX |
| | Median | X.X | X.X | X.X | X.X | X.X | X.X |
| | Maximum | XX | XX | XX | XX | XX | XX |
| Testname (unit) | n | X | X | X | X | X | X |
| | Mean | X.X | X.X | X.X | X.X | X.X | X.X |
| | SD | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| | Minimum | XX | XX | XX | XX | XX | XX |
| | Median | X.X | X.X | X.X | X.X | X.X | X.X |
| | Maximum | XX | XX | XX | XX | XX | XX |

Note: Study Part 1 is up to Day 9 and Study Part 2 is from Day 10 and afterwards.

### 11. LISTING SHELLS

The following listing shells provide a framework for the display of data from this study. The shells may change due to unforeseen circumstances. These shells may not be reflective of every aspect of this study, but are intended to show the general layout of the listings that will be presented and included in the final report. These listings will be generated off of the SDTM Version 1.4. All listings will be presented in Courier New size font 9.


Appendix 16.1.10.1 Clinical Laboratory Reference Ranges

| Laboratory Group | Test Name | Sex | Age Category | Reference Range | Unit |
|---|---|---|---|---|---|
| Serum Chemistry | Test Name<br>Test Name | XXXXXX | XX-XX<br>XX-XX | XX-XX<br>XX-XX | units<br>units |
| | Test Name<br>Test Name | XXXXXX | XX-XX | XX-XX<br>XX-XX | units<br>units |
| Hematology | Test Name<br>Test Name<br>Test Name<br>Test Name | XXXXXX<br>XXXXXX<br>XXXXXX | XX-XX<br>XX-XX<br>XX-XX | XX-XX<br>XX-XX<br>XX-XX<br>XX-XX | units<br>units<br>units<br>units |
| Urinalysis | Test Name<br>Test Name<br>Test Name<br>Test Name | XXXXXX<br>XXXXXX<br>XXXXXX | XX-XX<br>XX-XX<br>XX-XX<br>XX-XX | XX-XX<br>XX-XX<br>XX-XX<br>XX-XX | units<br>units<br>units<br>units |

<similar for remaining Laboratory Groups and Test Names>


#### Appendix 16.2.1 Subject Discontinuation (Safety Population)

| Subject | C+udiz | Randomized | Sequence/Arm | | Completed | | |
|---|---|---|---|---|---|---|---|
| Number | Period | Part 1 | Part 2 | Date | _ | Primary Discontinuation Reason | Specify |
| X | XXXX | XXXX | X | DDMMYYYYY | YES | | |
| X | XXXX | XXXX | X | DDMMYYYYY | NO | Adverse Event | XXXXXXXXXX |

Note: Product X: < >


#### Appendix 16.2.2 Protocol Deviation

| Subject | Any | Study | Study | Deviation | Deviation | Other, | Deviation | Deviation |
|---|---|---|---|---|---|---|---|---|
| Number | Deviation | Period | Product | Category | Type | Specify | Date | Term |
| X | YES | XXX | X | XXXX | XXXX | | DDMMYYYY | XXXXXXXXXX |

Note: Product X: < >


### Appendix 16.2.4.1.1 Demographics (Safety Population)

| Subject | Randomized S | Randomized Sequence/Arm | | Age* | | | | Height | Weight | Body Mass<br>Index | Informed<br>Consent |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Number | Part 1 | Part 2 | Birth | (yrs) | Sex | Race | Ethnicity | (cm) | (kg) | $(kg/m^2)$ | Date |
| Х | XXXX | X | DDMMYYYY | XX | XXXXXX | XXXXXX | XXXXXX | XXX | XX.XX | XX.XX | DDMMYYYYY |
| X | XXXX | X | DDMMYYYYY | XX | XXXXXX | XXXXXX | XXXXXX | XXX | XX.XX | XX.XX | DDMMYYYY |
| X | XXXX | X | DDMMYYYYY | XX | XXXXXX | XXXXXX | XXXXXX | XXX | XX.XX | XX.XX | DDMMYYYYY |

Note: \* Age is calculated from the date of first study product use.


### Appendix 16.2.4.1.2 Reproductive Status (Safety Population)

| Subject<br>Number | A Woman of<br>Childbearing<br>Potential? | Last<br>Menstrual<br>Period | Last<br>Pregnancy | Outcome | | Lactating, Pregnant, or Plan to Become Pregnant? | Reproductive<br>Status | | Agree to Use<br>Double Barrier |
|---|---|---|---|---|---|---|---|---|---|
| X | XXXXXX | DDMMYYYY | XXXXXXX | XXXXXX | DDMMYYYYY | XXXXXX | XXXXXXX | XXXXXXX | XXX |


### Appendix 16.2.4.2 Physical Examination (Safety Population)

| Subject<br>Number | Study<br>Period | Time Point | Date | Body System<br>or Organ Class | Reason for<br>Not Done | Finding | Clinically<br>Significant? | Comment |
|---|---|---|---|---|---|---|---|---|
| Х | Screen | XXXXXX | DDMMYYYY | XXXXXXXX | | XXXXXX | XXXXXX | |


#### Appendix 16.2.4.3.1 Medical History (Safety Population)

| | | | Medical | Start | | End | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>Number | Study<br>Period | Time Point | History<br>Present | Date Time | | Date | Time | Reported Term for the Medical History | Clinically<br>Significant | |
| | Saroon | | VVV | | LILI • MM | | LILI • MM | | VVV | _ |

Programmer Note: Date can be YYYY, MMMYYYY, or DDMMMYYYY based on individual subject data.

Appendix 16.2.4.3.1 Allergy History (Safety Population)

| Subject<br>Number | Study<br>Period | Time Point | Allergy<br>Present | Category<br>of Allergy | State<br>Date | End<br>Date | Clinical<br>Significance | Investigator<br>Judgement |
|---|---|---|---|---|---|---|---|---|
| X | Screen | xxxxxxx | XXX | XXXXXXXXXX | DDMMMYYYY | DDMMMYYYY | XXXXX | XXXXXXXX |

Programmer Note: Date can be YYYY, MMMYYYY, or DDMMMYYYY based on individual subject data.


Appendix 16.2.4.3.2 Surgical History (Safety Population)

| Subject<br>Number | - | Time Point | Surgical<br>History<br>Present | Date of<br>Surgical Event | 2 4 | Clinically<br>Significant |
|---|---|---|---|---|---|---|
| × | Screen | XXXXXXX | XXX | DDMMMYYYY | | |

Programmer Note: Date can be YYYY, MMYYYY, or DDMMYYYY based on individual subject data.

Appendix 16.2.4.4 Smoking History (Safety Population)

| Subject | Study | Cigarettes | Start | Type of | Cigarette | Cigarette | Cigarette | Cigarette | | Question* | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Number | Period | Per Day | Date | Cigarette | Brand | Style | Flavor | Length | 1 | 2 | 3 | 4 |
| | Screen | YY | | Menthol | | | YYYYYY | YYYYYY | YYY | | VV | YYY |

Programmer Note: Date can be YYYY, MMMYYYY, or DDMMMYYYY based on individual subject data.

- Note: Question 1 = Has the subject used any other nicotine-containing products other than manufactured combustible cigarettes (e.g., e-cigarettes, roll-your-own cigarettes, bidis, snuff, nicotine inhaler, pipe, cigar, chewing tobacco, nicotine patch, nicotine spray, nicotine lozenge, or nicotine gum) within the last 14 days?
  - Question 2 = Has the subject used any prescription smoking cessation treatments, including, but not limited to, varenicline (Chantix®) or bupropion (Zyban®) within the last 3 months?
  - Question 3 = Is the subject a self-reported puffer (i.e., adult smoker who draws smoke from the cigarette into the mouth and throat but does not inhale)?
  - Question 4 = Is the subject planning to quit smoking during the study or postponing a quit attempt in order to participate in the study?

Program: /CAXXXXX/sas prg/stsas/lis/programname.sas DDMMYYYY HH:MM


Appendix 16.2.4.5 Caffeine, Alcohol, and Drug History (Safety Population)

| Cubicat | | Alcohol | | | | Caffeine | | | | Drug | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Number | Consumption? | Abuse? | Туре | Amount | Frequency | Consumption? | Туре | Amount | Frequency | Abuse? | End Date | Used | Amount | Frequency |
| X | XX | XXX | XXX | XXX | XXXXX | XX | XXX | XXX | XXXXX | XX | DDMMYYYY | XXX | XXX | XXXXX |

Programmer Note: Date can be YYYY, MMYYYY, or DDMMYYYY based on individual subject data.


Appendix 16.2.5.1.1 Inclusion Criteria

1. <>

2. <> 3. <>

4. <>

5. < >

etc.

## Nerudia Ltd. NER 01/003 *my*blu™ E-cigarettes

Clinical Study Report No. CA22736

Page 1 of X Appendix 16.2.5.1.2 Exclusion Criteria

1. < >

2. <>

3. < >

4. < >

5. < > etc.


#### Appendix 16.2.5.2 Subject Eligibility (Safety Population)

| Subject<br>Number | Study<br>Period | Time Point | Date | Time | Did Subject meet all eligibility criteria? | Criterion Not Met* | Comment |
|---|---|---|---|---|---|---|---|
| X | Screen | XXXX | DDMMYYYYY | HH:MM | YES | | |
| X | Screen | XXXX | DDMMYYYY | HH:MM | NO | EXCLUSION X | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| X | Screen | XXXX | DDMMYYYY | HH:MM | YES | | |
| X | Screen | XXXX | DDMMYYYY | HH:MM | NO | INCLUSION X | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |

Note: \* Please refer to Appendix 16.2.5.1.1 and Appendix 16.2.5.1.2 for specific inclusion and exclusion criteria.


### Appendix 16.2.5.3 Randomization (Safety Population)

| Subject<br>Number | Study<br>Period | Time Point | Date | Time | Randomization<br>Performed | Randomized<br>Sequence | Randomized<br>Arm |
|---|---|---|---|---|---|---|---|
| X | X | XXXXXX | DDMMYYYY | HH:MM | XXX | XXXX | X |

Note: Product X: < > Arm X: < >


Appendix 16.2.5.4.1 Usual Brand Cigarette (Safety Population)

| Subject<br>Number | Study<br>Period | Time Point | Date | Time | Number of Cigarettes<br>per Pack | Number of Unopened<br>Packs from Subject | Comment |
|---|---|---|---|---|---|---|---|
| X | X | XXXXXX | DDMMYYYY | HH:MM | XX | XXX | |


Appendix 16.2.5.4.2 Test Product Administration (Safety Population)

| Subject<br>Number | Study<br>Period | Product | Time Point | Start<br>Date | Start<br>Time | End<br>Time | Total Number of Inhalations | 3 Seconds<br>Per Puff? | Comment for<br>Duration | Missed<br>Puff? | Comment for<br>Missed Puff |
|---|---|---|---|---|---|---|---|---|---|---|---|
| X | X | X | XXXXXX | DDMMMYYYY | HH:MM | HH:MM | XXX | XXX | | XXX | |

Note: Product X: < >


### Appendix 16.2.5.4.3 Ad Libitum Product Use (Safety Population)

| Subject<br>Number | Study<br>Period | Product | Time Point | Start<br>Date | Start<br>Time | Stop<br>Date | Stop<br>Time | No. of Pods<br>Dispensed | No. of Pods<br>Used | |
|---|---|---|---|---|---|---|---|---|---|---|
| X | X | × | XXXXXX | DDMMMYYYY | HH:MM | DDMMMYYYY | HH:MM | XXX | XXX | <br> |

Note: Product X: < >


Appendix 16.2.5.4.4 Product Use Behavior - Pod Weight (Safety Population)

| Subject<br>Number | | Product | Time Point | Pre Weight<br>(g) | Post Weight<br>(g) | Comment |
|---|---|---|---|---|---|---|
| X | X | Х | HH:MM | X.XXXX | X.XXXX | |

Note: Product X: < >


Appendix 16.2.5.5.1 Blood Draw Times (Safety Population)

| Subject<br>Number | | Product | Time Point | Date | Actual<br>Time | Comments |
|---|---|---|---|---|---|---|
| X | X | X | XXXXXXXX | DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY | HH:MM:SS | |

Note: Product X: < >


### Appendix 16.2.5.5.2 Urine Collection (Safety Population)

| Subject<br>Number | Study<br>Period | Product | Time Point | Start /Stop<br>Date / Time | Void/Container Storage<br>Date / Time | Tare Weight<br>(g) | Total Weight (g) | Urine Weight<br>(g) | Comment |
|---|---|---|---|---|---|---|---|---|---|
| X | X | X | XXXXXXXX | DDMMYYYY/HH:MM:SS<br>DDMMMYYYY/HH:MM:SS | DDMMYYYY/HH:MM:SS<br>DDMMYYYYY/HH:MM:SS | XXXX | XXXX | XXXX | |

Note: Product X: < >


#### Appendix 16.2.5.6 Meal Times (Safety Population)

| Subject<br>Number | Study<br>Period | Product | Time Point | Category<br>of Meal | Received and Consumed the Meal | Start<br>Date | Start<br>Time | Comments | |
|---|---|---|---|---|---|---|---|---|---|
| X | X | X | XXXXXX | XXXXXXX | XXXX | DDMMMYYYY | HH:MM:SS | | _ |

Note: Product X: < >


Appendix 16.2.5.7 Prior and Concomitant Medications (Safety Population)

| Subject<br>Number | Any<br>Medications? Product | Medication<br>(WHO DD*) | Dosage Route | Start<br>Date | Start<br>Time | Stop<br>Date | Stop<br>Time | Frequency | Indication | Continuing? | ^Prior<br>to<br>Use |
|---|---|---|---|---|---|---|---|---|---|---|---|
| X | NO | None | | | | | | | | | |
| X | NO | None | | | | | | | | | |
| X | YES X | XXXXXXXX | | K DDMMYYYYY<br>K DDMMYYYYY | | | | | XXXXXXXX | XXX<br>XXX | YES<br>NO |

Note:  $\star$  Concomitant medications are coded with WHO Drug Dictionary Version 01Sep2019-b3.

WHO DD = World Health Organization Drug Dictionary  $^{\circ}$  is derived based on the first study product use.

Product X: < >

Program: /CAXXXXX/sas\_prg/stsas/lis/programname.sas DDMMMYYYY HH:MM

Programmer Note: Other dose unit, route, frequency may presented if applicable.

### Appendices for blood biomarkers will have the following format:

Study Blood

-1

14

Appendix 16 2 6 2 1 Blood COHb Saturation (Outcomes Population)

| ybbe | 10.2.0 | .2.1 b1000 C | OID Sacurat | TOIL (Outcomes I | оритастоп) | |
|---|---|---|---|---|---|---|
| Blood COHb<br>% Saturation | | | | 4 - Day -1<br>% Change | Day 14<br>Change | |
| XXX<br>XXX<br>XXX | XXX<br>XXX<br>XXX | XXX<br>XXX<br>XXX | XXX<br>XXX<br>XXX | XXX<br>XXX<br>XXX | XXX<br>XXX<br>XXX | XXX<br>XXX<br>XXX |


Note: Arm I:  $myblu^{m}$ 

Subject

XXXXX

Arm J: Combustible Cigarette

Arm K: Dual Use

Number Sequence Day

Program: /CAXXXXX/sas\_prg/stsas/lis\_PROGRAMNAME.sas DDMMMYYYY HH:MM

Programming Notes: Day 14 - Day -1 is only presented for Arm I

### Appendices for urine biomarkers except nicotine and metabs will have the following format:


Appendix 16.2.6.2.2 Urine NNAL (Outcomes Population)

| Subject<br>Number | Study<br>Arm | Study<br>Day | <br>xg/mL) | NNAL<br>(xg/24 hours) | xg/g cr | Day<br>Change | 9 - Day 1<br>% Change | Day<br>Change | 14 - Day -1<br>% Change | Day 1<br>Change | 14 - Day 9<br>% Change |
|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXXX | X | -1<br>9 | XXX | XXX<br>XXX | XXX<br>XXX | XXX | XXX<br>XXX | XXX | XXX<br>XXX | XXX<br>XXX | XXX<br>XXX |
| | | 14 | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |

Note: cr = creatinineArm I:  $myblu^{m}$ 

Arm J: Combustible Cigarette

Arm K: Dual Use

Program: /CAXXXXX/sas\_prg/stsas/lis\_PROGRAMNAME.sas DDMMMYYYY HH:MM

Programming Notes: Day 14 - Day -1 is only presented for Arm I


Appendix 16.2.6.2.15.1 Urine Nicotine and Metabolites (Outcomes Population)

| Subject<br>Number | Study<br>Day | Nicotine<br>(ng/mL) | Nicotine<br>Glucuronide<br>(ng/mL) | Cotinine<br>(ng/mL) | Cotinine<br>Glucuronide<br>(ng/mL) | Trans-3-hydroxy<br>Cotinine<br>(ng/mL) | Trans-3-hydroxy<br>Cotinine<br>Glucuronide<br>(ng/mL) |
|---|---|---|---|---|---|---|---|
| <br>XXXXXX | -1 | XXX | XXX | XXX | XXX | XXX | XXX |
| | 9 | XXX | XXX | XXX | XXX | XXX | XXX |
| | 14 | XXX | XXX | XXX | XXX | XXX | XXX |

Program: /CAXXXXX/sas\_prg/stsas/lis\_PROGRAMNAME.sas DDMMMYYYY HH:MM


#### Appendix 16.2.6.3.1 PES Questionnaire (Outcomes Population)

- 1. Was it satisfying?
- 2. Did it taste good?
- 3. Did you enjoy the sensations in your mouth?
- 4. Did it calm you down?
- 5. Did it make you feel more awake?
- 6. Did it make you feel less irritable?
- 7. Did it help you concentrate?
- 8. Did it reduce your hunger for food?
- 9. Did it make you dizzy?
- 10. Did it make you nauseous?
- 11. Did it immediately relieve your craving for a cigarette?
- 12. Did you enjoy it?
- 13. Did it relieve withdrawal symptoms?
- 14. Did it relieve the urge to smoke?
- 15. Was it enough nicotine?
- 16. Was it too much nicotine?
- 17. Was it easy to use?
- 18. Were there bothersome side effects?
- 19. Were you comfortable using the product in public?
- 20. Did you still have a craving for a cigarette after using the product?
- 21. Are you concerned that you would become dependent on this product?

Program: /CAXXXXX/sas prg/pksas/PROGRAMNAME.SAS DDMMMYYYY HH:MM

### Nerudia Ltd.

### NER 01/003 myblu™ E-cigarettes

### Clinical Study Report No. CA22736

Appendix 16.2.6.3.2 PES Questionnaire Responses (Outcomes Population)


| Subject | | Study | | | Question | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Number | Product | Day | Session | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | | 21 |
| XXXXXX | X | X | Controlled | Χ | X | X | X | X | X | X | X | X | X | X | X |
| | | | Ad libitum | X | X | X | X | X | X | X | X | X | X | X | X |

Note: Product X: < >

Scale: 1 = not at all, 2 = very little, 3 = a little, 4 = moderately, 5 = a lot, 6 = quite a lot, 7 = extremely Refer to Appendix 16.2.6.3.1 for the description of questions.

Program: /CAXXXXX/sas prg/pksas/PROGRAMNAME.SAS DDMMMYYYY HH:MM

### Nerudia Ltd.

### NER 01/003 myblu™ E-cigarettes

## Clinical Study Report No. CA22736


Appendix 16.2.6.3.3 PES Questionnaire Subscales (Outcomes Population)

| Subject | | Study | | | Subscale | | |
|---|---|---|---|---|---|---|---|
| Number | Product | Day | Session | Satisfaction | Psychological Reward | Aversion | Relief |
| XXXXXX | X | XXXX | Controlled | X | X | X | X |
| XXXXXX | X | XXXX | Ad libitum | X | X | X | X |

Note: Product X: < >

"Satisfaction" (Average of items 1, 2, 3, and 12); "Psychological Reward" (Average of items 4 through 8);
"Aversion" (Average of 9, 10, 16, and 18);

"Relief" (Average of items 11, 13, 14, 15, and reversed for item 20)

Program: /CAXXXX/sas prg/pksas/PROGRAMNAME.SAS DDMMYYYYY HH:MM


### Appendix 16.2.6.4 Product Liking Questionnaire Responses (Outcomes Population)

| Subject<br>Number | Product | Study<br>Day | Session | How much do you like the test e-cigarette you are using? (VAS Score) |
|---|---|---|---|---|
| XXXXXX | X | X | Controlled<br>Ad libitum | XX<br>XX |

Note: Product X: < >

Program: /CAXXXXX/sas\_prg/pksas/PROGRAMNAME.SAS DDMMMYYYY HH:MM
Appendix 16.2.6.5 Future Intent to Use Questionnaire Responses (Outcomes Population)

| Subject | | Study | | | VAS Score | s |
|---|---|---|---|---|---|---|
| Number | Product | Day | Session | Question 1 | Question 2 | Question 3 |
| XXXXXX | X | Χ | Controlled | XX | XX | XX |
| | | | Ad libitum | XX | XX | XX |

Note: Question 1: How likely are you to continue to smoke after you complete this study?

Question 2: If available, how likely are you to buy your assigned study product in the future?

Question 3: How likely are you to buy an e-cigarette other than your assigned product in the future?

Product X: < >

Program: /CAXXXXX/sas prg/pksas/PROGRAMNAME.SAS DDMMMYYYY HH:MM

Appendix 16.2.6.6.1 PSCDI, PSECDI Questionnaire (Outcomes Population)

- 1. How many cigarettes [times] per day do you usually smoke [use your electronic cigarette]? ([assume that one "time" consists of around 15 puffs or lasts around 10 minutes]) (Scoring: 0-4 times/day = 0, 5-9 = 1, 10-14 = 2, 15-19 = 3, 20-29 = 4, 30+ = 5)
- 2. On days that you can smoke [use your electronic cigarette] freely, how soon after you wake up do you smoke your first cigarette of the day [first use your electronic cigarette]? (Scoring: 0-5 mins = 5, 6-15 = 4, 16-30 = 3, 31-60 = 2, 61-120 = 1, 121+ = 0)
- 3. Do you sometimes awaken at night to have a cigarette [use your electronic cigarette]? (Scoring: Yes = 1, No = 0)
- 4. If yes, how many nights per week do you typically awaken to smoke [use your electronic cigarette]? (Scoring: 0-1 nights = 0, 2-3 nights = 1, 4+ nights = 2)
- 5. Do you smoke [use an electronic cigarette] now because it is really hard to quit? (Scoring: Yes = 1, No = 0)
- 6. Do you ever have strong cravings to smoke [use an electronic cigarette]? (Scoring: Yes = 1, No = 0)
- 7. Over the past week, how strong have the urges to smoke [use an electronic cigarette] been? (Scoring: None/Slight = 0, Moderate/Strong= 1, Very Strong/Extremely Strong = 2)
- 8. Is it hard to keep from smoking [using an electronic cigarette] in places where you are not supposed to? (Scoring: Yes = 1, No = 0)

When you haven't used tobacco [an electronic cigarette] for a while or when you tried to stop smoking [using]...

- 9. Did you feel more irritable because you couldn't smoke [use an electronic cigarette]? (Scoring: Yes = 1, No = 0)
- 10. Did you feel nervous, restless, or anxious because you couldn't smoke [use an electronic cigarette]? (Scoring: Yes = 1, No = 0)
- 11. Total scoring: 0 3 = not dependent, 4 8 = low dependence, 9 12 = medium dependence, 13+ = high dependence.

Program: /CAXXXXX/sas prg/pksas/PROGRAMNAME.SAS DDMMMYYYY HH:MM

## Nerudia Ltd.

## NER 01/003 *my*blu™ E-cigarettes

# Clinical Study Report No. CA22736


Appendix 16.2.6.6.2 PSCDI, PSECDI Questionnaire Responses (Outcomes Population)

| Subject | Study | Study | | | | | | | Quest | ion | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Number | Arm | Day | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | Total Score |
| XXXXXX | X | X | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | | X | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |

Note: Arm I:  $myblu^{m}$ 

Arm J: Combustible Cigarette

Arm K: Dual Use

Refer to Appendix 16.2.6.6.1 for the description of questions.

Program: /CAXXXXX/sas\_prg/pksas/PROGRAMNAME.SAS DDMMMYYYY HH:MM

Appendix 16.2.6.7.1 MTWS-R Questionnaire (Outcomes Population)

Please rate yourself for the period of the last 24 hours.

- 1. Angry, irritable, frustrated
- 2. Anxious, nervous
- 3. Depressed mood, sad
- 4. Difficulty concentrating
- 5. Increased appetite, hungry, weight gain
- 6. Insomnia, sleep problems, awakening at night
- 7. Restless
- 8. Desire or craving to smoke

Program: /CAXXXXX/sas prg/pksas/PROGRAMNAME.SAS DDMMMYYYY HH:MM

## NER 01/003 *my*blu™ E-cigarettes

## Clinical Study Report No. CA22736


Appendix 16.2.6.7.2 MTWS-R Questionnaire Responses (Outcomes Population)

| Subject | Study | Study | | | | | Questi | on | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Number | | Day | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | Total Score |
| XXXXXX | Х | X | <br>X | X | Х | Х | X | X | X | X | XX |
| | | X | X | X | X | X | X | X | X | X | XX |

Note: Arm I:  $myblu^{m}$ 

Arm J: Combustible Cigarette

Arm K: Dual Use

Scale: 0 = none, 1 = slight, 2 = mild, 3 = moderate, 4 = severe Refer to Appendix 16.2.6.7.1 for the description of questions.

Program: /CAXXXXX/sas\_prg/pksas/PROGRAMNAME.SAS DDMMMYYYY HH:MM

# Clinical Study Report No. CA22736

1. <>

2. <>

3. <>

4. < >

5. <>

6. < >

7. <>

8. < >

9. <>

10. < >

Program: /CAXXXXX/sas\_prg/pksas/PROGRAMNAME.SAS DDMMMYYYY HH:MM

## Nerudia Ltd.

### NER 01/003 myblu™ E-cigarettes

### Clinical Study Report No. CA22736

Appendix 16.2.6.8.2 QSU-Brief Questionnaire Responses (Outcomes Population)

| Subject<br>Number | Study<br>Arm | Study<br>Day | 1 | 2 | 3 | 4 | 5 | Quest | | 8 | 9 | 10 | <br>1 | Factor Score 2 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXXXX | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| XXXXXX | X | X | X | X | X | X | X | X | X | X | X | X | X | X |

Note: Arm I: myblu™

Arm J: Combustible Cigarette

Arm K: Dual Use

Scale: 1 = Strongly disagree, 7 = Strongly agree

Factor 1 (anticipation of pleasure from smoking): average of items 1, 3, 6, 7, and 10.

Factor 2 (relief of nicotine withdrawal): average of items 2, 4, 5, 8, and 9.

Refer to Appendix 16.2.6.8.1 for the description of questions.

Program: /CAXXXX/sas prg/pksas/PROGRAMNAME.SAS DDMMYYYYY HH:MM


#### Appendix 16.2.6.9 Individual Puff Topography Parameters (Outcomes Population)

| Subject<br>Number | Study<br>Day | Product | Date | | Subject | Cigarette<br>Number/<br>ENDS Number | | Puff<br>Duration<br>(sec) | Puff<br>Volume<br>(mL) | Peak<br>Flow<br>(mL/sec) | Flow | Inter-Puff<br>Interval<br>(sec) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 1 | -1 | N/A | XXXXXXXXX | X:XX:X | Yes | X | X | X.XX | XX | XX | XX | XX |

#### Appendix 16.2.7.1.1 Adverse Events (I of II) (Safety Population)

| Subject S | C+udiz | C+ndr | | | | Onset | | Resolved | | Duration |
|---|---|---|---|---|---|---|---|---|---|---|
| _ | Period | Study<br>Product | UE?^ | Adverse Event* | Preferred Term | Date | Time | Date | Time | (DD:HH:MM) |
| 1 | X | X | Yes | XXXXXXXXXXXX | XXXXXXXXXX XXXXXXX | DDMMYYYY | | DDMMMYYYY | X:XX | XX:XX:XX |

Note: & = Abbreviation for study product use-emergent (UE),

\* = Adverse events are classified according to the MedDRA Version XX.X.

Product X: < >

Appendix 16.2.7.1.2 Adverse Events (II of II) (Safety Population)

| | | | | Onset | | | | | | Relation-<br>ship to | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>Number | | Study<br>Product | Adverse<br>Event | Date | Time | Freq | Severity | Ser* | | Study<br>Product | Action | Unexpected<br>Adverse Event Co | omment |
| 1 | XXX | X | <br>XXXXXXXXXXXXXXXXXXXX | DDMMYYYY | X:XX | <br>Inter | <br>. Mild | XXX | Resolved | XXXXXXXX | None | XXX | |

Note: Ser\* represents Serious event.

Freq represents Frequency: SI = Single Episode, Inter. = Intermittent, Cont. = Continuous

Product X: < >

Appendix 16.2.7.2 Adverse Event Non-Medication Therapy (Safety Population)

#### Procedure

| _ | | | | | Onset | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| _ | Subject<br>Number | | Study<br>Product | Adverse<br>Event | Date | Time | Indication | Given? | Start<br>Date | Start<br>Time | End<br>Date | End<br>Time | Procedure | Dosing<br>Frequency |
| - | 1 | XXX | × | xxxxxxxx | DDMMMYYYY | x:xx | xxxx | Yes | DDMMMYYYY | HH:MM | DDMMMYYYY | HH:MM | *********** | |

Note: Product X: <>

Appendix 16.2.7.3 Adverse Event Preferred Term Classification (Safety Population)

| Cubica | + C+11d-1 | C+11dr | Adverse | | | Unset | |
|---|---|---|---|---|---|---|---|
| Number | t Study<br>Period | Study<br>Product | Adverse<br>Event | Preferred Term | Body System | Date | Time |
| 1 | X | X | XXXXXX XXXXX XXXX XXXXX | XXXXXXXXX XXXXXX | XXXXXXXXXXXXXXXXXX | DDMMYYYY | X:XX |

Note: \* = Adverse events are classified according to the MedDRA Version XX.X. Product X: < >

#### Appendices 16.2.8.1.2 to 16.2.8.1.4 will have the following format.


Appendix 16.2.8.1.1 Clinical Laboratory Report - Serum Chemistry (Safety Population)

| Subject<br>Number | Age/<br>Sex | Study<br>Period | Day | Date | Parameter1<br>< Range><br>(Unit) | Parameter2<br>< Range><br>(Unit) | Parameter3<br>< Range><br>(Unit) | Parameter4<br>< Range><br>(Unit) | Parameter5<br>< Range><br>(Unit) | Parameter6<br>< Range><br>(Unit) |
|---|---|---|---|---|---|---|---|---|---|---|
| X | XX | Screening<br>XXXXXX | | DDMMYYYY<br>DDMMYYYYY | XX HN<br>XX HN | XX<br>XX | XX<br>XX | XX<br>XX<br>XX | XX HN<br>XX HN | XX<br>XX |
| | | XXXXXX | X | DDMMYYYY | XX HN | XX | XX | XX | XX HN | XX |

Note: H = Above Reference Range, L = Below Reference Range PI flag: <math>Y = Clinically significant, N = not clinically significant

Program: /CAXXXXX/ECR/sas\_prg/stsas/lis\_PROGRAMNAME.sas DDMMMYYYY HH:MM

Programmer Note: Replace Parameter1, 2 etc. with actual lab tests in the study.

Appendix 16.2.8.1.5 Clinical Laboratory Report - Comments (Safety Population)

| Subject<br>Number | Age/<br>Sex | Study<br>Period | Day | Date | Department | Test | Result | Unit | Comment |
|---|---|---|---|---|---|---|---|---|---|
| X | XX | Screening | | DDMMYYYY | XXXXXX | XXXXXXXXXXXXX | XX | XXXXXX | XXXXXXXXXXXXX |

Appendix 16.2.8.1.6 Alcohol Breath Testing (Safety Population)

| | | | Alcohol Brea | ath Testing | |
|---------|--------|------------|--------------|-------------|--------|
| Subject | Study | | | | |
| Number | Period | Time Point | Date | Time | Result |
| Х | XX | XXX | DDMMYYYY | HH:MM | XXXX |

Appendix 16.2.8.2 Vital Signs (Safety Population)

| | | | | | | Bloo | d Pressure (mmHg) | | Respir- | - Temper- | - | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | t Study<br>Visit | Product | Time Point | Date | Time | Tost | <br>Systolic/Diastolic | Pulse<br>(bpm) | ation | ature<br>(℃) | Weight<br>(ka) | Commont |
| Number | VISIC | Product | THRE POINT | Date | 11111E | rest | Systolic/Diastolic | (DDIII) | (rpm) | ( C) | (Kg) | Comment |
| X | Screening | | XXXXXXXXXX | DDMMYYYY | X:XX | SIT5 | XXX/ XX | XX | XX | XX.X | XXX.X | |
| | X | X | XXXXXXXXXX | DDMMYYYYY | XX:XX | SIT5 | XXX/ XX | XX | XX | XX.X | | |

Note: Product X: < >

Page 1 of 1

Appendix 16.2.8.3 12-Lead Electrocardiogram (Safety Population)

| | Study<br>Period | Time Point | Date | Time | Overall<br>Interpretation | Heart<br>Rate<br>(bpm) | PR<br>(msec) | QRS<br>(msec) | QT<br>(msec) | QTcF*<br>(msec) | Specify | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 1 | Screen | | DDMONYYYY | X:XX:XX | ANCS | XX | XXX | XX | XXX | XXX | EARLY REPOLARIZATION; LE | FT |
| | XXXXX | XXXXXXXXX | DDMONYYYY<br>DDMONYYYY | | | XX | XXX | XX<br>XX | XXX | XXX | LEFT AXIS DEVIATION | |

Note: ANCS = Abnormal, Not Clinically Significant

QTcF\* = QT corrected for heart rate using Fridericia's correction. # = QTc > 450, @ = QTc change from baseline greater than 30 msec

Program: /CAXXXXX/sas\_prg/stsas/standardlis/cdash\_lis\_ecg.sas 27NOV2015 18:35

# Nerudia Ltd.

# NER 01/003 *my*blu™ E-cigarettes

# Clinical Study Report No. CA22736

Appendix 16.2.8.4 Carbon Monoxide Breath Test (Safety Population)

Subject Study

| Number | | Date | Time | Result | (ppm) | Comment |
|--------|--------|----------|-------|--------|-------|---------|
| Х | Screen | DDMMYYYY | HH:MM | XXX | | |

Program: /CAXXXXX/ECR/sas\_prg/stsas/lis\_PROGRAMNAME.sas DDMMYYYYY HH:MM


Appendix 16.2.8.5 Administration of Albuterol (Safety Population)

| Subject<br>Number | | Time Point | | Date | Time |
|---|---|---|---|---|---|
| X | XXXXX | XXXXXXXX | Time of 1st Albuterol puff administered:<br>Time of 2nd Albuterol puff administered:<br>Time of 3rd Albuterol puff administered:<br>Time of last Albuterol puff administered: | DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY | HH:MM<br>HH:MM<br>HH:MM<br>HH:MM |
| | XXXXX | XXXXXXX | Time of 1st Albuterol puff administered:<br>Time of 2nd Albuterol puff administered:<br>Time of 3rd Albuterol puff administered:<br>Time of last Albuterol puff administered: | DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY | HH:MM<br>HH:MM<br>HH:MM |

Appendix 16.2.8.6 Spirometry (Safety Population)


| | Study<br>Period | | Event* | Date | Time | FVC<br>(L) | FVC<br>%Predicted | FEV1<br>(L) | FEV1<br>%predicted | FVC:FEV1<br>Ratio | FVC:FEV1<br>Ratio<br>%Predicted | FEF<br>25-75% | FEF 25-75%<br>%Predicted | | FVC<br>Change |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| X | Screen | XXX | Pre | DDMMYYYYY | HH:MM | XX | XX | XX | XX | XX | XX | XX | XX | | |
| | | | Post | DDMMYYYY | HH:MM | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | XXXX | XXX | Pre | DDMMYYYY | HH:MM | XX | XX | XX | XX | XX | XX | XX | XX | | |
| | | | Post | DDMMMYYYY | HH • MM | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |

Note: \* pre = pre-bronchodilator, post = post-bronchodilator

# Nerudia Ltd. NER 01/003 *my*blu™ E-cigarettes

### Clinical Study Report No. CA22736


Appendix 16.2.8.6 Tobacco Cessation Information (Safety Population)

| Subject | at Ctuder | | Question | | | |
|---|---|---|---|---|---|---|
| | ct Study<br>r Period | Date | Time | 1 | 2 | Comment |
| X | XXXXXX | DDMMYYYY | HH:MM | XXX | XXX | |
| X | XXXXXX | DDMMMYYYY | HH:MM | XXX | XXX | |

Note: Question 1 = Has the subject been advised that in order to reduce the health effects of smoking and using smokeless tobacco products, the best thing to do is to quit?

Question 2 = Has the subject been provided the Quit Assist card and referred to the Quit Assist website?